# The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for A Placebo Controlled,
Double-blind, Multi-centre, Single Dose, Parallel Group,
Randomised Clinical Trial of GSK2862277 in Patients
undergoing Oesophagectomy Surgery

Compound Number : GSK2862277

Effective Date : 17-NOV-2015

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol TFR116341.
- This RAP is intended to describe the planned efficacy, safety & tolerability, pharmacokinetics and pharmacodynamic analyses required for the study.
- This version includes amendments to the originally approved RAP.
- This RAP will be provided to the study team members to convey the content of i) the interim analyses output (including sample size re-estimation) and ii) the Statistical Analysis Complete (SAC) deliverable.
- Note: Analyses and outputs to support the exploratory translational sub-study will be covered in a separate stand-alone RAP and such outputs are not expected to form part of the SAC deliverable for the main study

#### **Author's Name and Functional Area:**

| PPD | | |
|--------------|-------------------------------|-------------|
| Manager, Sta | tistics (Clinical Statistics) | 17-NOV-2015 |
| _ | Clinical Statistics) | |

#### Approved via e-mail by:

| PPD | 17-NOV-2015 |
|--------------------------------|--------------|
| Director (Clinical Statistics) | 17-INOV-2013 |

Copyright 2015 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | REPC | ORTING & ANALYSIS PLAN SYNPOSIS | 5 |
| ١. | 1.1. | RAP Amendments | |
| 2. | SUMN | MARY OF KEY PROTOCOL INFORMATION | 10 |
| | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | 10 |
| | 2.2. | Study Objective(s) and Endpoint(s) | 10 |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses | 12 |
| 3. | DI ANI | INED ANALYSES | 10 |
| ა. | 3.1. | Interim Analyses | |
| | 3.1. | 3.1.1. Interim analysis #1: Unblinded safety review after approx | |
| | | 10 patients have completed Day 7 visit; roughly 5 per | • |
| | | study drug arm | 13 |
| | | 3.1.2. Interim analysis #2: Unblinded safety review, futility | 10 |
| | | analysis and sample size re-estimation after approx 40 | |
| | | patients have completed Day 7 visit; roughly 20 per stud | V |
| | | drug arm. | • |
| | 3.2. | Final Analyses | |
| | | • | |
| 4. | ANAL | YSIS POPULATIONS | |
| | 4.1. | Protocol Deviations | 20 |
| _ | CONC | CIDEDATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING VENTIONS | 21 |
| | CON | VENTIONS | 21 |
| 6. | STUD | DY POPULATION ANALYSES | 22 |
| | 6.1. | Overview of Planned Analyses | |
| | | · | |
| 7. | PRIM | ARY STATISTICAL ANALYSES | |
| | 7.1. | Efficacy Analyses | |
| | | 7.1.1. Overview of Planned Efficacy Analyses | |
| | | 7.1.2. Planned Efficacy Statistical Analyses | <mark>25</mark> |
| 8. | SECC | ONDARY STATISTICAL ANALYSES | 20 |
| Ο. | 8.1. | Efficacy Analyses | |
| | 0.1. | 8.1.1. Overview of Planned Efficacy Analyses | |
| | | 8.1.2. Planned Efficacy Statistical Analyses | |
| | 8.2. | Safety Analyses | |
| | 0.2. | 8.2.1. Overview of Planned Analyses | |
| | 8.3. | Pharmacokinetic Analyses | |
| | 0.0. | 8.3.1. Overview of Planned Pharmacokinetic Analyses | |
| | | 8.3.2. Drug Concentration Measures | |
| | | 8.3.3. Pharmacokinetic Parameters | |
| | | 8.3.3.1. Deriving Pharmacokinetic Parameters | |
| | | 8.3.3.2. Statistical Analysis of Pharmacokinetic | |
| | | Parameters | 37 |
| | 8.4. | Pharmacodynamic (Biomarker) Analyses | 38 |

# CONFIDENTIAL

TFR116341

| | | 8.4.1. | Overview of Planned Pharmacodynamic (Biomarker) | 0.0 |
|---|---|---|---|---|
| | | 8.4.2. | Analyses | |
| | | | Allalyses | 39 |
| 9. | OTHE | R STATIS | TICAL ANALYSES | 42 |
| | 9.1. | Explorato | ory Statistical Analyses | 42 |
| 10. | REFE | RENCES. | | 43 |
| 4.4 | 4 DDE | IDIOEO | | 4.4 |
| 11. | 11.1. | | | 44 |
| | | | Population | 45 |
| | | 11.1.1. | Exclusions from Per Protocol Populations | 45 |
| | 11.2. | Appendix | c 2: Time & Events | 46 |
| | | 11.2.1. | Protocol Defined Time & Events | 46 |
| | 11.3. | Appendix | 3: Treatment States and Phases | 50 |
| | | 11.3.1. | Treatment Phases | |
| | | 11.3.2. | Treatment States | |
| | | | 11.3.2.1. Treatment States for AE Data | |
| | 11.4. | | 4: Data Display Standards & Handling Conventions | |
| | | 11.4.1. | Study Treatment & Sub-group Display Descriptors | |
| | | 11.4.2. | Baseline Definition & Derivations | |
| | | | 11.4.2.1. Baseline Definitions | 52 |
| | | | 11.4.2.2. Derivations and Handling of Missing Baseline Data | 52 |
| | | 11.4.3. | Reporting Process & Standards | |
| | 11.5. | _ | (5: Derived and Transformed Data | |
| | | 11.5.1. | General | |
| | | 11.5.2. | Study Population | |
| | | 11.5.3. | Safety | |
| | | 11.5.4. | Efficacy | |
| | | 11.5.5. | Pharmacokinetic | |
| | | 11.5.6. | Pharmacodynamic (Biomarker) | 61 |
| | | 11.5.7. | Exploratory Endpoints | 61 |
| | 11.6. | | ে6: Premature Withdrawals & Handling of Missing Data | |
| | | 11.6.1. | Premature Withdrawals | |
| | | 11.6.2. | Handling of Missing Data | |
| | | | 11.6.2.1. Handling of Missing Dates | |
| | | | 11.6.2.2. Handling of Partial Dates | 64 |
| | | | 11.6.2.3. Handling of Missing Data for Statistical | 0.4 |
| | 44 7 | A 11 | Analysis | 64 |
| | 11.7. | | (7: Values of Potential Clinical Importance | |
| | | 11.7.1. | Laboratory Values | |
| | | 11.7.2. | ECG | |
| | 11.8. | 11.7.3. | Vital Signs<br>८ 8: Biomarker Details | |
| | 11.0.<br>11.9. | | र ७: Examination of Covariates, Subgroups & Other Strata | |
| | 11.3. | 11.9.1. | Handling of Covariates, Subgroups & Other Strata | |
| | 11 10 | | c 10: PVPI and EVLW – Supplementary Information | |
| | | | Data derivations to be performed by GSK | |

# CONFIDENTIAL

TFR116341

| | 11.10.2. | Theoretical Underpinning of Transpulmonary | |
|---|---|---|---|
| | | Thermodilution Measurements | 72 |
| 11.11. | Appendix | 11: Model Checking and Diagnostics for Statistical | |
| | Analyses | | 77 |
| | 11.11.1. | Bayesian Analyses (SAS Proc MCMC) | |
| | | 11.11.1.1 Prior Distributions | |
| | | 11.11.1.2. Initial Values | |
| | | 11.11.1.3. Convergence Diagnostics | <mark>7</mark> 9 |
| | | 11.11.1.4. Additional Model Checking (optional at the | |
| | | discretion of the study statistician) | 80 |
| | | 11.11.1.5. Possible corrective actions for non-converging | |
| | | MCMC models | 81 |
| | 11.11.2. | Mixed modelling assumptions (SAS Proc MIXED) | 81 |
| 11.12. | Appendix | 12: Details of Simulation exercise that produced | |
| | operation | al characteristics used in the protocol | 83 |
| | | Simulations supporting interim analysis 2 | 83 |
| | 11.12.2. | Simulations providing operating characteristics of the | |
| | | target sample size (40 per arm) | 91 |
| 11.13. | | : 13: Abbreviations & Trade Marks | 106 |
| | | Abbreviations | |
| | | Trademarks | |
| 11.14. | | : 14: List of Data Displays | |
| | | Data Display Numbering | |
| | 11.14.2. | Mock Example Shell Referencing | 108 |
| | | Deliverable [Priority] | |
| | 11.14.4. | Study Population Tables | 109 |
| | 11.14.5. | Efficacy Tables | 112 |
| | 11.14.6. | Efficacy Figures | 117 |
| | 11.14.7. | Safety Tables | 1 <mark>20</mark> |
| | 11.14.8. | Safety Figures | 125 |
| | 11.14.9. | Pharmacokinetic Tables | 126 |
| | 11.14.10 | .Pharmacokinetic Figures | 128 |
| | 11.14.11 | .Pharmacodynamic (Biomarker) Tables | 130 |
| | 11.14.12 | Pharmacodynamic (Biomarker) Figures | 132 |
| | | Pharmacogenetic Tables | |
| | | ICH Listings | |
| | | Non-ICH Listings | |
| 11.15. | Appendix | 15: Example Mock Shells for Data Displays | 143 |
| 11.15. | 11.14.10<br>11.14.11<br>11.14.12<br>11.14.13<br>11.14.14<br>11.14.15 | Pharmacokinetic Figures | 128<br>130<br>132<br>134<br>135 |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | This RAP details all planned analyses and outputs required for the final Clinical Study Report (CSR) of study GSK2862277 TFR116341. |
| Protocol | This RAP is based on protocol amendment 4 (Dated: 16/FEB/2015) of study GSK2862277 (GSK Document No. : 2014N197251_04 and eCRF Version (1). |
| Primary<br>Objective | To evaluate whether a single nebulised dose of GSK2862277 prevents peri-<br>operative lung injury compared to placebo, as assessed by measurement of<br>pulmonary vascular permeability (PVPI). |
| Primary<br>Endpoint | Baseline adjusted change in PVPI on completion of surgery |
| Study<br>Design | A Placebo Controlled, Double-blind, Multi-centre, Single Dose, Parallel Group,<br>Randomised Clinical Trial of GSK2862277 in Patients undergoing<br>Oesophagectomy Surgery |
| | • No formal sample size calculations were performed, however, the number of patients is based on computer simulations of baseline adjusted change in PVPI and PaO2/FiO2 on completion of surgery outcomes. Posterior probabilities of each outcome are assessed in combination against chosen threshold criteria to determine the likelihood of success/failure of the study to detect true treatment differences. A sample size of 40 subjects p.a. has an equivalent of a Type I error rate of 4.65% and a probability of 80.64% of detecting plausible effect sizes. A sufficient number of subjects will be enrolled such that 80 subjects complete dosing and assessments. |
| | Patients enrolled in the study will be scheduled to undergo planned/elective trans-thoracic surgery for oesophagectomy. Prior to surgery patients will receive a single nebulised dose of GSK2862277 or placebo. |
| | • A factorial treatment structure is used in the randomisation (Treatment and the lung which BAL is sampled from, both two level factors). Summary tables of the raw/observed data will be produced with all possible groupings (See Section 11.4.1). Although each statistical model will contain adequate terms to account for the full factorial treatment structure the majority of statistical analyses for non BAL related endpoints will implicitly assume that the Treatment by BAL interaction is negligible and present results as treatment comparisons averaged over the levels of the BAL factor; without formally testing for it (mainly due to the small sample size). Informal checking of this assumption may consist of examining the posterior distribution for the interaction term and visually assessing whether it is non zero. If this is deemed to have occurred the corresponding summary tables and analysis outputs will be modified. For BAL related endpoints the starting assumption for summary tables and statistical modelling will be the interaction term is present, but outputs may be modified if the interaction is subsequently deemed negligible. |
| | Due to the nature of the endpoints in this study (e.g. the invasive medical procedures needed to obtain PVPI) it is often not practical/ethical to schedule |

| Overview | Key Elements of the RAP |
|---|---|
| | true baseline samples (pre-randomisation / pre-dose). However, in mitigation, it should be noted that the surgical procedure is expected to be the principal factor driving changes in many of these study endpoints (e.g. PVPI and PaO2/FiO2) and the scheduled baseline is measured before the surgical intervention. Therefore, potential interpretational difficulties (e.g. attributing causality: chance result or real treatment effect acting over the dose to baseline time period) should large differences between baseline values on the treatment arms are acknowledged but accepted (this is an exploratory and not confirmatory study). If the observed difference between treatments at baseline is deemed to be large / clinically important appropriate sensitivity analyses may be performed (for example, but not limited to, omitting the baseline term from the corresponding statistical model). |
| Planned | Interim analyses are detailed within Section 3.1 where applicable. |
| Analyses | <ul> <li>All decisions regarding final analysis, as defined in this RAP document, will be<br/>made prior to Database Freeze of the study data.</li> </ul> |
| Analysis<br>Populations | The 'Safety Population' will be used to evaluate study population andsafety and 'PK' population to evaluate pharmacokinetics. |
| | <ul> <li>Per protocol populations have been defined that exclude "open and shut"<br/>cases; and will be used as part of efficacy and PD/Biomarkers analyses.</li> </ul> |
| Hypothesis | <ul> <li>The study was designed to estimate the effect of a single nebulised 26 mg dose<br/>of GSK2862277 relative to placebo on primary and secondary efficacy<br/>endpoints.</li> </ul> |
| | <ul> <li>No formal statistical hypothesis tests will be conducted; instead an estimation<br/>approach will be undertaken.</li> </ul> |
| Primary<br>Analyses | <ul> <li>The protocol proposed an end of study decision pathway, consisting of the<br/>primary endpoint and PaO2/FiO2 on completion of surgery (adjusting for the<br/>baseline values of each endpoint)</li> </ul> |
| | <ul> <li>Evaluation of this decision pathway via joint modelling of the 2x endpoints<br/>constitutes the primary analysis.</li> </ul> |
| | <ul> <li>The primary analysis utilises a Bayesian framework with Monte Carlo Markov<br/>Chain (MCMC) sampling techniques. The decision pathway will be evaluated<br/>via posterior distributions of appropriate combinations of the model parameters.</li> </ul> |
| | <ul> <li>The decision pathway is not binding upon GSK but provides an a priori<br/>yardstick to measure the success of the trial against.</li> </ul> |
| | Note: The marginal distribution of baseline adjusted PVPI on completion of surgery is obtained as part of the steps to evaluate the decision grid (hence this primary analysis does cover the primary objective/endpoint stated in the protocol). |
| Secondary<br>Analyses | Baseline adjusted change in PVPI on completion of surgery: Bayesian ANCOVA model(s) with baseline and centre as fixed effects with covariate exploration / model building activities (e.g. duration of surgery and duration of one lung ventilation as plausible continuous covariates). Acts as confirmation |

| Overview | Key Elements of the RAP |
|---|---|
| | that the marginal distribution from the Primary analysis is appropriate. |
| | Baseline adjusted change in extravascular lung water index (EVLWI) and baseline adjusted change in PaO2/FiO2, on completion of surgery will be analysed in a similar manner to the Secondary Analysis of PVPI (single time point analysis), described above. |
| | Bayesian repeated measures analysis of post-operative PVPI, EVLWI and PaO2/FiO2 (separate model for each endpoint; assuming a mixed effects model structure). Baseline adjusted medians and 95% credible intervals will be constructed for the differences/ratios between GSK2862277 26 mg and Placebo at each of the post-operative time points. |
| | <ul> <li>Safety data will be presented in tabular format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards.</li> <li>Incidence and titres of serum anti-GSK2862277 antibodies post dosing will be summarised by treatment and listed by subject</li> </ul> |
| | <ul> <li>Individual GSK2862277 plasma concentration-time profiles and median/mean (±SD) profiles will be plotted and listed. Derived PK parameters will be summarised and listed. BAL fluid and plasma urea data, along with the derived Dilution Factor will be summarised and listed. BAL fluid concentrations of GSK2862277, the volume of ELF in BAL fluid and pooled ELF concentration of GSK2862277 will be summarised and graphically presented. No formal statistical analyses will be conducted.</li> </ul> |
| | Biomarkers in BAL will be analysed in a Bayesian framework assuming a mixed effects model structure. Summary statistics from derived posterior probability distributions (such as treatment medians and 95% credible intervals) will be constructed for the differences/ratios between GSK286227 26 mg and Placebo at each time point (and possibly within each BAL sampling location too). |
| Exploratory<br>Analyses | Daily SOFA scores will be analysed using Bayesian repeated measures analyses. Adjusted medians and 95% credible intervals will be presented in tables and graphically for each treatment by day, together with estimated treatment differences GSK2862277 26 mg – Placebo and the corresponding 95% credible intervals. Note: Strong assumptions will be made to predict a baseline SOFA score for each subject to evaluate change from baseline SOFA (exploratory) |
| | Blood/Cellular Biomarkers will be analysed in a similar fashion to the BAL biomarkers. |
| | Other clinical parameters would be summarised by treatment and listed by subject. Statistical modelling would be conditional on the observed data. |

# 1.1. RAP Amendments

Revision chronology:

| RAP Section(s) | Amendment details |
|---|---|
| Reporting and Analysis Plan Final [10-JUL-2015] | |
| Reporting and Analysis | Plan Final Amendment 1 [17-NOV-2015] – Pre unblinding for IA1 |
| Cover Page | Indicated RAP contains amended text |
| 1 | Clarified Analysis Populations for Efficacy PD/Biomarkers will be Per protocol (i.e. will not include "Open and Shut" cases) |
| 1.1 | Added Revision Chronology Table |
| 3.1.2 | Clarified IA2 will use mixture of Safety and Per protocol populations |
| 7.1.1 & 8.1.1 | Clarified Per Protocol 2 population to be used instead of Safety |
| 8.4.1 | Clarified Per Protocol 2 population to be used instead of Safety, except for BAL related outputs where Per Protocol 1 population is required |
| 8.4.1 Table 8 | Updated List of Planned Biomarkers to reflect current plans at time of RAP amendment 1 |
| 11.1.1 | Clarified that an upcoming eCRF version will have a variable indicating if a subject was an "open and shut case" and manual programming may be required to implement the populations if this variable is not retrospectively populated for existing subjects. |
| 11.6.2.1 | Added section for missing date/times for surgical procedures and biomarker samples to account for known missing data for subject PPD (known at time RAP amendment #1 written). |

| RAP Section(s) | Amendment details |
|---|---|
| , , | Plan Final [10-JUL-2015] |
| | Plan Final Amendment 1 [17-NOV-2015] – Pre unblinding for IA1 |
| 11.7.1 | Based upon medical monitor advice: |
| | Corrected Low Flag value for Hemoglobin (Males and Females) because it was specified in g/dL and not g/L |
| | Changed PR interval Lower and Upper PCI values |
| | Change from Baseline "Increase from Baseline QTc": Moved the range from the Lower to the Upper column (leaving Lower column blank) |
| | Re-drew the Vital Sign Parameter (Change from<br>Baseline) tables to only have one entry for Decreases<br>and Increases respectively |
| 11.8 | Updated List of Planned Biomarkers to reflect current plans at time of RAP amendment 1 |
| 11.14 | Amended populations for efficacy/Biomarker related outputs and corrected typos in timing/priority (e.g. "IA [2]" corrected to "IA2 [1]") |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the substance of the originally planned primary statistical analysis specified in the protocol / protocol amendment 4 (Dated: 16/FEB/2015). Clarification of how the four level treatment structure is incorporated into the decision grid and a mechanism to adjust for other covariates such as centre have been included in this RAP.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate whether a single<br>nebulised dose of GSK2862277<br>prevents peri-operative lung injury<br>compared to placebo, as assessed<br>by measurement of pulmonary<br>vascular permeability. | Baseline adjusted change in PVPI on completion of surgery |
| Secondary Objectives | Secondary Endpoints |
| To evaluate whether a single<br>nebulised dose of GSK2862277<br>prevents peri-operative lung injury<br>compared to placebo, as assessed by<br>measurement of pulmonary oedema. | Baseline adjusted change in EVLWI on completion of surgery. |
| To evaluate the safety and tolerability<br>of GSK2862277 administered<br>preoperatively | <ul> <li>AEs</li> <li>Clinical laboratory safety data.</li> <li>ECG readings</li> <li>Vital signs</li> </ul> |
| To evaluate whether a single nebulised dose of GSK2862277 prevents peri-operative lung injury compared to placebo, as assessed by degree of hypoxaemia | Baseline adjusted change in PaO2/FiO2 on completion of surgery |
| To evaluate differences in expression<br>profile of BAL biomarkers from both<br>ventilated and collapsed lungs<br>immediately after surgery | Levels of BAL biomarkers (e.g. IL-6, sRAGE, protein levels) on completion of surgery. |
| To evaluate the effect of a single IH dose of GSK2862277 compared to placebo, on attenuating lung and distal organ injury over the post-operative period | <ul> <li>Change over time in PaO2/FiO2 post-operatively on Day 2 through to Day 4 (as available; SpO2/FiO2 when arterial line removed)</li> <li>Change over time in PVPI and EVLWI post-operatively on Day 2 through to Day 4</li> <li>Daily SOFA scores on Day 2 through to Day 4</li> </ul> |
| To describe plasma pharmacokinetics<br>of a single inhaled dose of<br>GSK2862277. | Plasma concentrations of GSK2862277 and derived pharmacokinetic parameters. |
| To quantify the concentration of | BAL concentrations of GSK2862277 and derived |

| Objectives | Endpoints |
|---|---|
| GSK2862277 in BAL and to compare to plasma levels of GSK2862277 | pharmacokinetic parameters Ratio of BAL concentration to plasma concentration. |
| To evaluate the levels and specificity<br>of any anti-drug antibodies formed<br>following dosing with GSK2862277. | Incidence and titers of serum anti-GSK2862277 antibodies post dosing |
| Exploratory Objectives | Exploratory Endpoints |
| To evaluate the effect of GSK2862277 compared to placebo on clinical and patient outcomes. | <ul> <li>Further exploratory evaluation of effectiveness may be conducted where data permit. Endpoints may include, but are not limited to:</li> <li>Diagnosis of ARDS out to day 28;</li> <li>28 day survival;</li> <li>Ventilator Free Days; ICU &amp; hospital length of stay;</li> <li>Organ Failure Free Days;</li> <li>Haemodynamic assessments (e.g. Cardiac Index, Global End Diastolic Volume, etc)</li> <li>Oxygenation Index</li> </ul> |
| To evaluate changes in TNFR related<br>and disease biology biomarkers in the<br>blood of patients who have been<br>treated with GSK286227 compared to<br>placebo, on completion of surgery and<br>in the immediate post-operative<br>period. | Difference from placebo in levels of plasma biomarkers<br>(e.g. IL-6, sRAGE) on completion of surgery and through<br>to Day 4 |

# 2.3. Study Design



# 2.4. Statistical Hypotheses

## **Precision Estimation**

No formal statistical hypotheses will be tested in this study. Safety related objectives will be assessed via summary tables, listings and figures.

In addition to summary tables, listings and figures, study objectives relating to efficacy (for example, lung physiology and biomarkers) may be evaluated using posterior distribution(s) for the

effect of GSK2862277 relative to Placebo. Point estimates and corresponding 95% credible intervals will be constructed for the difference between the mean of the test treatment and the mean of the reference treatment,  $\mu(\text{test})$  -  $\mu(\text{reference})$ . No adjustment for multiplicity will be performed due to the Bayesian analysis framework.

**Note:** If data require log transformation prior to analysis then point estimates and corresponding 95% credible intervals will be constructed for the ratio of test treatment to placebo treatment  $\mu$  (test) /  $\mu$  (reference) in place of those for differences in means.

## 3. PLANNED ANALYSES

# 3.1. Interim Analyses

There are two interim analyses planned for this study both of which will use unblinded data (an unblinded sample size re-estimation will be performed as part of interim analysis #2). Further details are given in Section 3.1.1 and Section 3.1.2. The interim analyses will be performed by the study statistician (or designate). The appropriate internal GSK procedures will be followed to ensure that access to unblinded subject level data is restricted to the specific study team members who require access.

# 3.1.1. Interim analysis #1: Unblinded safety review after approx 10 patients have completed Day 7 visit; roughly 5 per study drug arm.

The principal objective will be to determine whether there are any emerging safety trends/ signals which might require modifications to be made and/or suspension of recruitment pending further data review. Unless there are safety concerns recruitment into the study may continue whilst interim analysis #1 (IA1) is being performed. IA1 will use the "Safety" population applicable at the time of the data cut.

The following safety outputs will be provided:

- Demographic information
- AE/SAEs
- Laboratory data
- Vital signs
- ECG data
- Concomitant medications
- Listing of surgical procedure information for each subject

For further details of the output see Appendix 14.

Note: An additional informal check of the available plasma PK values may be made to give confidence dosing is occurring as intended. Samples will be batched and sent for analysis at designated intervals during the study and the results made available (batches will be timed to coincide with the interim analyses). The check would be basic; namely confirming subjects on active doses of GSK2862277 with available plasma PK concentrations at the time of the interim had at least one quantifiable post dose value of GSK2862277. No outputs will be reported from this step and the timing of the interim analyses will not be delayed on account of this. Appropriate

remedial action(s) would be taken if this check revealed potential problems with the dosing (for example, but not limited to, re-training of selected sites on the use of the equipment, or processing all the collected PK samples with formal PK and/or PK/PD modelling with a view to a dose adjustment – details would be documented in any associated protocol amendment and/or the CSR).

# 3.1.2. Interim analysis #2: Unblinded safety review, futility analysis and sample size re-estimation after approx 40 patients have completed Day 7 visit; roughly 20 per study drug arm.

A "soft lock" of the database for those subjects in scope for interim analysis #2 (IA2) is planned. This should ensure the IA2 eCRF data are as clean as possible and that data for the potential analyses in Figure 1 are available in a reasonable timeframe. IA2 will use a mixture of the "Safety" and "Per Protocol" populations applicable at the time of the data cut.

In addition a Sample size re-estimation will take place at IA2 to determine if the overall target sample size should remain at 80 subjects (~40 p.a.).

The outcome of interim analysis #2 will be communicated by GSK to the sites as either "Continue" or "Pause and Review".

Upon a "Pause and Review" communication the available data will be reviewed by the study team (un-blinded) and additional data may be requested from the sites to determine whether to:

- Stop the study early for futility
- Modify aspects of its design
- Resume and continue unaltered

Figure 1 indicates the flow of additional data to be reviewed upon a "Pause and Review" outcome and possible actions; although it should be stressed that Figure 1 is non-binding. Emerging patterns in the data may suggest other analyses not described here that may influence the action taken.

Although interim analysis #2 is scheduled to occur after approximately 20 patients p.a. have available data up to Day 7, it is possible that recruitment rates may be lower than anticipated in which case the interim analysis may occur after a fixed time with whatever data are available.

The futility analysis component of Interim analysis #2 will use the baseline adjusted endpoints on completion of surgery:

- PVPI Ratio: Mean Active/Mean Placebo,
- P to F Ratio Difference: Mean Active Mean Placebo

and will utilise predictive inference, decision pathway and confidence thresholds.

The interim analysis will assume that there is no interaction between study drug (active and placebo) and the location of the BAL lung sampling (collapsed or ventilated). Therefore the 4 treatments will be combined to two treatments (based on study drug) and

references to treatment arms in this section assume usage of Alternative Treatment descriptors #1 (See Section 11.4.1). The algorithm suggested in Section 9.3.1 of the protocol has been modified to allow adjustments for other covariates.

The algorithm for the interim analysis is as follows:

- 1. Apply any transformations to the endpoint(s) (and baseline(s)) and center any continuous covariates.
- 2. Fit a model similar in form to that described in Section 7.1.2 to the observed IA2 data. Note: Should use separate variance covariance matrices (one per treatment arm).
- 3. The equivalent of adjusted least square means will be constructed for each endpoint on each treatment arm.
- 4. Once MCMC model convergence has been achieved the current iteration's values for the variance covariance matrix and the adjusted least square mean vector define a multivariate normal distribution for a future subjects data (a separate distribution per treatment arm)
- 5. Use the newly defined multivariate normal distributions to simulate enough subjects to achieve an overall total of 40 per arm
- 6. Repeat steps 4 & 5 1000 times (i.e. 1,000 samples once the MCMC model has converged).
- 7. For each treatment arm, use the median values of the adjusted least square means and the median values of each element of the variance covariance matrix to derive the hyperparameters of the Normal-Inverse-Wishart distribution for each treatment (i.e. constructed using the model **adjusted** IA2 immediately post surgical values rather than being derived directly from the raw/observed data) see Table 14 for how to obtain these parameters.
- 8. Derive Multivariate sample statistics from each simulated dataset (see Section 11.12.1 for the list of sample statistics to derive). The sample statistics will be used to update the parameters of the Normal-Inverse-Wishart distribution for each treatment (see Table 15).
- 9. Use the updated Normal-Inverse-Wishart distributions to estimate the end of study mean treatment effects (i.e. condition on the Expected value of the VCV) and then determine the parameters describing the distribution of the mean end of study treatment difference (See Section 11.12.1).
- 10. Determine whether the probability of observing ANY decrease in PaO2/FiO2 means and Any increase in PVPI means is greater than 0.1
- 11. If so then record that simulated study as being futile
- 12. Repeat steps 8 to 10 1000 times
- 13. Determine the proportion of the 1000 simulated studies which meet the futility threshold
- 14. If the proportion is larger than 0.3 then the recommendation is to "Pause and Review", otherwise the recommendation is to "Continue"

| Interim | Details |
|---|---|
| Analysis #2 | |
| Additional details on the Method | <ul> <li>PVPI and P<sub>a</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> on completion of surgery</li> <li>Baseline: PVPI and P<sub>a</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> immediately prior to surgery (day 1)</li> <li>Any transformation of a response variable is also expected to be applied to the corresponding baseline variable. Final decisions on transformations will be based on the observed data and model diagnostics (PVPI is expected to require a Ln (natural logarithm) transformation)</li> <li>Any observations with missing model covariates (e.g. baseline) would be excluded from the model fitting process (i.e. also excluding the record from any centering of covariates)</li> </ul> |
| | <ul> <li>The above endpoints and baselines will be the average of any replicates available at the planned time points</li> <li>The model specifications described in Section 7.1.2 (primary analysis) will also apply to the model fitted to the observed set of IA2 data where applicable. Exceptions include only using the burn in and thinning parameters to achieve MCMC model convergence (the number of posterior draws will be limited to 1,000 to match the required number of future simulated study outcomes). In addition the IA2 model does not require directly fitting 4 separate treatment parameters. Therefore the following is an example construction for the adjusted least square equivalent Ln{PVPI}</li> <li>μ̂<sub>Pbo,PVPI</sub> + (**eenters* / #Centers*)</li> </ul> |
| Output | <ul> <li>By subject time profiles of PVPI and PaO2/FiO2 grouped by treatment will be produced using the available IA2 data.</li> <li>Scatterplots of the observed IA2 data from each subjects will be produced (grouped by treatment and IA2 timepoint)</li> <li>Descriptive statistics for absolute and change from baseline PVPI and PaO2/FiO2 grouped by treatment will be tabulated.</li> <li>A set of summary text describing the IA2 process and recommendation will be produced. Note: In addition the full output from SAS PROC MCMC will be produced for statisticians to assess the suitability of the model but this is not expected to be disseminated further due to its technical nature.</li> </ul> |
| Pause and<br>Review | <ul> <li>In the event of a "Pause and Review" recommendation the analyses described in Figure 1 may be attempted in the order described therein.</li> <li>Analyses in Figure 1 are expected to be the same as their respective end of study analyses (e.g. analyses involving BAL will account for the BAL lung sampled in the statistical modelling and if necessary compare active to placebo within each of those strata).</li> <li>No formal decision criteria for Figure 1 are specified here. The results of the analyses described in Figure 1 will be used to inform the decision to "Continue", "Modify" or "Stop" in discussions with the study team. Additional analyses may be performed if appropriate and documented in the CPSR.</li> </ul> |
| Sample Size<br>Restimation | The adjusted sample size (total number of subjects) will be determined by the clinical study team after reviewing the outcome of the following exercise. It is |

| Interim<br>Analysis #2 | Details |
|---|---|
| | expected to be the smallest value from either the current upper limit (80) or the re-estimated value (i.e. it is expected to remain capped at 80 subjects). There is no minimum limit, so it is therefore possible that the re-estimated sample size chosen by the clinical study team is the same value as the observed number of IA2 subjects, and hence the study will cease recruiting new subjects. • The re-estimation will use the median estimates of each of the elements in the VCV matrix obtained from the (adjusted) modelling of the observed IA2 data. It will use the similar methodology to the protocol (see Section 11.12.2 for details of the simulation process), except that total sample size will be varied until the resulting operating characteristics for the "Overall success outcome" using the "Null" and "Minimum desired profile" scenarios match the ones obtained for a total sample size of 80 (roughly 4.65% and 80.64% respectively). If the point estimates for the variances from the observed IA2 data are larger than the assumed values used in the protocol then the procedure will start at 80 subjects and increase by 2 subjects until the criteria are met, and conversely if the observed variances are smaller the process will start at 80 subjects and decrease by 2 subjects until the criteria are met. Note: Larger increments may also be used to arrive in the "ball park" more quickly (e.g. 6, 10 or 20 subject increments) |

Figure 1 Flow chart of additional data and questions in the event of IA2 Pause and Review outcome (non-exhaustive list)



# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

# 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screen Failures | <ul> <li>Comprise all subjects who enrolled but are recorded as screen failures</li> </ul> | Screen Failures |
| Safety | <ul> <li>Comprise of all subjects who receive at least one complete dose of study treatment.</li> <li>This population will be based on the treatment the subject actually received.</li> </ul> | <ul><li>Study Population</li><li>Safety</li><li>Efficacy</li></ul> |
| Pharmacokinetic<br>(PK) | <ul> <li>Subjects in the 'Safety' population for whom<br/>a pharmacokinetic sample (plasma and/or<br/>BAL) was obtained and analysed.</li> </ul> | • PK |
| Per Protocol 1<br>(PP1) | Subjects in the 'Safety' population for whom<br>the treatment actually received was the same<br>one they were randomised to ( <b>both</b> study<br>drug and BAL sampling location) | Efficacy |
| | <ul> <li>Met the protocol defined inclusion/exclusion<br/>criteria (if criteria are changed during course<br/>of study apply the set applicable at the time<br/>of their enrolment)</li> </ul> | |
| | <ul> <li>Not an "open and shut" (inoperable) surgical case</li> </ul> | |
| Per Protocol 2<br>(PP2) | Subjects in the 'Safety' population for whom<br>the study drug actually received was the<br>same one they were randomised to (study<br>drug) | Efficacy |
| | <ul> <li>Met the protocol defined inclusion/exclusion<br/>criteria (if criteria are changed during course<br/>of study apply the set applicable at the time<br/>of their enrolment)</li> </ul> | |
| | Not an "open and shut" (inoperable) surgical case | |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Per Protocol 3 (PP3) | Subjects in the 'Safety' population for whom<br>the BAL lung actually sampled was the same<br>one they were randomised to | Efficacy |
| | Met the protocol defined inclusion/exclusion<br>criteria (if criteria are changed during course<br>of study apply the set applicable at the time<br>of their enrolment) | |
| | Not an "open and shut" (inoperable) surgical case | |
| Interim Analysis 1 (IA1)* | Subjects in the 'Safety' population at the time of the Interim Analysis 1 data cut | Outputs detailing population membership |
| Interim Analysis 2 (IA2)* | Subjects in the 'Safety' population at the time of the Interim Analysis 2 data cut | Outputs detailing population membership |

#### NOTES:

- Please refer to Appendix 1: List of Data Displays which details the population to be used for each displays being generated.
- \*= Population will only be produced to support the end of study reporting. Outputs required to support each of the interim analyses will use the applicable population at the time of the respective interim analysis data cut.

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - o For subjects involved in the interim analyses every effort will be made to review the (uncleaned) data from those subjects prior to unblinding those individuals. However given the interim database(s) may not be frozen these in-stream decisions may be revised if new information becomes apparent. Any such revision, and justification if necessary, would be noted in the study file.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 11.2 | Appendix 2: Time & Events |
| 11.3 | Appendix 3: Treatment States and Phases |
| 11.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 11.5 | Appendix 5: Derived and Transformed Data |
| 11.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| 11.7 | Appendix 7: Values of Potential Clinical Importance |
| 11.8 | Appendix 8: Biomarker Details |
| 11.9 | Appendix 9: Examination of Covariates, Subgroups & Other Strata |
| 11.10 | Appendix 10: PVPI and EVLW – Supplementary Information |
| 11.11 | Appendix 11: Model Checking and Diagnostics for Statistical Analyses. |
| 11.12 | Appendix 12: Details of Simulation exercise that produced operational characteristics used in the protocol |
| 11.13 | Appendix 13: Abbreviations & Trade Marks |
| 11.14 | Appendix 14: List of Data Displays |
| 11.15 | Appendix 15: Example Mock Shells for Data Displays |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the "Safety" population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Display Type | Data | Displays Gene | rated |
|---|---|---|---|
| | Table | Figure | Listing |
| Randomisation | | <u> </u> | |
| Randomisation | | | Y |
| Blind broken (excluding when part of interim analyses) | | | Y |
| Subject Accountability | | | |
| Study Population membership | Y | | Y |
| Subject Disposition | | | |
| Disposition | Υ | | |
| Reasons for Screening Failures | Υ | | Y |
| Reasons for Withdrawals | | | Y |
| Important Protocol Deviations | Υ | | Y |
| Inclusion and Exclusion Criteria Deviations | | | Y |
| Demography | | | |
| Demographic Characteristics | Υ | | Y |
| Race & Racial Combinations | Υ | | Y |
| European Medicines Agency: Summaries for the European | Υ | | |
| Clinical Trials Database (EudraCT) | Ī | | |
| Medical Condition & Concomitant Medications | | | |
| Concomitant Medication | Υ | | Υ |
| Medical Conditions (Current and Past) | <b>Y</b> 1 | | Y |
| Exposure | | | |
| Exposure | | | Y |

#### NOTES:

- Y = Yes display generated.
- 1 = Summarise Current and Past conditions in separate tables

# 7. PRIMARY STATISTICAL ANALYSES

# 7.1. Efficacy Analyses

# 7.1.1. Overview of Planned Efficacy Analyses

Further details regarding Transpulmonary Thermodilution (TPTD) measurements are provided in Appendix 10: PVPI and EVLW – Supplementary Information.

The primary efficacy analyses will be based on the "Per Protocol 2" population, unless otherwise specified.

Table 3 provides an overview of the planned efficacy analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 3 Overview of Planned Efficacy Analyses

| Endpoint / | | | Α | bsolu | te | | Change from Baseline | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | Stat | Stats Analysis | | Summary | | Individual | | Stats Analysis | | | Summary | | Individual | |
| Туре | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Transpulmonary Therm | odilu | tion | | | | | | | | | | | | |
| PVPI | | | | Υ | Υ | Υ | Y1. | | | | Υ | | | Y1. |
| $P_aO_2/F_iO_2$ | | | | Υ | Υ | Υ | Y1 | | | | Υ | | | Y1. |
| Joint Modelling of | Υ | Υ | Υ | | Υ | | | | | | | | | |
| PVPI and P <sub>a</sub> O <sub>2</sub> /F <sub>i</sub> O <sub>2</sub> | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Natural logarithms of the observed response will be performed if it is deemed appropriate prior to modelling. If
   Natural logarithms are used results will be back-transformed for display purposes.
- 1. Listing should also flag any discrepancies between the eCRF supplied PVPI and any in-house GSK re-derivations.

Figure 2 shows the proposed End of Study Decision Pathway based on joint modelling of PVPI and P<sub>a</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub>.

In crude terms decreases in PVPI and increases in  $P_aO_2/F_iO_2$  (relative to the changes seen on the placebo arm) are the desired outcomes for the study drug.

Figure 2 End of Study Decision Pathway



Note: In Figure 2 statements such as " $\leq 11.6\% \downarrow$ " translate as "the decrease (active relative to placebo) is **less** than 11.6%; i.e. when the ratio of the treatment means (Act/Pbo) is **greater** than 0.884". The implication being that there is a 75% chance or more that study drug hasn't decreased PVPI enough and the outcome is "Potentially Unsuccessful".

The posterior probability of each Figure 2 outcome will be derived and, if it exceeds its respective confidence level, that outcome will be deemed to have occurred. Combinations of occurring outcomes imply the following four end of study states:

| Overall success | ≥1 of the "Success" outcomes | AND | 0 "Failures" |
|---|---|---|---|
| <b>Potentially Unsuccessful</b> | 0 "Success" outcomes | AND | 1 "Failure" |
| Inconclusive | 0 "Success" outcomes | AND | 0 "Failures" |
| Inconsistent | ≥1 of the "Success" outcomes | AND | 1 "Failure" |

Note: The primary analysis will only use the pre-op and immediate post op values of PVPI and P<sub>a</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub>. Secondary analysis (a repeated measures version of the joint modelling) may also include the same set of timepoints and comparisons, but because the estimates across multiple timepoints may be correlated there may be minor differences in the results from the Primary and Secondary analysis models. In such a scenario the primary analysis model will take precedence. Only if the study statistician deems any

discrepancies to be large enough to be of concern will further discussion and/or comment be added to the CSR.

# 7.1.2. Planned Efficacy Statistical Analyses

# **Primary Statistical Analyses**

## Endpoint(s)

- PVPI and P<sub>a</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> on completion of surgery
- Baseline: PVPI and P<sub>a</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> immediately prior to surgery (day 1)
- Any transformation of a response variable is also expected to be applied to the corresponding baseline variable. Final decisions on transformations will be based on the observed data and model diagnostics (PVPI is expected to require a Ln (natural logarithm) transformation)
- Any observations with missing model covariates (e.g. baseline) would be excluded from the model fitting process (i.e. also excluding the record from any centering of covariates)
- The above endpoints and baselines will be the average of any replicates available at the planned time points

# Model Specification

- The (transformed) endpoints will be assumed to follow a multivariate normal distribution. Linear predictors will be derived for each subject (i.e. obtain a vector of means for the MVN distribution). Each treatment arm will also have a separate variance covariance matrix.
- The linear predictors will consist of mean vectors to capture the effect of treatment for each endpoint and a variety of other model terms (an example is given at the end of this text).
- Main Treatment Descriptors to be used (i.e. 4 levels of the treatment term)
- No intercept terms should be fitted for either endpoint (due to fitting all 4 levels of treatment).
- Baseline vectors will be fitted as continuous covariates (baseline values should be centered prior to inclusion in the model, centering to occur after any transformation of the individual subjects responses).
- Categorical fixed effect vectors should be added for Center by Endpoint (if recruitment is such
  that center terms are poorly estimated then appropriate action will be taken, including but not
  limited to, pooling of centers or removal of the term from the model).
- Non-informative priors will be utilized for each model parameter assigned either as a normal distribution centered on 0 with large variance 1E6 or as appropriate to the parameters distribution.
- The prior for the variance covariance matrices  $\Sigma_{Pbo}$  and  $\Sigma_{Act}$  will be an inverse Wishart distribution (separate VCVs are not required for the BAL factor levels).
- SAS PROC MCMC will be used to combine the non-informative priors with the data observed
  to obtain sufficient draws from the posterior distribution (after any thinning) such that the
  MCSE/SD values for parameters of interest are less than 0.01 (anticipated to be in the region
  of ~100,000 draws). If model convergence is poor then alternative initial parameter values
  should be considered.
- The randomization seed used in PROC MCMC should itself be generated with an element of randomness but there is no need to formally document this process (e.g. using Excel function RANDBETWEEN [1,9999999] and copying the result into the SAS code)
- Combinations of the fitted model parameters will be used to answer the clinically relevant questions.

# **Primary Statistical Analyses**

Median values of the baseline adjusted response for each endpoint and their associated 95% credible intervals (equi-tailed) will be produced from the posterior distributions obtained via appropriate combinations of the fitted model parameters; akin to lease square means (e.g.

Adjusted Pbo PVPI averaging over BAL = 
$$\frac{\hat{\mu}_{PC,PVPI} + \hat{\mu}_{PV,PVPI}}{2} + \left(\sum_{i=1}^{\#centers} Center_i / \#Centers\right).$$

- The joint (bivariate) posterior probability distribution of the endpoints (averaging over BAL) will be obtained for the comparison(s) implied in Figure 2 by appropriate combinations of the fitted model parameters. The marginal posterior distributions for the comparisons for each endpoint will also be obtained from this joint posterior sample and be used to construct medians and 95% equi-tail credible intervals for individual endpoints.
- Flag variables (taking binary values of 1 or 0) will be created to evaluate the steps in the end of study decision pathway for each simulated draw from the joint posterior distribution (Figure 2). The mean of each flag variable over the MCMC iterations is the estimate of the desired probability, and should be used to assess which study outcome has been observed. These flag variables (and constrained variables) may cause SAS to issue warning or error messages to the log due to their binary nature, especially if the result is clear cut and their value rarely changes (such warnings/errors should be reviewed but may be safely discounted)
- In addition posterior probabilities of the differences (or ratios) for other cut-points (which may be determined upon inspection of the data, or from developing business requirements), may also be computed.
- Where applicable estimates would be derived at the means of any model covariates, akin to
  least squares means in PROC MIXED, and back transformed if necessary. When covariates
  are centered before the model fitting their mean is zero so the covariate can be dropped from
  the derivation.

The following describes the anticipated linear predictor for an hypothetical subject from center 3, on active treatment, with BAL sampled from the collapsed lung and centered baseline values of -4.1 and -0.5 for P/F and PVPI respectively (note: additional covariates may be explored and added based on the observed data).

# **Primary Statistical Analyses**

$$\begin{bmatrix} \hat{y}_{1} & \hat{y}_{2} \\ \hat{y}_{1} & \hat{y}_{2} \end{bmatrix} = \begin{bmatrix} -4.1 & 0.5 \\ 0 & \hat{B}S_{PVFI} \end{bmatrix} + \begin{bmatrix} Center_{1,P/F} & Center_{1,PVFI} \\ Center_{2,P/F} & Center_{2,PVFI} \\ Center_{3,P/F} & Center_{3,PVFI} \\ Center_{4,P/F} & Center_{4,PVFI} \\ Center_{5,P/F} & Center_{5,PVFI} \end{bmatrix} + \begin{bmatrix} I(Pho, Collapsed) * [\hat{\mu}_{PO, PVFI} & \hat{\mu}_{PO, PVFI}] + I(Pho, PVFI) + I(Pho,$$

$$I(Pbo,Collapsed)*[\hat{\mu}_{PC,P/F} \quad \hat{\mu}_{PC,PVPI}] + I(Pbo,Ventilated)*[\hat{\mu}_{PV,P/F} \quad \hat{\mu}_{PV,PVPI}] + I(Act,Collapsed)*[\hat{\mu}_{AC,P/F} \quad \hat{\mu}_{AC,PVPI}] + I(Act,Ventilated)*[\hat{\mu}_{AV,P/F} \quad \hat{\mu}_{AV,PVPI}]$$

Where

 $Center_5$  term(s) constrained to be zero and  $I(\bullet)$  is an Indicator function with value 1 if condition met and zero otherwise [Here I(Pbo, Collapsed), I(Pbo, Ventialted), I(Act, Ventilated) = 0, I(Act, Collapsed) = 1,

$$I(C_3) = 1$$
 and  $I(C_1)$ ,  $I(C_2)$ ,  $I(C_4)$  &  $I(C_5) = 0$ 

To link to observed data assume : 
$$\begin{bmatrix} y_{1} & y_{1} \\ y_{1} & y_{2} \end{bmatrix}^{MVN} \sim \left( \begin{bmatrix} y_{1} & y_{1} \\ \hat{y}_{1} & \hat{y}_{2} \end{bmatrix}, [\Sigma_{Act}] \right)$$
 where  $\Sigma_{Pbo}$  &  $\Sigma_{Act}$ 

are 2x2 Variance Covariance matrices for the treatment arms (ignoring the BAL factor) Posterior distributions are enumerated with appropriate combinations

of 
$$\hat{\mu}_{PC,P/F}$$
,  $\hat{\mu}_{PC,PVPI}$ ,  $\hat{\mu}_{PV,P/F}$ ,  $\hat{\mu}_{PV,PVPI}$ ,  $\hat{\mu}_{AC,P/F}$  &  $\hat{\mu}_{AC,PVPI}$ ,  $\hat{\mu}_{AV,P/F}$  &  $\hat{\mu}_{AV,PVPI}$  e.g Sample from Posterior Distn for Diff in Mean P/F averaging over BAL factor =

$$\left(\frac{\hat{\mu}_{AC,P/F} + \hat{\mu}_{AV,P/F}}{2}\right) - \left(\frac{\hat{\mu}_{PC,P/F} + \hat{\mu}_{PV,P/F}}{2}\right)$$

## **Model Checking & Diagnostics**

- Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.
- Posterior distributions for the Interaction between Study Drug and BAL will be produced and
  examined as part of the model fitting process (separate distribution per endpoint). If any of the
  endpoints is deemed to have a non-zero interaction then the treatment comparisons (study
  drug) will be obtained within each level of BAL, for BOTH endpoints and the same decision
  pathway will be applied to each. An example of the combinations required to obtain the
  Interaction term for PVPI is

$$\left(\frac{\hat{\mu}_{PC,P/F} + \hat{\mu}_{AV,P/F}}{2}\right) - \left(\frac{\hat{\mu}_{PV,P/F} + \hat{\mu}_{AC,P/F}}{2}\right)$$

 A SAS coding trick may be required to fit separate variance covariance matrices to work around a known bug in the SASv9.3 TS1M2 MCMC procedure. Separate response variables

## **Primary Statistical Analyses**

may be required for each treatment arm (with all values set to missing if the record was from a subject not on that treatment). Multiple MVN model statements would link these endpoints to a distinct VCV matrix. See MCMC training course notes "An intro. to Bayesian methods using SAS" by PPD GSK, February 2014" Slide 56+ for details.

## **Model Results Presentation**

- Posterior treatment effects (adjusted Active and Placebo means averaging over the levels of BAL) and differences (or ratios) to placebo (marginals from the joint posterior probability distribution of the comparisons) will be displayed graphically. In addition a bivariate contour plot of the joint posterior distribution for the comparisons in Figure 2 may be produced (with the decision criteria overlaid onto it and the marginal distributions displayed) – this may require bespoke programming.
- Median and 95% (equi-tail) credible intervals for the LSmean equivalents and Median and 95% (equi-tail) credible intervals for differences (or ratios) to placebo will be summarized.
- Posterior probabilities for the end of study decision pathway (and other cut points)

# **Sensitivity and Supportive Statistical Analyses**

- Other potential a priori covariates include "Endpoint by duration of surgical procedure" and
  "Endpoint by duration of one lung ventilation" interaction terms. Each duration term would enter
  the model as a centered continuous covariate. The study statistician may explore the
  appropriateness of these terms, and whether they should enter as linear or higher order terms
  via scatterplots of covariate vs each endpoint. Given the relatively small sample sizes and
  exploratory nature of the trial the final analysis model used to make inferences may be
  selected via a combination of expert judgment and formal statistical model selection techniques
  (e.g. Bayes factors).
- Intermediate model building outputs would not need to be formally reported only the final chosen model would have associated Tables, Figures and Listings.
- Optional (at discretion of study statistician): For robustness, assuming non-informative priors
  are used, the equivalent PROC MIXED model may be fitted and the LSMeans and estimates of
  differences compared to the results obtained from the PROC MCMC analysis. Output from this
  analysis may be listed as a stand alone output or as part of the MCMC raw SAS listings
  (conditional on PROC MIXED being used) with no corresponding Tables or Figures.
- The above analyses may be repeated using the Per Protocol 1 population if deemed necessary by the study statistician

# 8. SECONDARY STATISTICAL ANALYSES

# 8.1. Efficacy Analyses

# 8.1.1. Overview of Planned Efficacy Analyses

The secondary efficacy analyses will be based on the "Per Protocol 2" population, unless otherwise specified.

Table 4 provides an overview of the planned efficacy analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 4 Overview of Planned Efficacy Analyses

| Endpoint / Parameter/ | | Absolute | | | | | | | C | hange | from | Basel | ine | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | Stat | s Anal | lysis | Sum | mary | Indiv | ridual | Sta | Stats Analysis | | Sum | Summary | | idual |
| | Т | F | L | Τ | F | F | L | Τ | F | L | T | F | F | L |
| Transpulmonary Thermodilution⁵ | | | | | | | | | | | | | | |
| Joint Modelling of PVPI and P <sub>a</sub> O <sub>2</sub> /F <sub>i</sub> O <sub>2</sub> | Υ | Υ | Υ | | Y1 | | | | | | | | | |
| Pulmonary Vascular | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | | Υ | | | Υ |
| Permeability Index (PVPI) | · · | ' | | | | | ' | | | | · | | | ' |
| Extravascular Lung Water Index (EVLWI) <sup>4</sup> | Υ | Υ | Y | Y | Υ | Υ | Υ2 | | | | Y | | | <b>Y</b> 3 |
| Extravascular Lung<br>Water (EVLW) | | | | | | | Υ2 | | | | | | | |
| Arterial Line Used | | | | <b>Y</b> <sup>7</sup> | | | Υ | | | | | | | |
| Cardiac Output (CO) | | | | | | | Y2 | | | | | | | |
| Cardiac Index (CI) <sup>4</sup> | | | | Υ | | | Y2 | | | | Υ | | | <b>Y</b> 3 |
| Global End-Diastolic<br>Volume (GEDV) | | | | | | | <b>Y</b> <sup>2</sup> | | | | | | | |
| Global End-Diastolic Volume Index (GEDI) <sup>4</sup> | | | | Y | | | <b>Y</b> <sup>2</sup> | | | | Υ | | | <b>Y</b> 3 |
| Mean Arterial Pressure (MAP) | | | | Y | | | Υ | | | | Υ | | | Υ |
| Systemic Vascular<br>Resistance (SVR) | | | | | | | Υ | | | | | | | |
| Systemic Vascular<br>Resistance Index<br>(SVRI) <sup>4</sup> | | | | Y | | | Y | | | | Y | | | Y |
| Stroke Volume<br>Variation (SVV) | | | | Y | | | Υ | | | | Υ | | | Υ |
| Global Ejection<br>Fraction (GEF) | | | | Y | | | Υ | | | | Υ | | | Y |
| Heart Rate (HR) | | | | Υ | | | Υ | | | | Υ | | | Υ |
| Blood Pressure (AP): | | | | Y | | | Υ | | | | Y | | | Y |
| Systolic and Diastolic | | | | V | | | V | | | | V | | | V |
| Central Venous | | | | Υ | | | Υ | | | | Υ | | | Υ |

| Endpoint / Parameter/ | | | Α | bsolu | te | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | Stat | s Ana | ysis | Sumi | mary | Indiv | idual | Sta | ts Ana | lysis | Sum | mary | Indiv | idual |
| | Т | F | Г | Т | F | F | L | Т | F | L | Т | F | F | L |
| Pressure (CVP) | | | | | | | | | | | | | | |
| Predicted Body | | | | Υ | | | Υ | | | | | | | |
| Weight⁴ | | | | | | | | | | | | | | |
| Predicted Body | | | | Υ | | | Υ | | | | | | | |
| Surface Area <sup>4</sup> | | | | | | | | | | | | | | |
| Body Surface Area4 | | | | Υ | | | Υ | | | | | | | |
| Oxygenation | | | | | | | | | | | | | | |
| $P_aO_2/F_iO_2$ 4 | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | | Υ | | | Υ |
| SpO <sub>2</sub> /F <sub>i</sub> O <sub>2</sub> <sup>4</sup> | | | | Υ | Υ | Υ | Υ | | | | Υ | | | Υ |
| Correlation between | | | | | Y1 | | | | | | | | | |
| $P_aO_2/F_iO_2$ and | | | | | | | | | | | | | | |
| SpO <sub>2</sub> /F <sub>i</sub> O <sub>2</sub> <sup>4</sup> | | | | | | | | | | | | | | |
| Mean Airway Pressure | | | | Υ | | | Υ | | | | Υ | | | Υ |
| (Paw) | | | | | | | | | | | | | | |
| Oxygenation Index | | | | Υ | | | Υ | | | | Υ | | | Υ |
| SOFA | | | | | | | | | | | | | | |
| SOFA scores <sup>6</sup> | Υ | Υ | Υ | Υ | | Υ | Υ | | | | Υ | | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
  - 1. Represented as scatterplot matrix
  - 2. List replicate values and the derived mean
  - 3. Derive mean of the replicate values prior to computing the change from baseline
  - 4. Derived in house by GSK from data collected on eCRF.
  - Site instructed to set up machine to display the Absolute values and not the corresponding indexed values. If
    the site omitted to do this (monitors examining the PDF hard copy of the PiCCO output is an example of how
    GSK may be alerted) then GSK will derive corresponding absolute versions using the formulas in Section
    11.5.4.
  - 6. Add footnotes to change from baseline SOFA outputs explaining the strong assumptions required to obtain the Baseline (see Section 11.4.2.1)
  - 7. Summarise the Number of distinct individuals and % of big N for each Response category

# 8.1.2. Planned Efficacy Statistical Analyses

# Secondary Statistical Analyses (Repeated Measures Joint Modelling of PVPI and PaO2/FiO2)

#### Endpoint(s)

- All Post Surgery PVPI and P<sub>a</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub>
- Baseline: PVPI and P<sub>a</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> immediately prior to surgery (day 1)
- Any transformation of a response variable is also expected to be applied to the corresponding baseline variable. Final decisions on transformations will be based on the observed data and model diagnostics (PVPI is expected to require a Ln (natural logarithm) transformation)
- Any observations with missing model covariates (e.g. baseline) would be excluded from the model fitting process (i.e. also excluding the record from any centering of covariates)
- The above endpoints and baselines will be the average of any replicates available at the

# Secondary Statistical Analyses (Repeated Measures Joint Modelling of PVPI and PaO2/FiO2)

planned time points

# **Model Specification**

- Repeated measures version of the primary analysis (Section 7.1.2). Only changes related to the repeated measures are described in detail.
- 4x Post surgery Planned Timepoints: on completion of surgery day1, day 2 day 3 and day 4 (where available)
- Center by endpoint model parameters to be duplicated in the linear predictor (one repeat for each planned timepoint)
- Additional model parameters (continuous & centered) to capture the Baseline by planned timepoint interaction
- Obtain Bivariate and associated marginal distributions for the active Vs placebo comparisons (averaging over levels of BAL sampling) for each planned timepoint
- Care should be taken in how the data are sorted/arranged, since the ordering of variables will
  now contain information on both endpoint and timepoint. A simplified example linear predictor
  is shown below for baseline, immediately post op day1 and day 2 timepoints for a hypothetical
  subject from center 3, on active treatment, with BAL sampled from the collapsed lung with
  centered baseline values of -4.1 and -0.5 for P/F and PVPI respectively (note: additional
  covariates may be explored and added based on the observed data and the additional
  timepoints would be added in a similar style and alternative orderings of the data may be used
  if easier to implement in SAS):

# Secondary Statistical Analyses (Repeated Measures Joint Modelling of PVPI and PaO2/FiO2)

$$\begin{bmatrix} P/F & P/F & PVPI & PVPI \\ D_1 & D_2 & D_1 & D_2 \\ \hat{y}_1 & \hat{y}_2 & \hat{y}_3 & \hat{y}_4 \end{bmatrix} = [I(C_1) \ I(C_2) \ I(C_3) \ I(C_4) \ I(C_5)] *$$

$$\begin{split} & \left[ -4.1 \ -4.1 \ 0.5 \ 0.5 \right] \! \left[ Diag \! \left( \hat{B}S_{D1,P/F} \ \hat{B}S_{D2,P/F} \ \hat{B}S_{D1,PVPI} \ \hat{B}S_{D2,PVPI} \right) \! \right] + \\ & I \! \left( Pbo, Coll \right) * \left[ \hat{\mu}_{D1,PC,P/F} \ \hat{\mu}_{D2,PC,P/F} \ \hat{\mu}_{D1,PC,PVPI} \ \hat{\mu}_{D1,PC,PVPI} \ \hat{\mu}_{D2,PC,PVPI} \right] + \\ & I \! \left( Pbo, Vent \right) * \left[ \hat{\mu}_{D1,PV,P/F} \ \hat{\mu}_{D2,PV,P/F} \ \hat{\mu}_{D1,PV,PVPI} \ \hat{\mu}_{D2,PV,PVPI} \ \hat{\mu}_{D2,AC,PVPI} \right] + \\ & I \! \left( Act, Coll \right) * \left[ \hat{\mu}_{D1,AC,P/F} \ \hat{\mu}_{D2,AC,P/F} \ \hat{\mu}_{D1,AC,PVPI} \ \hat{\mu}_{D2,AV,PVPI} \ \hat{\mu}_{D2,AV,PVPI} \right] + \\ & I \! \left( Act, Vent \right) * \left[ \hat{\mu}_{D1,AV,P/F} \ \hat{\mu}_{D2,AV,P/F} \ \hat{\mu}_{D1,AV,PVPI} \ \hat{\mu}_{D2,AV,PVPI} \right] \end{split}$$

Where

Center<sub>5</sub> term(s) constrained to be zero and  $I(\bullet)$  is an Indicator function with value 1 if condition met and zero otherwise [Here I(Pbo, Coll), I(Pbo, Vent), I(Act, Vent) = 0, I(Act, Coll) = 1, I(C<sub>3</sub>) = 1 and I(C<sub>1</sub>), I(C<sub>2</sub>), I(C<sub>4</sub>) & I(C<sub>5</sub>) = 0]

To link to observed data assume:

$$\begin{bmatrix} P/F & P/F & PVPI & PVPI \\ D1 & D2 & D1 & D2 \\ y_1 & y_2 & y_3 & y_4 \end{bmatrix}^{MVN} \sim \begin{bmatrix} P/F & P/F & PVPI & PVPI \\ D1 & D2 & D1 & D2 \\ \hat{y}_1 & \hat{y}_2 & \hat{y}_3 & \hat{y}_4 \end{bmatrix}, [\Sigma_{Act}] \text{ where } \Sigma_{Act} \text{ is a } 4x4$$

Variance Covariance matrix for the active treatment arm

Posterior distributions are enumerated with appropriate combinations of

$$\begin{split} \hat{\mu}_{D1,PC,P/F}, \hat{\mu}_{D1,PV,P/F}, \hat{\mu}_{D1,PC,PVPI}, \hat{\mu}_{D1,PV,PVPI}, \hat{\mu}_{D1,AC,P/F}, \hat{\mu}_{D1,AV,P/F}, \hat{\mu}_{D1,AC,PVPI}, \hat{\mu}_{D1,AV,PVPI}, \\ \hat{\mu}_{D2,PC,P/F}, \hat{\mu}_{D2,PV,P/F}, \hat{\mu}_{D2,PC,PVPI}, \hat{\mu}_{D2,PV,PVPI}, \hat{\mu}_{D2,AC,P/F}, \hat{\mu}_{D2,AV,P/F}, \hat{\mu}_{D2,AC,PVPI}, \hat{\mu}_{D2,AV,PVPI} \\ e.g \text{ Sample from Posterior Distn for Day 2 Diff in Mean P/F averaging over BAL} = \end{split}$$

$$\left(rac{\hat{\mu}_{D2,AC,P/F} + \hat{\mu}_{D2,AV,P/F}}{2}
ight) - \left(rac{\hat{\mu}_{D2,PC,P/F} + \hat{\mu}_{D2,PV,P/F}}{2}
ight)$$

# **Model Checking & Diagnostics**

- Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.
- Checks similar to those for the Primary analysis of the interaction terms for Study Drug and BAL within each timepoint will be produced and if any of them suggest an interaction then ONLY the treatment comparisons within THAT timepoint only will be modified to account for the location of the BAL sampling

## **Model Results Presentation**

Sets of outputs analogous to the Primary analysis will be produced for each planned timepoint;

# Secondary Statistical Analyses (Repeated Measures Joint Modelling of PVPI and PaO2/FiO2)

although the end of study decision pathway would not be applied to the resulting probabilities.

# **Sensitivity and Supportive Statistical Analyses**

- A similar approach will be performed to the primary analysis. Refer to the Sensitivity and Supportive Statistical Analyses within the Primary Analysis Section 7.1.2
- The analysis may be repeated using the exploratory endpoint (Imputed PaO2/FiO2).

# Secondary Statistical Analyses (Univariate analyses – post surgery timepoint only) Endpoint(s)

- PVPI on completion of surgery
- EVLWI on completion of surgery
- P<sub>a</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> on completion of surgery

# **Model Specification**

- A similar Bayesian repeated measures modeling approach will be implemented (c.f. the Joint modeling approach in the Secondary Analysis of PVPI and P<sub>a</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub>; but with only one endpoint).
- If deemed necessary natural logarithms of the observed responses may be implemented on a per endpoint basis.

# **Model Checking & Diagnostics**

- Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.
- Checks similar to those for the Primary analysis of the interaction terms for Study Drug and BAL within each timepoint may be produced

#### **Model Results Presentation**

- Posterior means and treatment ratios will be displayed graphically.
- Median, mean and 95% credible intervals for treatment means and ratios of all time points, to immediately prior to surgery.
- Posterior probabilities that the ratios at all time points are less than 1, and other specific values

## **Sensitivity and Supportive Statistical Analyses**

 A similar approach will be performed to the primary analysis. Refer to the Sensitivity and Supportive Statistical Analyses within the Primary Analysis Section 7.1.2

#### Secondary Statistical Analyses (SOFA)

#### Endpoint(s)

• SOFA scores on Day 2 through to Day 4.

#### **Model Specification**

• A Bayesian repeated measures model will be fit to SOFA scores (observed and imputed) measured on Day 2, Day 3 and Day 4. The following categorical terms will be fit in the model: Day, Treatment and Treatment \* Day, where Day is the repeated measures factor and treatment uses the 4x main treatment levels. An assessment will be made by the study statistician regarding including Baseline SOFA as a continuous covariate. The model will assume non-informative priors for all parameters. The modeling will implicitly combine the BAL sampling levels by study drug arm. The adjusted means for each Study Drug by Day will be obtained and the posterior distributions of these quantities will be displayed graphically, and the median and 95% credible interval (equi-tailed) will be calculated. Posterior distributions of (combined) Active - Placebo for each post surgery time point will be generated. The posterior

## Secondary Statistical Analyses (Univariate analyses – post surgery timepoint only)

probabilities that these differences, representing the true effect size, at each time point are less than 0, less than -1, less than -2 and less than -3 will be produced, in addition to other values which will be determined upon inspection of the data.

# **Model Checking & Diagnostics**

- Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.
- Checks similar to those for the Primary analysis of the interaction terms for Study Drug and BAL within each timepoint may be produced

#### **Model Results Presentation**

- Adjusted medians and 95% credible intervals will be presented for each study drug by day, together with the median estimated study drug differences (Active – Placebo) and the corresponding 95% credible intervals.
- Plots of medians and 95% credible intervals from the model will be generated for each study drug by time point. Additionally, plots of differences and 95% credible intervals for the comparison of interest will be generated
- Bayesian posterior probabilities that the true differences for each of the active treatments and placebo are greater than various levels will be produced, assuming non informative priors

## Sensitivity and Supportive Statistical Analyses

 A similar approach will be performed to the primary analysis. Refer to the Sensitivity and Supportive Statistical Analyses within the Primary Analysis Section 7.1.2

# 8.2. Safety Analyses

# 8.2.1. Overview of Planned Analyses

The safety analyses will be based on the "Safety" population, unless otherwise specified.

Table 5 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 5 Overview of Planned Safety Analyses

| Endpoint / Parameter/ | | Ab | solute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| Display Type | Sui | mmary | Indiv | ridual | Sum | mary | Indiv | ridual |
| | T | F | F | L | T | F | F | L |
| Adverse Events | | | | | | | | |
| All AE's <sup>1.</sup> | Υ | | | Υ | | | | |
| All Drug-related AE's | Υ | | | | | | | |
| Serious AE's | Υ | | | Υ | | | | |
| Withdrawal AE's | | | | Υ | | | | |
| European Medicines | Υ | | | | | | | |
| Agency: Summaries for | | | | | | | | |
| the European Clinical | | | | | | | | |
| Trials Database (EudraCT) | | | | | | | | |
| Clinical Laboratory | | | | | | | | |
| Clinical Chemistry <sup>2</sup> | Υ | | | Υ | | | | |
| Hematology <sup>2</sup> | Υ | | | Υ | | | | |
| Urinalysis <sup>3</sup> | Υ | | | | | | | |
| ECG | | | | | | | | |
| ECG Findings | Υ | | | Υ | Υ | | | |
| ECG Values | Υ | | | Y <sup>4</sup> | | | | |
| Vital Signs | | | | | | | | |
| Vitals Values | Υ | | | Υ | | | | |
| Immunogenicity | | | | | | | | |
| Immunogenicity results | Υ | | | Υ | | | | |
| Surgical Procedure | | | | | | | | |
| Subject level information | | | | Υ | | | | |
| related to the Surgical | | | | | | | | |
| Procedure | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Listings will include subject's numbers for individual AE's & AE system organ classes, preferred terms and verbatim text.
- 2. Listings of chemistry (and/or haematology) abnormalities of PCI and all values for subjects with chemistry (and/or haematology) abnormalities of PCI. CRP to be excluded from these summaries (but will be included in the Biomarker outputs)
- 3. Urinalysis results may be mapped to common nomenclatures prior to summarising
- 4. Listings of ECG values of PCI and all ECG values for subjects with any PCI

# 8.3. Pharmacokinetic Analyses

# 8.3.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

Table 6 provides an overview of the planned analyses, with full details being presented in Appendix 14: List of Data Displays.

Table 6 Overview of Planned Pharmacokinetic Analyses

| Endpoint / Parameter/ | Untransformed | | | | | | | Log-Transformed | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | Stats Analysis | | Summary | | Individual | | Stats Analysis | | | Summary | | Individual | | |
| | T | F | L | T | F | F | L | Т | F | L | Т | F | F | L |
| Blood | | | | | | | | | | | | | | |
| Plasma Drug | | | | Υ | Υ | Υ | Υ | | | | | Υ | Υ | |
| Concentration | | | | I | I | I | I | | | | | I | I | |
| Derived PK | | | | <b>&gt;</b> | | | Υ | | | | V | | | |
| Parameters | | | | I | | | I | | | | I | | | |
| BAL | | | | | | | | | | | | | | |
| BAL Drug | | | | | | | Υ | | | | | | | |
| Concentration | | | | | | | I | | | | | | | |
| Plasma Urea & BAL | | | | | | | Υ | | | | | | | |
| Urea | | | | | | | I | | | | | | | |
| Dilution Factor | | | | | | | Υ | | | | | | | |
| Volume of ELF fluid <sup>1.</sup> | | | | Υ | | | Υ | | | | | | | |
| Volume of BAL fluid | | | | | | | Υ | | | | | | | |
| Total Drug in BAL fluid | | | | | | | Υ | | | | | | | |
| Derived ELF Drug | | | | <b>V</b> | | | Υ | | | | | Υ | | |
| Concentration <sup>1.</sup> | | | | ' | | | ı | | | | | ı | | |

## NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Corrected for Dilution Factor.

# 8.3.2. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 11.4.3 Reporting Process & Standards).

#### 8.3.3. Pharmacokinetic Parameters

# 8.3.3.1. Deriving Pharmacokinetic Parameters

• Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 11.4.3 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using WinNonLin Phoenix.
- All calculations of non-compartmental parameters will be based on actual sampling times.
- Pharmacokinetic parameters described in Table 7 will be determined from the plasma concentration-time data, as data permits.

Table 7 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| Tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| t½ | Apparent terminal half-life will be calculated as: |
| | t½ = In2 / lambda_z |

#### NOTES:

- Additional parameters may be included as required.
- Lambda\_z is the terminal phase rate constant estimated by linear regression analysis of the loge transformed concentration-time data

Section 11.5.5 details the BAL PK parameters to be derived, as data permits. These too will be summarised and listed.

#### 8.3.3.2. Statistical Analysis of Pharmacokinetic Parameters

There will be no formal statistical analyses of the pharmacokinetic parameter data. PK parameters will be calculated based on the available data and listed.

#### 8.4. Pharmacodynamic (Biomarker) Analyses

#### 8.4.1. Overview of Planned Pharmacodynamic (Biomarker) Analyses

The pharmacodynamic analyses will be based on the "Per Protocol 2" population, unless otherwise specified (e.g. for BAL related analyses which use "Per Protocol 1"). Further details of the biomarkers can be found in Appendix 8.

Table 8 provides an overview of the **planned** pharmacodynamic (Biomarker) analyses, with full details of data displays being presented in Appendix 14: List of Data Displays. Additional biomarkers may be added (or removed), and will follow a similar analysis strategy and any additional outputs would take the next available number.

Table 8 Overview of Planned Pharmacodynamic (Biomarker) Analyses

| Endpoint / Parameter/ | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | A | | | Absolu | ıte | | | | CI | hange | from | Basel | ine | |
| | Sta | ts Ana | lysis | Sum | mary | Indiv | /idual | Stat | s Ana | lysis | Sum | mary | Indiv | idual |
| | T | F | L | Т | F | F | L | Т | F | L | T | F | F | L |
| BAL | | | | | | | | | | | | | | |
| Free sTNFR1 | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| Total sTNFR1 | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| Complex sTNFR1 | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| TNFa | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| IL-6 | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| IL-8 | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| IL-1b | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| MCP-1 | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| CRP∆ | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| IL-1ra | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| IL-10 | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| Total protein | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| Total protein ratio | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| Surfactant Protein D | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| (SP-D) | | | | | | | | | | | | | | |
| RAGE | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| CC16 | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| vWF | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| sICAM | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| MPO | Υ | Υ | Υ | Υ | Υ | | Υ | | | | | | | |
| Serum (Plasma when s | | | | | 1 | T | 1 | 1 | 1 | 1 | | 1 | | |
| Free sTNFR1 | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | | Υ | | | Υ |
| Total sTNFR1 | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | | Υ | | | Υ |
| Complex sTNFR1 | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | | Υ | | | Υ |
| IL-6 | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | | Υ | | | Υ |
| IL-8 | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | | Υ | | | Υ |
| CRP∆ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | | Υ | | | Υ |
| Total Protein [Plasma] | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | | Υ | | | Υ |
| Surfactant Protein D (SP-D) | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | | Υ | | | Υ |

| Endpoint / Parameter/ | Untransformed/Transformed as appropriate | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | | Absolute | | | | | | | Change from Baseline | | | | | |
| | Stat | Stats Analysis | | | mmary Individual | | | Stats Analysis S | | | Sum | mary | Indiv | idual |
| | Т | F | L | T | F | F | L | Т | F | L | Т | F | F | L |
| RAGE | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | | Υ | | | Υ |
| CC16 | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | | Υ | | | Υ |
| vWF | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | | Υ | | | Υ |
| sICAM | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | | Υ | | | Υ |
| MPO | Υ | Υ | Υ | Υ | Υ | Y | Υ | | | | Υ | | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Δ=Run as part of Clinical Chemistry Labs and therefore may have different timepoints and require subsequent adjustments to the model / displays. For BAL there is only a single timepoint

#### 8.4.2. Planned Pharmacodynamic (Biomarker) Statistical Analyses

## Planned Statistical Analyses (BAL Biomarkers)

#### Endpoint(s)

- Absolute value of BAL biomarker (separate analysis per biomarker)
- Any observations with missing model covariates would be excluded from the model fitting process (i.e. also excluding the record from any centering of covariates)

#### **Model Specification**

- For each biomarker, the values will be inspected to determine whether a data transformation is required.
- Main Treatment Descriptors to be used (i.e. 4 levels of the treatment term)
- No intercept terms should be fitted for either endpoint (due to fitting all 4 levels of treatment).
- Categorical fixed effect should be added for Center (if recruitment is such that center terms
  are poorly estimated then appropriate action will be taken, including but not limited to, pooling
  of centers or removal of the term from the model).
- Non-informative priors will be utilized for each model parameter assigned either as a normal distribution centered on 0 with large variance 1E6 or as appropriate to the parameters distribution.
- Separate Variance parameters for each treatment arm.
- SAS PROC MCMC will be used to combine the non-informative priors with the data observed
  to obtain sufficient draws from the posterior distribution (after any thinning) such that the
  MCSE/SD values for parameters of interest are less than 0.01 (anticipated to be in the region
  of ~100,000 draws). If model convergence is poor then alternative initial parameter values
  should be considered.
- The randomization seed used in PROC MCMC should itself be generated with an element of randomness - but there is no need to formally document this process (e.g. using Excel function RANDBETWEEN [1,9999999] and copying the result into the SAS code)
- Combinations of the fitted model parameters will be used to answer the clinically relevant questions.
- Median values of the adjusted response for each level of the main treatment descriptors and their associated 95% credible intervals (equi-tailed) will be produced from the posterior

#### Planned Statistical Analyses (BAL Biomarkers)

distributions obtained via appropriate combinations of the fitted model parameters; akin to lease square means

- Posterior distributions will be obtained for the Active vs Placebo comparison within each level
  of the BAL sampling. These distributions will be used to determine the probability of any
  reduction and any increase c.f. placebo. In addition posterior probabilities of the differences (or
  ratios) for other cut-points (which may be determined upon inspection of the data, or from
  developing business requirements), may also be computed.
- Where applicable estimates would be derived at the means of any model covariates, akin to least squares means in PROC MIXED, and back transformed if necessary. When covariates are centered before the model fitting their mean is zero so the covariate can be dropped from the derivation.

#### **Model Checking**

- Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.
- Potential covariates may also be explored (e.g. duration of surgery, age, gender). Only outputs from the final model will be reported

#### **Model Results Presentation**

- By subject time profiles of biomarkers will be produced.
- Scatterplot matricies of the correlation structures between BAL biomarkers may be produced.
- Median and 95% (equi-tail) credible intervals for the LSmean equivalents and Median and 95% (equi-tail) credible intervals for differences (or ratios) to placebo will be summarized.
- Posterior probabilities for the cut points

#### Planned Statistical Analyses (Serum Biomarkers)

#### Endpoint(s)

- Absolute value of serum biomarker response (separate analysis per biomarker)
- Timepoints: Day 1 (on completion of surgery), day 2, day 3, day 4 and day 8
- Baseline: day 1 (Pre-dose)
- Any transformation of a response variable is also expected to be applied to the corresponding baseline variable. Final decisions on transformations will be based on the observed data and model diagnostics (all biomarkers are expected to require a Ln (natural logarithm) transformation)
- Any observations with missing model covariates (e.g. baseline) would be excluded from the model fitting process (i.e. also excluding the record from any centering of covariates)

#### **Model Specification**

- The (transformed) endpoints will be assumed to follow a multivariate normal distribution.
   Linear predictors will be derived for each subject (i.e. obtain a vector of means for the MVN distribution). Each treatment arm will also have a separate variance covariance matrix.
- The linear predictors will consist of mean vectors to capture the effect of treatment for each time point and a variety of other model terms (an example is given at the end of this text).
- Main Treatment Descriptors to be used (i.e. 4 levels of the treatment term)
- No intercept terms should be fitted for either endpoint (due to fitting all 4 levels of treatment).
- Baseline vectors will be fitted as continuous covariates (baseline values should be centered
  prior to inclusion in the model, centering to occur after any transformation of the individual
  subjects responses).

#### Planned Statistical Analyses (Serum Biomarkers)

- Categorical fixed effect vectors should be added for Center (if recruitment is such that center terms are poorly estimated then appropriate action will be taken, including but not limited to, pooling of centers or removal of the term from the model).
- Non-informative priors will be utilized for each model parameter assigned either as a normal distribution centered on 0 with large variance 1E6 or as appropriate to the parameters distribution.
- Each of the 4x variance covariance matrices will use an inverse Wishart distribution as its prior.
- SAS PROC MCMC will be used to combine the non-informative priors with the data observed
  to obtain sufficient draws from the posterior distribution (after any thinning) such that the
  MCSE/SD values for parameters of interest are less than 0.01 (anticipated to be in the region
  of ~100,000 draws). If model convergence is poor then alternative initial parameter values
  should be considered.
- The randomization seed used in PROC MCMC should itself be generated with an element of randomness - but there is no need to formally document this process (e.g. using Excel function RANDBETWEEN [1,9999999] and copying the result into the SAS code)
- Combinations of the fitted model parameters will be used to answer the clinically relevant questions.
- Median values of the baseline adjusted response for each treatment by timepoint combination and their associated 95% credible intervals (equi-tailed) will be produced from the posterior distributions obtained via appropriate combinations of the fitted model parameters; akin to lease square means
- Posterior distributions will be obtained for the Active vs Placebo comparison within each level
  of the BAL sampling for each time point. These distributions will be used to determine the
  probability of any reduction and any increase c.f. placebo. In addition posterior probabilities of
  the differences (or ratios) for other cut-points (which may be determined upon inspection of the
  data, or from developing business requirements), may also be computed.
- Where applicable estimates would be derived at the means of any model covariates, akin to least squares means in PROC MIXED, and back transformed if necessary. When covariates are centered before the model fitting their mean is zero so the covariate can be dropped from the derivation.

#### **Model Checking**

- Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.
- Potential covariates may also be explored (e.g. duration of surgery, age, gender). Only outputs from the final model will be reported

#### **Model Results Presentation**

- By subject time profiles of biomarkers will be produced.
- Scatterplot matricies of the correlation structures between BAL biomarkers may be produced (one page per timepoint – including baseline).
- Median and 95% (equi-tail) credible intervals for the LSmean equivalents and Median and 95% (equi-tail) credible intervals for differences (or ratios) to placebo will be summarized.
- Posterior probabilities for the cut points

#### 9. OTHER STATISTICAL ANALYSES

## 9.1. Exploratory Statistical Analyses

The strategy for each exploratory endpoint is to list and summarise by Study Medication (i.e. Assume BAL sampling location is irrelevant). Subsequent statistical analysis may be conditional on the observed data (at the discretion of the study statistician) and methods would be documented in the CSR.

Table 9 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 9 Overview of Planned Exploratory Statistical Analyses

| Endpoint / Parameter/ | | Ab | solute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| Display Type | Su | Summary | | idual | Sum | mary | Individual | |
| | T | F | F | L | Т | F | F | L |
| Clinical Outcomes | | | | | | | | |
| Diagnosis of ARDS out to | Υ | | | Υ | | | | |
| day 28 | | | | | | | | |
| 28 day survival | Υ | Υ | | Υ | | | | |
| Organ failure free days out | Υ | | | Υ | | | | |
| to day 28 | | | | | | | | |
| Resource Utilisation | | | | | | | | |
| Ventilator Free Days | Υ | | | Υ | | | | |
| ICU Length of Stay | Υ | | | Y | | | | |
| Hospital Length of Stay | Υ | | | Υ | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 10. REFERENCES

GlaxoSmithKline Document Number 2014N197251\_04 Study ID TFR116341. APlacebo Controlled, Double-blind, Multi-centre, Single Dose, Parallel Group, Randomised Clinical Trial of GSK2862277 in Patients undergoing Oesophagectomy Surgery. Report Date 16-FEB-2015.

Pandharipande PP, Shintani AK, Hagerman HE, St Jacques PJ, Rice TW, Sanders NW, Ware LB, Bernard GR, Ely EW. Derivation and validation of Spo2/Fio2 ratio to impute for Pao2/Fio2 ratio in the respiratory component of the Sequential Organ Failure Assessment score. Crit Care Med. 2009 Apr;37(4):1317-21. doi: 10.1097/CCM.0b013e31819cefa9.

Perkins G.D., Gates S, Park D., Gao F., Knox C, Holloway B, McAuley D.F, Ryan J., Marzouk J, Cooke M.W., Lamb S.E., Thickett D.R.. The Beta Agonist Lung Injury Trial (BALTI) Prevention: A Randomized Controlled Trial. AJRCCM. In press Jan 2014

Rice T.W. et al, 2007: Comparison of the SpO2/FIO2 Ratio and the PaO2/FIO2 Ratio in Patients With Acute Lung Injury or ARDS. CHEST (Critical Care Med.) 2007; 132:410–417

Vincent JL, Moreno R, Takala J, Willatts S, De Mendonça A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996; 22:707-10.

## 11. APPENDICES

| Section | Component |
|---|---|
| 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 11.2 | Appendix 2: Time & Events |
| 11.3 | Appendix 3: Treatment States and Phases |
| 11.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 11.5 | Appendix 5: Derived and Transformed Data |
| 11.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| 11.7 | Appendix 7: Values of Potential Clinical Importance |
| 11.8 | Appendix 8: Biomarker Details |
| 11.9 | Appendix 9: Examination of Covariates, Subgroups & Other Strata |
| 11.10 | Appendix 10: PVPI and EVLW – Supplementary Information |
| 11.11 | Appendix 11: Model Checking and Diagnostics for Statistical Analyses. |
| 11.12 | Appendix 12: Details of Simulation exercise that produced operational characteristics used in the protocol |
| 11.13 | Appendix 13: Abbreviations & Trade Marks |
| 11.14 | Appendix 14: List of Data Displays |
| 11.15 | Appendix 15: Example Mock Shells for Data Displays |

# 11.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

#### 11.1.1. Exclusions from Per Protocol Populations

A subject meeting any of the following criteria will be excluded from the Per Protocol population:

| Per<br>Protocol<br>Population<br>ID | Number | Exclusion Description |
|---|---|---|
| 1 | 01 | Subject did not satisfy all of the inclusion and exclusion criteria (from whichever version of the protocol was active at the time of their enrolment) |
| | 02 | Subject did not receive either i) the study drug they were randomised to, or ii) the actual BAL lung sampled was not the one they were randomised to have sampled |
| | 03 | Subject was classified as inoperable upon commencement of surgical procedures (an "open and shut" case) |
| 2 | 01 | Subject did not satisfy all of the inclusion and exclusion criteria (from whichever version of the protocol was active at the time of their enrolment) |
| | 02 | Subject did not receive the study drug they were randomised to |
| | 03 | Subject was classified as inoperable upon commencement of surgical procedures (an "open and shut" case) |
| 3 | 01 | Subject did not satisfy all of the inclusion and exclusion criteria (from whichever version of the protocol was active at the time of their enrolment) |
| | 02 | Actual BAL lung sampled for the subject was not the one they were randomised to have sampled |
| | 03 | Subject was classified as inoperable upon commencement of surgical procedures (an "open and shut" case) |

#### NOTES:

• The above definitions may be modified during the in-stream protocol deviation reviews (for example, subjects who were deemed to be in-operable upon commencement of their surgical procedure may be added to each of the per protocol populations – this may require anecdotal evidence followed up by bespoke communications between GSK and the sites as it is not possible to guarantee such scenarios could be accurately defined using rules based on duration of surgery alone) A planned eCRF update should add a variable indicating if an individual was an "open and shut case". Prior to this update manual coding may be required to correctly compute the above populations (and also if the new variable is not retrospectively populated for existing subjects, e.g. those in IA1)

## 11.2. Appendix 2: Time & Events

## 11.2.1. Protocol Defined Time & Events

Table 10 Time and Events Table (Screening)

| Procedures | Screening (7 to 28 days inclusive prior to surgery) | 1. | Rest the subject in a supine or semi-<br>recumbent position for at least 5 min and<br>then take three measurements 5 minutes |
|---|---|---|---|
| Informed Consent | Χ | | apart. |
| Demography | Χ | 2. | HIV testing dependent on local practice |
| Medical History | Χ | 3. | If repeat screening is required previous |
| Smoking Status & History | Х | ] . | results from ADA screening and |
| Quantiferon-GOLD for TB <sup>3</sup> | Х | | Quantiferon-GOLD testing can be used for |
| HepB, HepC, HIV testing <sup>2</sup> | Х | | up to 60 days. |
| Inclusion/Exclusion Criteria | Х | | |
| Concomitant Medication | Χ | | |
| Physical Examination | Х | | |
| Vital Signs | Х | | |
| 12-lead ECG <sup>1</sup> | Χ | | |
| Serious Adverse Events | Χ | | |
| Clinical Labs including Haematology and Chemistry | X | | |
| Pre-existing ADA screening <sup>3</sup> | Х | | |
| Pharmacogenetics (PGx) sample <sup>3</sup> | Х | | |
| IVRS | Х | | |

Table 11 Time and Events Table Day 1

| Procedures | Pre-dose <sup>4</sup> | 0 h1 | 1 h | Immediately prior or at start of surgery | On<br>completion<br>of surgery | activities may be conducted up-to 72 |
|---|---|---|---|---|---|---|
| Randomisation | X <sup>2</sup> | | | | | hours prior to administration of study |
| Brief Physical Examination | Χ | | | | | treatment. 3.Only applicable at designated sites |
| Concomitant Medication | | | | Χ | | 4.Can be taken up to 24 hours prior to |
| IVRS | X <sup>2</sup> | | | | | dosing |
| Vital Signs | Χ | | Χ | | | 5.If 12 lead ECG is not available, |
| 12-lead ECG | Χ | | <b>X</b> 5 | | | monitoring by 3 lead ECG/telemetry |
| Adverse Events | | | | Χ | | (or similar) is acceptable |
| Serious Adverse Events | | | | Χ | | NB: Time points (except pre-dose) refer |
| Clinical Labs including Haematology and Chemistry | Х | | | | | to post-start of drug administration on Day 1. Pre-dose is defined as the time from admission to hospital up to the administration of study treatment. |
| Blood sample for immunogenicity | Х | | | | | |
| Blood sample for PK | Χ | | Χ | | Х | |
| Blood sample for urea and total protein | | | | | Х | |
| Blood samples for translational sub-study <sup>3</sup> | Х | | | | Х | |
| Sample for Urinalysis | Χ | | | | | |
| Blood sample for serum biomarkers | Х | | | | Х | |
| Nebulised (IH) Study<br>Treatment | | Χ | | | | |
| Transpulmonary thermodilution | | | | Х | Х | |
| P/F Ratio: • Arterial blood sample • Record FiO <sub>2</sub> | | | | Х | Х | |
| Measure SpO <sub>2</sub> using pulse oximetry | | | | Х | Х | |
| BAL Sampling | | | | | Χ | |

Table 12 Time and Events Table (Days 2 to 28)

| Procedures | Day<br>2 | Day<br>3 | Day<br>4 | Daily until<br>discharge | Day<br>81 | Day of discharge | Day<br>28<br>(FU)<br>±3<br>days | 1. | If discharged<br>before Day 8<br>take blood and<br>urine samples on<br>day of discharge<br>PVPI will be |
|---|---|---|---|---|---|---|---|---|---|
| Concomitant Medication | Χ | Χ | Χ | Х | | Х | Χ | | measured via |
| IVRS | | | | | | Х | Χ | | single-indicator |
| Transpulmonary<br>thermodilution <sup>2</sup> | Х | Χ | Х | | | | | | transpulmonary<br>thermodilution as |
| P/F Ratio • Arterial blood sample (as | Х | Х | Х | | | | | | long as the<br>subject remains<br>in the ICU with a<br>patent indwelling |
| Measure SpO <sub>2</sub> using pulse oximetry | Χ | Χ | Χ | | | | | | PiCCO catheter,<br>up to Day |
| Additional SOFA Components³ Glasgow Coma Score (GCS) Record Mean Arterial Pressure⁴ or administration of vasopressors required Bilirubin Platelets Creatinine (or urine output) | X | X | X | | | | | <ol> <li>4.</li> </ol> | sequential Organ Failure Assessment (SOFA) Score will only be calculated up to Day 4. If no arterial blood sample calculate MAP using equation: 2X diastolic blood pressure + systolic blood |
| Vital Signs | | | Х | | | Х | Χ | | pressure. Then |
| 12-lead ECG | Χ | | Χ | | | X | | 5. | divide by 3. |
| Adverse Events | Χ | Χ | Χ | Х | Χ | Х | Χ | Ο. | Only applicable<br>at designated |
| Serious Adverse Events | Χ | Χ | Χ | Х | Χ | Х | Χ | | sites |
| Clinical Labs including<br>Haematology and Chemistry | Х | Χ | Х | | Х | | | 6. | Sample to be taken 24 to 26 |
| Blood sample for serum | Χ | Χ | Χ | | Χ | | | | hours post-dose |
| Blood samples for translational sub-study <sup>5</sup> | Х | | | | | | | | of study<br>treatment. |
| Blood sample for | | | | | Х | | Χ | 7. | Sample to be |
| Immunogenicity Blood sample for PK | X6 | <b>X</b> <sup>7</sup> | | | | | | | taken 46 to 50 |
| Sample for Urinalysis | Λ* | Λ' | | | Х | | | | hours post-dose<br>of study<br>treatment. |


TFR116341

| | | | Daily until | | Day of | Day<br>28 | | |
|---|---|---|---|---|---|---|---|---|
| Procedures | Day<br>2 | discharge | Day<br>81 | discharge ±3 | (FU)<br>±3<br>days | 3 | Organ Failure Free Days needs to be recorded every day until | |
| Organ Failure Free Days | | | | | | X8 | | Day 28 (See |
| ARDS diagnosis status | | | | | Χ | | | SPM). |
| Ventilator Free Days | | | | | | Х | | |
| ICU & Hospital Length of Stay | | | | | Χ | | | |
| Survival | | | | | | Χ | | |

### 11.3. Appendix 3: Treatment States and Phases

#### 11.3.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to Study Treatment Start date & time. Since this is a single dose study and the time spent on the nebuliser (On-treatment) is expected to be 3-5 minutes a separate "On-treatment" phase is not required for this study.

| Treatment Phase | Definition |
|-----------------|-------------------------------------------------|
| Pre-Treatment | Date & Time ≤ Study Treatment Start Date & Time |
| Post-Treatment | Date & Time> Study Treatment Start Date & Time |

#### 11.3.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start date & time of the study treatment.

#### 11.3.2.1. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date & Time ≤ Study Treatment Start Date & Time |
| Post-Treatment | AE Start Date & Time > Study Treatment Start Date & Time |
| During Surgery | If Start of Surgery Date & Time ≤ AE Start Date & Time < End of Surgery Date & Time |
| Onset Time<br>Since 1st Dose<br>(Days Hours<br>Minutes) | AE Onset Date & Time - Treatment Start Date & Time converted to D H M format by tu_times |
| Duration (Days<br>Hours Minutes) | AE Resolution Date & Time – AE Onset Date & Time converted to D H M format by tu_times If resolution time not available then AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on Inform OR value is missing |

## 11.4. Appendix 4: Data Display Standards & Handling Conventions

#### 11.4.1. Study Treatment & Sub-group Display Descriptors

| | Main Treatment Group Descriptions | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporting | |
| Code | Description | Description | Order [1] |
| А | Placebo (BAL Collapsed lung) | Placebo (BAL Collapsed lung) | 1 |
| В | Placebo (BAL Ventilated lung) | Placebo (BAL Ventilated lung) | 2 |
| С | GSK2862277 (BAL Collapsed lung) | GSK2862277 26mg IH (BAL<br>Collapsed lung) | 3 |
| D | GSK2862277 (BAL Ventilated lung) | GSK2862277 26mg IH (BAL<br>Ventilated lung) | 4 |

#### NOTES:

In addition two alternative sets of treatment descriptors are required. Unless otherwise stated the outputs should use the main treatment group descriptions

| Alternative Treatment Group Descriptions #1 | | | |
|---|---|---|---|
| | RandAll NG Alternative Data Displays for Reporting | | |
| Code | Description | Description | Order [1] |
| Α | Placebo (BAL Collapsed lung) | Placebo | 1 |
| В | Placebo (BAL Ventilated lung) | | |
| С | GSK2862277 (BAL Collapsed lung) | GSK2862277 26mg IH | 2 |
| D | GSK2862277 (BAL Ventilated lung) | | |

#### NOTES:

1. Order represents treatments being presented in TFL, as appropriate.

| Alternative Treatment Group Descriptions #2 | | | |
|---|---|---|---|
| | RandAll NG | Alternative Data Displays for Reporting | |
| Code | Description | Description | Order [1] |
| Α | Placebo (BAL Collapsed lung) | BAL Collapsed lung | 1 |
| С | GSK2862277 (BAL Collapsed lung) | | |
| В | Placebo (BAL Ventilated lung) | BAL Ventilated lung | 2 |
| D | GSK2862277 (BAL Ventilated lung) | | |

#### NOTES:

1. Order represents treatments being presented in TFL, as appropriate.

<sup>1.</sup> Order represents treatments being presented in TFL, as appropriate.

#### 11.4.2. Baseline Definition & Derivations

#### 11.4.2.1. Baseline Definitions

For all endpoints (expect as noted in baseline definitions) the baseline value will be the latest pre-dose assessment.

| Parameter | Study Ass | Baseline Used in | | |
|---|---|---|---|---|
| | Day 1<br>(Pre-Dose) | Day 1 (<br>Immediately<br>prior to start of<br>surgery) | Day 2 | Data Display |
| Primary | | | | |
| PVPI | | X | | Day 1 (Immediately prior to start of surgery) |
| Secondary | | | | |
| Transpulmonary Thermodilution output | | X | | Day 1 (Immediately prior to start of surgery) |
| PaO2/FiO2 Ratio | | X | | Day 1 (Immediately prior to start of surgery) |
| SOFA <sup>1</sup> | Х | | | Derived Day 1 (Predose) |
| Biomarkers | | | | |
| Biomarker (Blood /<br>Serum) | Х | | | Day 1 (Pre-dose) |
| Immunogenicity | Х | | | Day 1 (Pre-dose) |

#### NOTES:

- Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.
- 1 = See Section 11.5.4 for assumptions required to derive a Baseline SOFA score

#### 11.4.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 11.4.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

#### 11.4.3. **Reporting Process & Standards**

| Reporting Process | |
|---|---|
| Software | Software |
| The currently sup- | The currently supported versions of SAS software will be used. |
| Reporting Area (Fin | Reporting Area (Final reporting effort at end of study) |
| HARP Server | : uk1salx00175 |
| HARP Area | : gsk2862277/tfr116341/final |
| QC Spreadsheet | : gsk2862277/tfr116341/final/documents |
| Reporting Area (Inte | Reporting Area (Interim analysis 1) |
| HARP Server | : uk1salx00175 |
| HARP Area | : gsk2862277/tfr116341/ia1 |
| QC Spreadsheet : gsk2862277/tfr116341/ia1/documents | |
| Reporting Area (Interim analysis 2) | |
| HARP Server | : uk1salx00175 |
| HARP Area | HARP Area : gsk2862277/tfr116341/ia2 |
| QC Spreadsheet : gsk2862277/tfr116341/ia2/documents | |
| Analysis Datasets | |

#### Analysis Datasets

- Analysis datasets will be created according to Legacy GSK A&R dataset standards AND/OR the set of CDISC standards implemented at GSK at time of database freeze (SDTM IG Version X.X & AdaM IG Version X.X.
- Any interim analysis is expected to be performed using Legacy GSK A&R dataset standards but the final reporting is expected to be performed in CDISC. However, if recruitment rates are high and/or the study is stopped after an interim analysis then the final reporting may also use the Legacy GSK A&R dataset standards.
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated for the final reporting effort (but will not be generated for the ia1 and ia2 reporting efforts).

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - o 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - o 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for

#### **Reporting Standards**

reporting of data based on the raw data collected.

- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings. They may also be omitted from figures, summaries and statistical analyses if the time deviation was deemed to be clinically impactful.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits / data points may be included in figures if it is relevant. Relevant outputs would typically be those focused on safety, and unscheduled visits / data points may be included in derivations of some endpoints (e.g. maximum post dose change from baseline body temperature). Less relevant outputs are those which aid activities that would not inherently utilise unscheduled visits / data points such as statistical modelling. For example, an individual subject time profile of body temperature should include any unscheduled temperature values; but a figure summarising body temperatures by treatment prior to statistical modelling should not display the unscheduled visit / data points.
- All unscheduled visits will be included in listings.

| - 7 til diloolloddiod | 7 in another with the included in notinge. |
|---|---|
| <b>Descriptive Summa</b> | Descriptive Summary Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharm | acokinetic Concentration Data |
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharm | Reporting of Pharmacokinetic Parameters |
| Descriptive<br>Summary Statistics<br>(Log Transformed) | <ul> <li>N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between geometric coefficient of variation CVb (%) will be reported.</li> <li>[1] CV<sub>b</sub> (%) = √ (exp(SD²) - 1) * 100 (SD = SD of log transformed data)</li> </ul> |
| Parameters Not<br>Being Log | Tmax |

| Transformed | |
|---|---|
| | Additionally, include the first point, last point and number of points used in he determination of lambda_z for listings. |

#### **Graphical Displays**

- Refer to IDSL Statistical Principals 7.01 to 7.13.
- The currently supported versions of the SAS SGxxx graphics procedures should be default
  choice for graphical displays (except for graphics produced by CPMS who may use their
  preferred software). If SGxxx cannot produce a required graphic then alternative software may
  be used. The default graphics options in SGxxx procedures may supersede IDSL Statistical
  Principals 7.01 to 7.13 (e.g. font choices and styles); since the SGxxx procedures post date the
  authoring of the principles.
- Whenever possible a treatment attribute map dataset should be used to keep symbols and colour schemes consistent across outputs, and where possible across individual subjects. This should be stored in the refdata area of HARP

#### 11.5. Appendix 5: Derived and Transformed Data

#### 11.5.1. **General**

#### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from Study Treatment Start Date:
- If the reference has both Dates and Times then the Study Day should be computed using the Datepart only
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Treatment Start Date → Study Day = Ref Date -Treatment Start Date
  - Ref Date ≥ Treatment Start Date → Study Day = Ref Date (Treatment Start Date) + 1

#### **Change from Baseline**

• The change from baseline will be calculated by subtracting the baseline values from the individual post-randomisation values.

#### 11.5.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Age will be computed relative to SCREENING visit (so outputs will match inclusion criteria definition of age at time subjects sign the informed consent form)

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / Height (m)<sup>2</sup>

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
   Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Since this is a single dose study duration of exposure outputs may not be displayed

#### **Extent of Exposure**

 Subjects who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.

#### 11.5.3. Safety

#### **ECG Parameters**

#### **RR Interval**

• IF RR interval (msec) is not provided directly, then RR can be derived as :

[1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### **Adverse Events**

#### **AE'S OF Special Interest**

No AE's of special interest have been defined for this study.

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - $\circ$  Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1
- Categorical lab results from Urinanalysis may be mapped to a common nomenclature for the purposes of producing summary tables (for example, but not limited to, "+", "Pos" and "Positive" may all be summarised under "Positive"). The medical monitor will advise on the mappings based upon the observed categories within each test and a listing of the actual mappings

#### **Laboratory Parameters**

applied to each lab test will be produced.

#### 11.5.4. **Efficacy**

#### **Transpulmonary Thermodilution**

#### **Predicted Body Weight**

 $BW_{\text{Pr}ed} = 50 + (0.91*(Height - 152.4))$ 

Males:  $Where...BW_{Pred}(kg), Height(cm)$ 

 $BW_{\text{Pr}ed} = 45.5 + (0.91 * (Height - 152.4))$ 

• Females:  $Where...BW_{Pred}(kg), Height(cm)$ 

## **Body Surface Area (DuBois formulae)**

 $BSA = 0.007184*Weight^{0.425}*Height^{0.725}$ 

Where...BSA(m²),Weight(kg),Height(cm)

#### **Predicted Body Surface Area**

 $PBSA = 0.007184 * BW_{\text{pr}_{ed}}^{0.425} * Height^{0.725}$ 

• Where... $PBSA(m^2)$ ,  $BW_{Pred}(kg)$ , Height(cm)

### "Indexing" of values using the (Absolute value) data entered into the eCRF

•  $CI = \frac{CO}{BSA}$ , where  $CI(L/\min/m^2)$ ,  $CO(L/\min) & BSA(m^2)$ 

•  $GEDI = \frac{GEDV}{BSA_{Pred}}$ , where  $GEDI(mL/m^2)$ , GEDV(mL) &  $BSA_{Pred}(m^2)$ 

•  $EVLWI = \frac{EVLW}{BW_{Pred}}$ , where EVLWI(mL/kg), EVLW(mL) &  $BW_{Pred}(kg)$ 

• SVRI = SVR \* BSA, where  $SVRI(\text{dyn * s * cm}^{-5} * \text{m}^2)$ ,  $SVR(\text{dyn * s * cm}^{-5}) \& BSA(\text{m}^2)$ 

Note: These alternative derivations may be used as a rough and ready check of the internal consistency of the parameters but small differences may occur due to rounding so they will not appear in any listings/outputs/analyses:

$$SVRI = \frac{(MAP - CVP)}{CI} * 80 \text{ and } SVR = 80 * \frac{(MAP - CVP)}{CO}.$$

## Recovering the Absolute value from the "Indexed" value

• CO = CI \* BSA, where  $CI(L/min/m^2)$ ,  $CO(L/min) & BSA(m^2)$ 

•  $GEDV = GEDI * BSA_{Pred}$ , where  $GEDI(mL/m^2)$ ,  $GEDV(mL) \& BSA_{Pred}(m^2)$ 

•  $EVLW = EVLWI * BW_{Pred}$ , where EVLWI(mL/kg),  $EVLW(mL) & BW_{Pred}(kg)$ 

•  $SVR = \frac{SVRI}{BSA}$ , where  $SVRI(\text{dyn *s *cm}^{-5} * \text{m}^2)$ ,  $SVR(\text{dyn *s *cm}^{-5}) \& BSA(\text{m}^2)$ 

#### **Secondary Endpoints**

#### Calculation of PaO<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> and SpO<sub>2</sub>/F<sub>i</sub>O<sub>2</sub>

- The P<sub>a</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> endpoint will be calculated when patients are intubated and have an arterial line present. Prior to computing the ratio the P<sub>a</sub>O<sub>2</sub> will be converted from kPa units to mmHg using the conversion rate 1/0.133 and F<sub>i</sub>O<sub>2</sub> will be expressed as a proportion and not a percentage.
- S<sub>p</sub>O<sub>2</sub>/ F<sub>i</sub>O<sub>2</sub> will be calculated as a ratio of percentages, where patients are no longer intubated and the arterial line has been removed.

#### **SOFA (Sequential Organ Failure Assessment)**

Table below (SOFA Score points allocation algorithm) details how points should be allocated to each SOFA component. Prior to analysis the CONMEDS dataset will be reviewed by the medical monitor who will flag observations which are adrenergic agents and vasopressors. Adrenergic agents that do not appear in Vincent (1996), and for which a highest dose has been recorded, will be assigned a SOFA score of 2.

Zero points are assigned if none of the points scoring criteria are met. If any of the information required to derive an individual SOFA component score is missing or cannot be obtained then that component score will be set to a missing value.

Derivation of Baseline SOFA value: Not all required SOFA components are being measured on Day 1. When component data are available they should be used (Day 1 Pre-dose: lab samples). Since each subject is about to undergo surgery they will be assumed to have been sufficiently fit to satisfy the following assumptions: Respiration, Central Nervous System and Cardiovascular component scores fixed at 0 and Renal score derived solely from Creatinine Pre-dose lab result.

#### SOFA Score points allocation algorithm

| SOFA Score /<br>Variable (x) | 0 | 1 | 2 | 3 | 4 |
|---|---|---|---|---|---|
| Respiration:<br>P <sub>a</sub> O <sub>2</sub> /F <sub>i</sub> O <sub>2</sub><br>(mmHG) | x ≥ 400 | 300 ≤ x < 400 | 200 ≤ x < 300 | $100 \le x < 200$ With Respiratory sup (Note: if $P_aO_2/F_iO_2$ in subject not on respirators score of 2 should be | these categories but atory support then a |
| Coagulation: Platelets (10^3 / mm^3) | x ≥ 150 | 100 ≤ x<br>< 150 | 50 ≤ x < 100 | 20 ≤ x < 50 | x < 20 |
| Liver:<br>Bilirubin<br>(µmol/L) | x < 20 | 20 ≤ x <<br>33 | 33 ≤ x < 102 | 102 ≤ x < 204 | x ≥ 204 |

| Secondary Endp | Secondary Endpoints | | | | |
|---|---|---|---|---|---|
| Calculation of P <sub>a</sub> O <sub>2</sub> /F <sub>i</sub> O <sub>2</sub> and S <sub>p</sub> O <sub>2</sub> /F <sub>i</sub> O <sub>2</sub> | | | | | |
| Cardiovascular: Hypotension (Adrenergic agents administered for at least one hour; doses are in µg/kg/min) | Mean<br>Arterial<br>Pressure<br>≥ 70<br>mmHg | Mean<br>Arterial<br>Pressure<br>< 70<br>mmHg | Dopamine≤5.0 (µg/kg/min) or any dose of: Dobutamine Or any dose of an adrenergic agent not listed here or in Vincent(1996) | Dopamine 5.1-15.0<br>(µg/kg/min)<br>or Epinephrine≤0.1<br>or<br>Norepinephrine≤0.1 | Dopamine > 15.0<br>(µg/kg/min)<br>or Epinephrine>0.1<br>or<br>Norepinephrine>0.1 |
| Central Nervous System: Glasgow Coma Score | x ≥ 15 | 13 ≤ x ≤<br>14 | 10 ≤ x ≤ 12 | $6 \le x \le 9$ | x < 6 |
| Renal:<br>Creatinine<br>(μmol/L) | x ≤ 110 | 110 < x<br>≤ 170 | 170 < x ≤ 300 | $300 < x \le 440$ [Or Urine output < 500 mL/day] | x > 440 [Or Urine output < 200 mL/day] |

#### **Calculation of Oxygenation Index**

The oxygenation index will be calculated as:

Oxygenation Index (%) = 
$$\frac{FiO2 * Paw}{PaO2}$$

where Mean Airway Pressure (Paw) and PaO2 are measured in mmHg and FiO2 is entered as a % and not a proportion.

Conversion of Paw units from  $cmH_2O$  to mmHg will be performed using the ratio 1  $cmH_2O$  = 1/1.36 mmHg.

Conversion of PaO2 units from kPa to mmHg will be performed using the ratio 1 kPa = 1/0.133 mmHg.

#### 11.5.5. Pharmacokinetic

#### **Drug Concentration in BAL**

#### **Derivation of BAL/ELF Drug Concentration Data**

 Urea concentration data will be used to calculate the dilution effect of the lavage which is used to extract the epithelial lining fluid (ELF) from the lung. A correction for dilution will be applied to BAL drug concentrations as follows:

Epithelial Lining Fluid (ELF) Drug Concentration (pg/mL) = BAL Drug Concentration (pg/mL) x Dilution Factor

#### **Drug Concentration in BAL**

where

Dilution Factor= Plasma Urea / BAL Urea

Plasma urea is measured from the plasma samples planned to be taken at a similar time to the BAL sample time.

 Additionally the Volume of ELF in BAL fluid and the Total Drug in BAL fluid will be calculated as follows:

*Volume of ELF in BAL Fluid (mL) = BAL Fluid Volume (mL)/Dilution Factor* 

Total Drug in BAL (pg) = BAL Drug Concentration  $(pg/mL) \times BAL$  Volume (mL)

#### 11.5.6. Pharmacodynamic (Biomarker)

#### Pharmacodynamic (Biomarker)

#### **Biomarkers**

- In general, it is assumed that biomarker endpoints will require variance stabilising transformations, such as taking a log<sub>e</sub> transformation prior to analysis (and that summary statistics appropriate to log<sub>e</sub> normally distributed data will apply for all summaries). However, this assumption will be considered for each endpoint individually prior to the generation of summary tables or statistical analysis, and if deemed more appropriate, a log<sub>e</sub> transformation will not be applied, or non-parametric methods may be employed.
- If transformations are used then the results will be reported on the back-transformed scale unless otherwise stated.

#### 11.5.7. Exploratory Endpoints

#### **Exploratory Endpoints**

#### Predicting missing P<sub>a</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> using S<sub>p</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub>

Rice (2007) describe the following linear model to predict S<sub>p</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> using available P<sub>a</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> values.

$$S_pO_2/F_iO_2 = 64 + (0.84 * P_aO_2/F_iO_2)$$

For exploratory purposes (i.e. taking the very strong steps of disregarding the uncertainty of the
original linear regression parameter estimates and the inverse estimation aspect of the
proposal) the formulae will be re-arranged and used to impute missing P<sub>a</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> values when a
corresponding S<sub>p</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> value is available (e.g. when the arterial line has been removed):

 $P_aO_2/F_iO_2$  (Imputed) =  $(S_pO_2/F_iO_2 - 64) / 0.84$  when  $P_aO_2/F_iO_2$  is missing &  $S_pO_2/F_iO_2$  available  $P_aO_2/F_iO_2$  (Imputed) =  $P_aO_2/F_iO_2$  when  $P_aO_2/F_iO_2$  is non-missing

 $P_aO_2/F_iO_2$  (Imputed) = Missing in all other cases

## 11.6. Appendix 6: Premature Withdrawals & Handling of Missing Data

## 11.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as one who has completed all phases of the study including the follow-up visit.</li> <li>Withdrawn subjects may be replaced in the study, but any replacement would take the next available randomisation number and not be guaranteed to receive the same treatment as the withdrawn subject.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> <li>In the event that the study is prematurely discontinued, all available data will be listed and a review carried out by the study team to assess which statistical</li> </ul> |
| Surgery | <ul> <li>analyses are still considered appropriate.</li> <li>In some cases, a subject may be randomised to the study and surgery initiated, but subsequently halted due to a decision being made that the case is in fact inoperable. In the event of an open and shut case subjects will be withdrawn from the study by the investigator. As the subjects will have received a dose of study dose prior to surgery, every effort should be made to complete as many of the Day 28 follow-up assessments and procedures as possible, prior to hospital discharge.</li> </ul> |

## 11.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> </li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| PVPI and<br>EVLWI | <ul> <li>In the case that PVPI and EVLWI are missing and cannot be derived using the<br/>methods described in Section 11.5.4, they will remain missing.</li> </ul> |
| PK | Urea data: Below the Lower Limit of Quantification (LLQ) values will be imputed with the relevant (BAL fluid) LLQ divided by 2 for the purpose of deriving the Dilution Factor. |
| | <ul> <li>Plasma concentrations: Refer to Section 11.5.3 or for further guidance see the<br/>PK Guidance document, GUI_00000051487, and the DB/CPMS guidelines</li> </ul> |

| Element | Reporting Detail |
|---|---|
| | 'Standards for the Handling of NQ impacted PK Parameters' for more information. |
| Biomarkers | Values below LLQ will be set as LLQ/2 |
| | Values above the upper limit of quantification (ULQ) will be set as ULQ |
| | <ul> <li>Imputed values will be used for the purposes of the computation of change from<br/>baseline and for summaries, plots and analysis, if deemed applicable.</li> </ul> |
| | Number of data imputed will be highlighted in the summaries and listings will report the values as below LLQ or above ULQ. |
| | If multiple LLQ's and ULQ's are available per assay (i.e. multiple runs with different standard curves are utilised) then the LLQ and/or ULQ value used for the above purposes shall be the minimum of the available LLQs and/or the maximum of the BLQ's. |
| | If more than a third of observations are below LLQ or above ULQ then no imputation will be performed for that subject. |

## 11.6.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 3: Treatment States and Phases.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> <li>Start or end dates which are completely missing (i.e. no year specified) will remain missing, with no imputation applied.</li> </ul> |
| Surgical<br>Procedures<br>/ Biomarker<br>samples<br>(Serum and<br>BAL) | <ul> <li>If the date/time of an event occurring during the surgical procedures is unknown then it shall remain missing. Any associated data values may be listed using the timeslicing keys to determine the chronological ordering.</li> <li>Since each surgical procedure is bespoke it is not possible to impute a date/time, although depending upon the analysis and endpoint the planned time (or the time of a proximal event) may be sufficiently accurate to be used. Otherwise the data point may be omitted from the analysis and/or form part of a sensitivity analysis (e.g. Subject PPD has unknown BAL sample date/time and the proposed PK modelling may be sensitive to any assumed/imputed value, so the observation may be dropped).</li> </ul> |

## 11.6.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

## 11.6.2.3. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail | | |
|---|---|---|---|
| SOFA | <ul> <li>If any of the information required to derive an individual SOFA component sis missing or cannot be obtained then that component score will be set to a missing value.</li> <li>However, in the case of missing P<sub>a</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> ratios; S<sub>p</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> ratios and the following corresponding thresholds for S<sub>p</sub>O<sub>2</sub>/F<sub>i</sub>O<sub>2</sub> may be used (Pandharipa 2009):</li> </ul> | | |
| | SOFA Respiratory<br>Score | $P_aO_2/F_iO_2$ | S <sub>p</sub> O <sub>2/</sub> F <sub>i</sub> O <sub>2</sub> |
| | 1 | < 400 | < 512 |
| | 2 | < 300 | < 357 |
| | 3 | < 200 | < 214 |
| | 4 | < 100 | < 89 |
| | causes then those comp response at that time poi | onent scores may be popul<br>nt on the corresponding tre<br>th requires imputation linea | ne to procedural / operational lated with the average eatment arm. Alternatively if r interpolation using the Day |

## 11.7. Appendix 7: Values of Potential Clinical Importance

## 11.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | 0.3 | 0.54 |
| Hematocrit | Ratio of 1 | Female | 0.3 | 0.54 |
| | /1 | Male | 90 | 180 |
| Hemoglobin | g/L | Female | 90 | 180 |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.6 | 3.0 |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | 20 |
| Platelet Count | x109/ L | | 100 | 600 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

Note: For the following lab tests the corresponding normal ranges should be used as the PCI range: Reticulocyte Count, RBC Count, MCV, MCH, MCHC, Monocytes, Eosinophils and Basophils

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | mmol/L | | 25 | 60 |
| Calcium | mmol/L | | 1.8 | 2.75 |
| Creatinine | mmol/L | | 30 | 160 |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 2.5 | 5.5 |
| Sodium | mmol/L | | 120 | 160 |
| Total CO2 | mmol/L | | 16 | 35 |
| BUN | mmol/L | | 3 | 15 |
| Chloride | | | no PCI required for this study | no PCI required for this study |

| Liver Function | | | |
|---|---|---|---|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 4x ULN |
| AST/SGOT | U/L | High | ≥ 4x ULN |
| AlkPhos | U/L | High | ≥ 4x ULN |
| T Bilirubin (Note: Direct Bilirubin PCI not required for this study) | µmol/L | High | ≥ 2xULN |
| T. Bilirubin + ALT | µmol/L<br>U/L | High | 2xULN T. Bilirubin<br>+<br>≥ 4x ULN ALT |

## 11.7.2. ECG

| ECG Parameter | Units | Clinical Con | cern Range |
|--------------------------------------|-------|--------------|------------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QT Interval | msec | ≥ 300 | ≤ 500 |
| Absolute QTc Interval (QTcB or QTcF) | msec | ≥ 300 | ≤ 450 |
| Absolute PR Interval | msec | < 90 | > 200 |
| Absolute QRS Interval | msec | < 70 | > 120 |
| Absolute RR Interval | msec | < 375 | > 1700 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | > 60 |

## 11.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |


#### TFR116341

| Vital Sign Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| (Change from Baseline) | | Decreases of magnitude | Increases of magnitude |
| Systolic Blood Pressure | mmHg | >50 | >50 |
| Diastolic Blood Pressure | mmHg | >30 | >30 |
| Heart Rate | bpm | >50 | >50 |

## 11.8. Appendix 8: Biomarker Details

**Note:** These are the planned biomarkers at time of RAP writing. Additional items may be added or existing ones removed.

| Parameters (BICATCD Code) | Sample | Unit | LLQ | ULQ |
|---|---|---|---|---|
| Target Engagement * | | | | |
| Free sTNFR1 | Serum & BAL | | | |
| Total sTNFR1 | Serum & BAL | | | |
| Complex TNFR1 | Serum & BAL | | | |
| Pro-Inflammatory Biomarkers * | | | | |
| TNFa | BAL | | | |
| IL-6 | Serum & BAL | | | |
| IL-8 | Serum & BAL | | | |
| IL-1b | BAL | | | |
| MCP-1 | BAL | | | |
| Anti-Inflammatory Biomarkers * | | | | • |
| CRP (Reactive Protein C) <sup>△</sup> | Plasma & BAL | | | |
| IL1-ra | BAL | | | |
| IL-10 | BAL | | | |
| Protein Permeability Index * | | | | |
| Total Protein in BAL | BAL | | | |
| Total Protein in Plasma | Plasma | | | |
| Total Protein Ratio (Ratio is derived from BAL and Plasma values) | Plasma & BAL | | | |
| Markers of Epithelial Cell Injury | | | | |
| Surfactant Protein D | Serum & BAL | | | |
| RAGE (Receptor for Advanced Glycation End products)* | Serum & BAL | | | |
| Club Cell 16 (also known as CC10 and CC16) | Serum & BAL | | | |
| Markers of Endothelial Injury | | | | |
| vWF | Serum & BAL | | | |
| sICAM-1* | Serum & BAL | | | |
| Markers of Neutrophil Activation* | | | | |
| MPO | Serum & BAL | | | |


TFR116341

#### NOTE:

- \* Expect biomarker parameters to be increased in oesophagectomy patients.
- Serum sampling times: Day 1 Prior to Surgery, Day 1 On Completion of Surgery, Day 2, Day 3, Day 4 and Day 8/Day of Discharge.
- BAL sampling time: Day 1 On Completion of Surgery.
- N/A = No ranges are normally provided for parameters.
- Display biomarkers in the order presented in the Table, and use Functional Category labels provided to further group them.
- $\Delta$  = Measured in plasma as part of Clinical Chemistry Labs so may have different sampling scheme and require appropriate adjustments to displays and/or models

## 11.9. Appendix 9: Examination of Covariates, Subgroups & Other Strata

#### 11.9.1. Handling of Covariates, Subgroups & Other Strata

- The randomisation is stratified by Centre (site). However, the number of subjects recruited at a site may be small (it is conceivable that a site may not recruit sufficient subjects to have an individual from each of the four treatment arms). Therefore the statistical models should include a fixed categorical effect for centre by intent, but this centre term may be dropped. Alternatively low recruiting centres may be pooled by NHS region, or another suitable characteristic (e.g. shared research fellow) if deemed appropriate.
- The following is a list of covariates that may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses (such outputs would take the next available number).
- Additional covariates of clinical interest may also be considered.
- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined prior to unblinding the trial.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

| Category | Potential Covariates and / or Subgroups |
|---|---|
| Randomisation strata | • Centre (site) |
| | Research fellow assisting with study procedures |
| | NHS authority the site belongs to (a potential mechanism to cluster centres that may behave similarly within the UK) |
| Subject characteristics | Gender |
| | • Age |
| | Race / Ethnicity |
| | Height / Weight / BMI |
| Medical History | Prior Oesophageal Chemotherapy |
| | Smoking history |
| | Medical history |
| Surgical Procedure | Duration of Surgery |
| | Duration of One Lung Ventilation |
| | Duration of anaesthesia |
| | Inotrope usage |


#### TFR116341

| Category | Potential Covariates and / or Subgroups |
|---|---|
| Immunogenicity | Did subject develop serum anti-GSK2862277<br>antibodies |
| Clinical Outcomes / Resource<br>Utilisation | Did subject develop ARDS during study |
| | Vent free days |
| | ICU length of stay |
| | Hospital length of stay |
| | Organ failure free days |

#### 11.10. Appendix 10: PVPI and EVLW – Supplementary Information

#### 11.10.1. Data derivations to be performed by GSK

When appropriate, "Indexed" versions of the parameters will be derived as per Section 11.5.4.

In the event that the sites did not configure their PiCCO machine to display the Absolute parameter sets and the only information available is the Indexed version of a PiCCO parameter then the Absolute value will be recovered from the indexed version using the appropriate equation from Section 11.5.4.

## 11.10.2. Theoretical Underpinning of Transpulmonary Thermodilution Measurements

This section briefly describes the theory behind the PiCCO machine. Not all of the items described are provided / outputted by the machine (see Table 13 for the parameters databased via the eCRF).

The transpulmonary thermodilution provides the measurement of cardiac output (CO), the global end-diastolic volume (GEDV) and intra-thoracic blood volume (ITBV) by passing a thermal indicator (cold solution) through the right heart, lungs and left heart and measuring the temperature changes at a known distance downstream, typically in the femoral artery. The ITBV (a measure of all the blood contained within the chest), is measured by the GEDV, which is the sum of the end-diastolic volumes of all heart chambers, and pulmonary blood volume (PBV).

Figure 3 Transpulmonary Thermodilution Curve showing mean transit time and downslope decay time (DSt) of the slope. The time point (A) represents the time of injection. The product of cardiac output and MTt equals the intrathoracic thermal volume. Multiplication of the cardiac output and the DSt equals the pulmonary thermal volume (PTV).


The product of the CO and the mean transit time (MTt) of the thermal indicator, is the intrathoracic thermal volume (ITTV = ITBV + EVLW), i.e., the distribution volume of the thermal indicator. The product of the CO and exponential downslope time (DSt) is the pulmonary thermal volume (PTV). The GEDV is calculated as the difference between the intrathoracic and pulmonary thermal volume (GEDV = ITTV – PTV). (See Figure 4.)

Figure 4 Determination of GEDV by transpulmonary thermodilution. The ITTV describes the distribution volume of the thermal indicator, including the volumes in the right atrium (RA), right ventricle (RV), left atrium and left ventricle (LV).



Intrathoracic blood volume (ITBV) is calculated from the GEDV by assuming a relationship of a constant ratio of 1.25. (ITBV =  $1.25 \times GEDV$ ). This ratio allows the calculation of ITBV and consequently the calculation of the EVLW (ITTV – ITBV).

PVPI is the ratio between EVLW and the pulmonary blood volume (PBV), which is deduced from the difference between the PTV and EVLW (PBV = PTV - EVLW).

Table 13 Endpoints and abbreviations used in Transpulmonary Thermodilution

| Timeframe | Grouping | Abbreviation / Item | Databased | Description |
|---|---|---|---|---|
| Continuous <sup>1</sup> | | | | |
| | Continuous | Heart Rate | Yes | Heart Rate |
| | cardiac output | AP | Yes | Arterial Pressures [Systolic<br>Blood Pressure / Diastolic Blood<br>Pressure] |
| | | CVP | Yes | Central Venous Pressure<br>[manually entered into PiCCO<br>machine] |
| | | CPO | No | Cardiac Power Output |
| | | CPI | No | Cardiac Power Index |
| | Calibrated Continuous cardiac output | PCCO | No | Pulse Contour Cardiac Output:<br>Calculated beat by beat as<br>Stroke Volume * Heart Rate |
| | | PCCI | No | Pulse Contour Cardiac Index |
| | Stroke Volume | SV | No | Stroke Volume |
| | | SVI | No | Stroke Volume Index: <b>Assumed</b> to be Stroke Volume indexed by predicted body surface area |
| | | 1 | | |
| | Afterload | SVR | Yes | Systematic Vascular Resistance: Determinant of afterload. Computed as $\frac{MAP-CVP}{Flow(CO)}*80 \text{ where}$ |
| | | | | Flow(CO)=Pressure/Resistance. Vasoconstriction implied if Flow(CO) is decreasing and Vasodilation implied if Flow(CO) is increasing provided pressure is constant |
| | | SVRI | No | Systematic Vascular Resistance<br>Index: SVR * BSA (Body<br>Surface Area - DuBois) |
| | | MAP | Yes | Mean Arterial Pressure |

| Timeframe | Grouping | Abbreviation / Item | Databased | Description |
|---|---|---|---|---|
| | Volume<br>responsiveness | SVV | Yes | Stroke Volume Variation: Variation in Stroke Volume over the breathing cycle for a specific time frame (only available in mechanically ventilated patients in sinus rhythm) |
| | | PPV | No | Pulse Pressure Variation: Variation in Pulse Pressure over the breathing cycle for a specific time frame (only available in mechanically ventilated patients in sinus rhythm) |
| | Contractility | dPmax | No | Left contractility paramater |
| | Contractility | urillax | INU | Len contractinty paramater |
| Discontinuous | Thermodilution<br>Cardiac Output | CO (also<br>known as<br>CO <sub>TDa</sub> ) | Yes<br>(triplicates) | Cardiac Output (thermodilution): Volume of blood pumped by heart in one minute. |
| | | CI | No | Cardiac Index: Cardiac Output indexed by body surface area (DuBois) |
| | Volumetric<br>Preload | GEDV | Yes<br>(triplicates) | Global End Diastolic Volume:<br>Filling volume of all four heart<br>chambers |
| | | GEDI | No | Global End Diastolic Volume<br>Index: GEDV indexed to<br>predicted body surface area |
| | Contractility | GEF | Yes | Global Ejection Fraction |
| | | CFI | No | Cardiac Function Index: Measure of contractility (performance of cardiac muscle). Ratio of flow and preload: CFI = CO / GEDV |
| | Pulmonary<br>Edema | EVLW (also<br>known as<br>ELW) | Yes<br>(triplicates) | Extra Vascular Lung Water:<br>Includes intra-cellular, interstitial<br>and intra-alveolar water (not<br>pleural effusion) |
| | | EVLWI (also<br>known as<br>ELWI) | No | Extra Vascular Lung Water Index: EVLW indexed to predicted body weight |

| Timeframe | Grouping | Abbreviation | Databased | Description |
|---|---|---|---|---|
| | | / Item<br>PVPI | Yes | Pulmonary Vascular Permeability Index: EVLW indexed to Pulmonary Blood Volume |
| | Used internally | ITBV | No | Intra-thoracic Blood Volume |
| | by the PiCCO | PBV | No | Pulmonary blood volume |
| | machine | PTV | No | Pulmonary thermal volume |
| | | MTt | No | Mean transit time |
| | | DSt | No | Downslope decay time |
| | | ITTV | No | Intrathoracic thermal volume |
| | | LAV / RAV | No | Left / Right atrium Volume |
| | | LVV / RVV | No | Left / Right ventricle Volume |
| Constant | Information / Demographics | BSA | No | Body Surface Area (DuBois): Manually derived from observed weight and height |
| | | PBW | No | Predicted Body Weight |
| | | PBSA | No | Predicted Body Surface Area: Derived using same approach as DuBois but uses Predicted body weight instead of observed weight |
| | | Arterial Line<br>Used | Yes | Typically Femoral (Brachial is the other option) |

A snapshot of the values for the continuous measurements would be taken when the 3x
 Thermodilutions are performed

# 11.11. Appendix 11: Model Checking and Diagnostics for Statistical Analyses

#### 11.11.1. Bayesian Analyses (SAS Proc MCMC)

- The following points are for guidance and illustration only and do not guarantee a successful model convergence. They cannot cover all eventualities and do not remove the requirement to do what is best for the specific set of observed data being modelled.
- Unless otherwise stated, data collected at screening and at unscheduled time points will not be included in the statistical analyses, i.e., only planned/scheduled post-screening data will be included.
- All credible intervals reported will be equal tail, unless otherwise specified.
- Convergence for the parameters in the model needs to be verified.
- The randomization seed used in PROC MCMC should itself be generated with an element of randomness but there is no need to formally document this process (e.g. using Excel function RANDBETWEEN [1,9999999] and copying the result into the SAS code)
- Unless the parameter is a flag variable (e.g. taking binary values of 1 or 0) the medians of the posterior distribution should be used.
- Warnings/Erros in the SAS log regarding flag variables may be safely discounted
- All effects will be entered on the same PARMS statement initially. If necessary to aid model convergence parameters may be split across several PARMS lines.
- Centring of continuous covariates will take place at the input dataset stage, using only individuals who contribute usable data to the model fitting process.
- Individuals with missing covariates would be dropped from the model fitting process (alternative imputation strategies may be explored if required, e.g. substituting the covariate mean for a missing value)
- Bespoke conjugate samplers (functions that can be called from within PROC MCMC)
  may be used to improve the computational performance and reduce the computational
  overheads. If such an approach is used it may require different parameterisations /
  prior specification but it should be set up act commensurate to the approaches
  described.

#### 11.11.1.1. Prior Distributions

Unless otherwise specified, the following will be the default approach to selecting prior distributions:

- Non-informative priors of the form Normal(0, Var=1E6) will be assigned to each fixed-effect parameter in the proposed statistical model.
- Non-informative inverse-gamma priors of the form IG(a=2.001,b=0.001) will be used for scale parameters (variances). If these parameters do not lead to convergence than choose "a" small and "b" smaller than the expected standard

deviation (the expected standard deviation can be obtained from empirical estimates or by fitting the model using likelihood approaches such as in PROC MIXED).

- For scale parameters (variances) that may take values close to zero a non-informative prior of the form Uniform(0, XXX) may be assigned for the standard deviation (SD) in place of the inverse gamma, where XXX is a suitably chosen range that covers clinically plausible values for the SD.
- For repeated measures models, non-informative Inverse-Wishart priors of the form  $IW(\upsilon, \Sigma)$  will be assigned for the unstructured VCV. The parameter  $\upsilon$  represents the dimension of VCV (number of rows or columns) and the matrix  $\Sigma$  is an identity matrix of the same dimension as VCV.
  - o If there are issues with these distribution parameters then the identity version of  $\Sigma$  may be replaced with a diagonal matrix that uses best guesses for the residual variance at each repeated measure timepoint (or empirical estimates or the residual estimate from fitting likelihood based models using PROC MIXED). This only needs to be of the correct order of magnitude.
  - O Alternatively, a Spatial power (with planned times as the "distances") for the VCV may be explored. The prior for the correlation parameter  $\rho$  is Uniform[-1,1], whereas the variance parameter  $\sigma^2$  is assumed to follow the IG(a=2.001,b=0.001) prior distribution.

It is good practice to ensure that each prior distribution is visualized to ensure it appears sensible, i.e., that it allows parameter values that generate clinically plausible response values and that it is truly non-informative over the region of the likelihood function where the data lies.

#### Note:

• The Gamma(a, b) density function takes the form

$$p(u) = \frac{b(bu)^{a-1}e^{-bu}}{\Gamma(a)}, u > 0$$

The mean is a/b and the variance is  $a/b^2$ .

• The IG(a, b) density function takes the form

$$p(u) = \frac{b^a u^{-(a+1)} e^{-b/u}}{\Gamma(a)}, u > 0$$

The mode is b/(a+1), the mean is b/(a-1), if a>1, and the variance is  $b^2/[(a-1)^2(a-2)]$ , if a>2.

• There is no requirement to formally report the prior visualisation outputs.

#### 11.11.1.2. Initial Values

Unless otherwise specified, initial parameter values of zero will be used for the fixed-effect parameters. For remaining model parameters initial values may be drawn at random from their respected prior distribution. If convergence of the Markov chain Monte Carlo (MCMC) algorithm is problematic then alternative estimates may be used (for example, these could be based on maximum likelihood estimates, or by setting any "intercept" parameter to lie roughly in the region of the observed data values).

#### 11.11.1.3. Convergence Diagnostics

To be able to perform Bayesian inference using MCMC simulations the samples for all the parameters in the model need to be obtained from the corresponding target posterior distribution. To ensure that this is the case the following is a list of convergence diagnostics that can be applied for each parameter:

Comparing MCSE vs posterior standard deviation:

- The Monte Carlo Standard Errors (MCSE) should be compared with the standard deviation of the posterior distribution (SD) to ensure that only a fraction of the posterior variability is due to the simulation, i.e., the ratio MCSE/SD should be as small as possible, typically close to 0.01.
- Adequate values for the number of MCMC samples / thinning / number of burn-in samples should be chosen to ensure that the ratio MCSE/SD for the key parameters in the model is approximately 0.01 (key parameters are those associated with treatment, or pre-specified comparisons of interest).
- For other model parameters, try to get the MCSE/SD values as close to 0.01 as possible, but if there is significant autocorrelation then values below 0.05 would be considered acceptable.
- In addition, if possible, the number of tuning units and maximum number of tuning iterations may be increased to find a better proposal distribution for the model parameters, which in turn may reduce the MCSE/SD ratio.
- Where possible the code should be written to allow the SAS compiler to identify and make use of conjugacy, since this can greatly reduce the corresponding MCSE/SD ratio.
- Models selected with MCSE/SD values > 0.01 would need a brief remark/justification added to the CSR to clarify why it was not possible to reach the target and why it is believed the subsequent model still has utility from an inference perspective.

#### Geweke diagnostics:

- The Geweke diagnostic test checks whether the mean estimates have converged by comparing means from the early and latter part of the Markov chain using a zscore t-test.
- Large absolute values of the z-score statistic indicate rejection of the null hypothesis of no difference between the mean estimates obtained from the early and latter parts of the chain.

#### Diagnostic plots and visual inspection:

- Trace plots of samples versus the simulation index can used to assess some aspects of convergence. The centre of the chain should appear stable with very small fluctuations, i.e., the distribution of points should not change as the chain progresses and the posterior mean and variance are relatively constant.
- Autocorrelation plots can be used to assess degree of autocorrelation (should decline rapidly and show no oscillation patterns).
- The posterior density should look reasonable for each parameter (e.g. for posterior parameters expected to follow a normal distribution, the density plot should not appear bi-modal, but for parameters acting as binary flags, then bi-modal is acceptable).
- Examination of correlation structures between relevant posterior parameters should be used to provide information about what potential issues may be and also what corrective action(s) may be worthwhile attempting (scatterplots of the samples from the posterior distributions of the parameters).

Convergence for all the parameters in the model needs to be verified.

## 11.11.1.4. Additional Model Checking (optional at the discretion of the study statistician)

Additional model checking can be performed using the posterior predictive distribution.

- For each observation generate as many expected values from the posterior predictive distribution as the number of MCMC samples.
- Residuals for each observation are obtained by subtracting the expected values from the observed values.
- For each subject calculate an average residual and an average expected value.
- Model fitting can be checked by looking for patterns when plotting the average residual versus the average predicted value as in a maximum likelihood estimation setting.

When non-informative priors are used and there is only a small amount of missing data a faster/easier alternative to the posterior predictive distribution model checking would be to fit the equivalent model using a frequentist approach (e.g. in SAS PROC MIXED) and utilise the built in diagnostic tools.

#### 11.11.1.5. Possible corrective actions for non-converging MCMC models

Possible corrective actions include but are not limited to

- Moving parameters (or combinations of parameters) onto separate PARMS statements (to form blocks that are updated independently in the MCMC algorithms)
- Increasing the number of MCMC draws from the posterior distributions
- Increasing the length of the burn in period
- Increasing the thinning parameter (to reduce the autocorrelation)
- Centring covariates (to reduce correlations between the posterior parameters)
- Re-parameterising the model (e.g. using log-normal prior distributions to stop values being sampled that are below zero)
- Re-scaling the parameters (e.g. if one parameter takes values orders of magnitudes different to the other model parameters then dividing it by a suitable constant but back transforming the rescaled parameter prior to its use in any subsequent manipulations)
- Visualising the likelihood function of the dataset to determine if there are more appropriate starting estimates (or profiled versions of the likelihood for subsets of model parameters where difficulties are being encountered if it is a high dimensionality problem)
- Consulting with internal GSK experts to resolve the issues

#### 11.11.2. Mixed modelling assumptions (SAS Proc MIXED)

The following applies to statistical models fitted using SAS Proc MIXED:

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.

- o In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
- Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the (studentised) residuals and a plot of the (studentised) residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

If there are any departures from the distributional assumptions, alternative models may be explored using appropriate transformed data.

# 11.12. Appendix 12: Details of Simulation exercise that produced operational characteristics used in the protocol

This section describes in detail how simulations were used to choose the cut-off points and probability thresholds included in the protocol decision rules and how simulations were used to assess the operating characteristics of the target sample size (40 per arm).

#### 11.12.1. Simulations supporting interim analysis 2

This section is divided into a broad overview of the strategy and additional sub-sections containing further detail on specific topics

- Feasibility considerations limited maximum number of subjects to 80.
- Assumption of 2x endpoints per subject available at 2x time points (pre-surgery (baseline) and immediately post surgery). PVPI was assumed to require Ln (natural logarithm) transformation. No covariate adjustments were allowed in these simulations, but the actual IA2 analysis may incorporate covariate adjustments (e.g. for centre effects)
- Goal of simulation strategy was to optimise the timing and frequency of interim analyses and the decision rules therein.
- Various scenarios of possible GSK2862277 treatment effects; expressed as
  differences from the placebo means were evaluated in conjunction with different IA2
  recruitment targets (hypothetical placebo means assumed to be the same as the
  baseline adjusted values estimated from the BALTI dataset (Perkins, 2014)). Table 20
  details the possible treatment effects evaluated. Table 16 details the potential IA2
  timings and thresholds evaluated.
- For each scenario the simulation process is split into "Outer" and "Inner" loops. Differences over the outer loops explore the impact of the "information content" within data available at the time of IA2. Differences over the inner loops explore the impact of the decision criteria and rules for a given set of "observed" interim data. In practice there will only be one set of observed study data. The *a priori* expectation was that the later the timing of IA2 (with respect to the possible 80 subjects) the more consistent the information content would be across outer loops and, therefore, less variability between outer loop outcomes.
- Logistics of implementing these complex simulations sometimes dictated the approaches taken (e.g. using conjugacy rather than MCMC simulations to enumerate distributions).
- Outer loops: For efficiency 10,000 sets of individual subject level data for the maximum possible study size are generated for each scenario (i.e. 80 subjects per dataset). Repeatedly subsetting these 80 subjects and creating summary statistics from each subsample allows multiple IA2 timings to be evaluated without constantly

having to re-simulate subject level data. Sufficient summary statistics were created using the first 12 subjects (6 per arm.), the first 14 subjects (7 p.a.), etc, through to 78 subjects (39 p.a.) in increments of 2 subjects. Thus, each of the 10,000 sets has 34 associated sets of summary statistics. Operating characteristics of potential IA2 timings (e.g. after 15 subjects per arm) were evaluated by selecting the corresponding 10,000 sets of associated summary statistics and putting each of them through the inner loop process. These are the summary statistics (and dimensions) produced which act as inputs to the inner loop process:

- Placebo Mean Vector [2x1], Variance Covariance matrix [2x2] and Correlation matrix [2x2]
- o Number of subjects on Placebo [scalar]
- Active Mean Vector [2x1] Variance Covariance matrix [2x2] and Correlation matrix [2x2]
- Number of subjects on Active [scalar]

Note: This step may be introducing some form of correlation between the simulation runs because the same subject level data is being used repeatedly (e.g. the summary statistics for 6 and 7 subjects per arm will only differ due to the 1x additional subject). Unfortunately computational run time, the number of scenarios and the protocol development timeline prohibited completely independent subject simulations to create the various summary statistics used as inputs to the inner loops.

• <u>Inner loops</u>: The starting assumption for each inner loop was that the "observed" data at the time of the interim have been used to derive multivariate sample summary statistics (computed separately per treatment arm). By using the VCV matrix from the Baseline adjusted BALTI dataset and the baseline adjusted Placebo means in the scenarios simulation of separate baseline data points was not necessary for the inner loops in this exercise.

Initially these summary statistics are combined with a set of non-informative priors to produce the hyperparameters of a multivariate normal distribution for predicting an individual subjects future response (described for the placebo treatment arm; analogous results for the active arm):

Mechanism for updating hyperparameters to simulate remaining

| | | | subjects (Pbo arm) | |
|---|---|---|---|---|
| P | ar' | Prior<br>Value<br>s | Data (Sample<br>Summary statistics) | Posterior Parameters |
| 1 | | ГаП | - (O 1 T 7 ) C | |

Table 14

| Par' | Prior<br>Value | Data (Sample<br>Summary statistics) | Posterior Parameters |
|---|---|---|---|
| | S | | |
| $\mu_{0,Pbo}$ | $\lceil 0 \rceil$ | $\bar{\mathbf{x}}$ (2x1 Vector of | $-\left(k_0 * \mu_{0,Pbo}\right) + \left(n_{pbo} * \overline{\mathbf{x}}\right)$ |
| | $\begin{bmatrix} 0 \\ 0 \end{bmatrix}$ | Pbo Sample means) | $\mu_{1,Pbo} = \frac{\left(k_0 * \mu_{0,Pbo}\right) + \left(n_{pbo} * \overline{\mathbf{x}}\right)}{\left(k_0 + n_{pbo}\right)}$ |
| $k_{0,Pbo}$ | 0 | $n_{pbo}$ at IA2 | $k_{1,Pbo} = \left(k_0 + n_{pbo}\right)$ |
| $ u_{0,Pbo}$ | 0 | $n_{pbo}$ at IA2 | $v_{1,Pbo} = \left(v_0 + n_{pbo}\right)$ |
| $\Psi_{0,Pbo}$ | $\begin{bmatrix} 0 & 0 \end{bmatrix}$ | $\mathbf{C} = (n_{pbo} - 1) * VCV$ $\mathbf{C} \text{ is a } 2x2 \text{ matrix}$ | $\Psi_{1,Pbo}$ = |
| | $\begin{bmatrix} 0 & 0 \end{bmatrix}$ | C is a 2x2 matrix | $\left(\left(k_{0}*n_{-k_{0}}\right)\right)$ |
| | | VCV is sample variance | $\Psi_{0,Pbo} + \mathbf{C} + \left( \left( \frac{k_0 * n_{pbo}}{k_0 + n_{pbo}} \right) * \left( \overline{\mathbf{x}} - \mu_{0,Pbo} \right) * \left( \overline{\mathbf{x}} - \mu_{0,Pbo} \right) \right)$ |
| | | covariance matrix | ( ··· o · · · · pbo ) |

The Posterior parameters (subscripted with a 1) from Table 14 are used to sample the parameters of the Multivariate normal distribution for a future subject and generate sufficient data to "complete the study recruitment for the arm". Each of the following steps constitutes one "inner loop":

- O Draw a sample VCV matrix  $\Sigma_{Pbo}$  (Note:  $\Sigma_{Pbo}$  relates to an individual subject, not a mean) from the inverse Wishart distribution parameterized using the posteriors  $\Psi_{1,Pbo}$  and  $\nu_{1,Pbo}$
- $\circ$  Conditional on the sampled  $\Sigma_{Pbo}$  draw a single sample (denoted  $\mu_{Fut,Pbo}$ ) from a MVN distribution with a mean vector parameterised using the posterior for  $\mu_{\mathrm{l},Pbo}$  and a VCV matrix parameterised using  $\frac{\mathrm{Sampled}\,\Sigma_{Pbo}}{k_{\mathrm{l},Pbo}}$
- o Draw sufficient subjects to reach a total of 40 per arm from the (same within an inner loop) MVN distribution i.e. from  $\sim^{MVN} (\mu_{\text{Fut,Pbo}}, \Sigma_{Pbo})$ . For example if the timing of the interim analysis was after 15 subjects then sample 25 future subjects from the MVN.
- Repeat this inner looping a total of 1,000 times

Conceptually 1,000 hybrid datasets are formed by repeatedly joining the observed data at time of the interim onto the 1,000 simulated sets of future subjects from the inner loops. Each of these "end of study datasets" (Eos) could then be analysed separately to obtain the joint probability of seeing any decrease in mean PaO2/FiO2 in conjunction with any increase in mean PVPI (relative to placebo).

However for computational speed the mechanism of updating the MVN hyperparameters was also used to obtain the end of study posterior distributions for the mean of each treatment arm. This is achieved by deriving the same set of sample summary statistics from each set of future simulated subjects (the "future data") and using the previous posteriors as priors. This results in Table 15. A further assumption uses the expected value of the inverse-Wishart distribution as the "sampled"  $\Sigma_{Eos}$  when obtaining the MVN distribution for the Mean treatment effect parameters for each arm. To further speed computations matrix algebra is used to obtain a MVN distribution for the end of study mean treatment difference parameters.

Using this distribution of mean treatment differences at the end of the study the probability of seeing any decrease in PaO2/FiO2 in conjunction with any increase in PVPI can be determined (since this problem is bivariate the SAS function PROBBNRM may be used).

Table 15 Mechanism for updating hyperparameters for end of study treatment effects (Pbo arm)

| Par' | Prior<br>Values | Data (Sample<br>Summary statistics<br>for future subjects) | Posterior |
|---|---|---|---|
| $\mu_{2,Pbo}$ | $\mu_{1,Pbo}$ (Table 14) | $\overline{\mathbf{X}}_{\mathrm{Fut,Pbo}}$ | $\mu_{2,Pbo} = \frac{\left(k_1 * \mu_{1,Pbo}\right) + \left(n_{rem} * \overline{\mathbf{x}}_{Fut,Pbo}\right)}{\left(k_{1,Pbo} + n_{rem}\right)}$ |
| $k_{2,Pbo}$ | k <sub>1,Pbo</sub> (Table 14) | $n_{rem} = 80 - n_{pbo}$ | $k_{2,Pbo} = \left(k_{1,Pbo} + n_{rem}\right)$ |
| $V_{2,Pbo}$ | $ u_{1,Pbo} $ (Table 14) | $n_{rem} = 80 - n_{pbo}$ | $v_{2,Pbo} = \left(v_{1,Pbo} + n_{rem}\right)$ |
| $\Psi_{2,Pbo}$ | $\Psi_{1,Pbo}$ (Table 14) | $\mathbf{C}_{Fut,Pbo} = (n_{rem} - 1)^*$ $VCV_{Fut,Pbo}$ | $\Psi_{2,Pbo} = \Psi_{1,Pbo} + \mathbf{C}_{Fut,Pbo} + \left( \left( \frac{k_1 * n_{rem}}{k_1 + n_{rem}} \right) * \left( \overline{\mathbf{x}}_{Fut,Pbo} - \mu_{1,Pbo} \right) * \left( \overline{\mathbf{x}}_{Fut,Pbo} - \mu_{1,Pbo} \right)^T \right)$ |

End of study Mean Pbo effect = 
$$\mu_{Eos, Pbo} \sim \left( \mu_{2, Pbo}, \frac{E[\Sigma_{Eos, Pbo}]}{k_{2, Pbo}} \right)$$

Hence

EoS Mean Trt Diffs = 
$$\mu_{Eos,Diff} \sim \left( (\mu_{2,Act} - \mu_{2,Pbo}), \frac{\left( \frac{\Psi_{2,Pbo}}{v_{2,Pbo} - 2 + 1} \right) + \left( \frac{\Psi_{2,Act}}{v_{2,Act} - 2 + 1} \right)}{\left( k_{2,Pbo} + k_{2,Act} \right)} \right)$$

Each of the parameters of the EoS Mean Trt Diffs MVN distribution for that inner loop is saved.

The output of the outer and inner loops for a given scenario is a dataset with approximately 10,000 \* 34 \* 1,000 sets of parameters that describe the end of study MVN distribution of mean treatment differences. In addition, each record also contains sufficient metadata to link it back to its generating circumstances.

Iterative discussions within the study team led to the critical boundaries for the endpoints that would be considered futile (i.e. any decrease in PaO2/FiO2 in conjunction with any increase in PVPI). Once set, the optimisation questions became "timing of IA2 and how much confidence was required to declare futility".

These outer/inner loop datasets allow multiple probability trigger thresholds to be evaluated without need to re-simulate (see topics below).

#### Generation of the individual subject data for the outer loop

Subject level PVPI and PaO2/FiO2 data from BALTI prevention trial (Perkins, 2014) were available for 56 subjects at pre-surgery and immediately post-surgery time points.

PC SAS (v9.3 TS1M2) PROC MCMC was used to fit the model in Equation 1 to the BALTI trial data and, once convergence achieved, simultaneously generate 10,000 sets of 80 subjects (40 per placebo arm using the fitted BALTI means and 40 per active arm using the BALTI means offset by a pre-specified amount; see Table 20). Each endpoint for each of the 80 subjects is represented as a distinct model parameter.

#### Equation 1 MVN Model fitted to BALTI dataset for the ith Subject

$$\begin{bmatrix} \hat{y}_1 & \hat{y}_2 \\ \hat{y}_1 & \hat{y}_2 \end{bmatrix}_i = \begin{bmatrix} BSP/F_i & \ln(BSPVPI_i) \end{bmatrix} \begin{bmatrix} \hat{B}S_{P/F} & 0 \\ 0 & \hat{B}S_{PVPI} \end{bmatrix} + \begin{bmatrix} \hat{\mu}_{BALTI,P/F} & \hat{\mu}_{BALTI,PVPI} \end{bmatrix}$$

i = 1 to 56

Where

 $BSP/F_i = Baseline (pre - surgery) PaO2/FiO2 for ith Subject (Centered)$ 

 $BSPVPI_i$  = Baseline (pre - surgery) PVPI for ith Subject (Centered)

To link to observed data assume : 
$$\begin{bmatrix} y_{1} & y_{2} \\ y_{1} & y_{2} \end{bmatrix}_{i}^{MVN} \begin{bmatrix} y_{1} & y_{2} \\ \hat{y}_{1} & \hat{y}_{2} \end{bmatrix}_{i}$$
,  $[\Sigma]$  where  $\Sigma$  is a 2x2

Variance Covariance matrix common to both treatments

Prior distributions are:

$$\begin{bmatrix} \hat{B}S_{P/F} & \hat{B}S_{PVPI} \end{bmatrix}^{MVN} \sim \begin{bmatrix} \begin{bmatrix} 0 & 0 \end{bmatrix}_{i}, \begin{bmatrix} 1E6 & 0 \\ 0 & 1E6 \end{bmatrix} \end{cases}; \text{ initial values} \begin{bmatrix} 0.36 & 0.4 \end{bmatrix} \\
\begin{bmatrix} \hat{\mu}_{BALTI,P/F} & \hat{\mu}_{BALTI,PVPI} \end{bmatrix}^{MVN} \sim \begin{bmatrix} \begin{bmatrix} 0 & 0 \end{bmatrix}_{i}, \begin{bmatrix} 1E6 & 0 \\ 0 & 1E6 \end{bmatrix} \end{bmatrix}; \text{ initial values} \begin{bmatrix} 20 & 0.5 \end{bmatrix} \\
\Sigma \sim \begin{bmatrix} 2, \begin{bmatrix} 1 & 0 \\ 0 & 1 \end{bmatrix} \end{pmatrix}$$

Example of supplied mean vectors for Placebo and Active arms for the "minimum desired profile"

$$\begin{bmatrix} P/F \\ LN \Big( PVPI \Big) \end{bmatrix} : \mu_P = \begin{bmatrix} 42.27 \\ 0.765 \end{bmatrix} \mu_a = \begin{bmatrix} 48.6105 \\ 0.602481 \end{bmatrix} \mu_{dif \& rat} = \begin{bmatrix} 6.3405 \\ -0.16252 \end{bmatrix} \& \begin{bmatrix} 1.15 \\ 0.85 \end{bmatrix} = \frac{15\%}{15\%} \updownarrow$$

Distribution used to simulate a future subject for the Placebo and Active arms

$$\begin{bmatrix} y_{Pbo,P/F} & y_{Pbo,PVPI} \end{bmatrix}_{k}^{MVN} \sim ([42.27 \quad 0.765]_{i}, \Sigma)$$

$$\begin{bmatrix} y_{Act,P/F} & y_{Act,PVPI} \end{bmatrix}_{k}^{MVN} \sim ([48.6105 \quad 0.602481]_{i}, \Sigma)$$

k = 1 to 40 and the sampled  $\Sigma$  is the same for each of the 2k subjects within a given MCMC iteration but a new  $\Sigma$  will be drawn for each of the 10,000 MCMC iterations (outer loops)

#### Generation of the summary statistics for the outer loops

SAS PROC IML was used to read in the PROC MCMC output (a dataset with one row per outer loop containing all subjects data for both treatment arms), and to process each row in turn as follows:

Manipulate/split the row contents into a matrix of dimension 2x40 (separate matrices of endpoints per treatment arm).

Subset each 2x40 matrix into possible interim analysis 2 timings by taking the first 5 observations and then 6<sup>th</sup>, 7<sup>th</sup>, etc until reaching the 39<sup>th</sup> and repeat the following

Centre each endpoint and derive the sample mean and sample variance covariance matrix (n-1 as the divisor) and also express the sample variance covariance matrix in terms of correlations and save the n per arm at the time of interim

Save each element of these matrices (to give one row per outer loop per possible interim analysis timing containing Pbo and Active summary statistics)

#### Choice of IA2 timing

Potential IA2 timings examined in this simulation exercise were at 15, 20 and 25 subjects per arm (plus a sanity check of 39 per arm).

#### Choice of IA2 futility threshold probability (applies within each inner loop)

A series of potential futility threshold probabilities for each inner loop were evaluated (ranging from 0.05 to 0.95 by increments of 0.05 using SAS formats). If the posterior probability of observing any decrease in PaO2/FiO2 in conjunction with any increase in PVPI exceeded the proposed threshold that inner loop was marked as futile.

## Choice of IA2 proportion of futile inner loop studies that will trigger the Pause and Review IA2 outcome (applies within each outer loop)

A series of threshold proportions were evaluated (ranging from 0.05 to 0.95 by increments of 0.05 using SAS formats). If the proportion of the (1,000) inner loops marked as futile exceeded the proposed threshold proportion that outer loop was said to have declared a "Pause and Review" outcome.

#### Selecting the timing and futility threshold

Each inner loop \* outer loop \* potential IA2 timing \* dataset scenario (Table 20) provides a posterior probability of observing any decrease in PaO2/FiO2 in conjunction with any increase in PVPI (giving 1,000\*10,000\*4\*5 = 20,000,000 values).

A series of SAS formats were created to dichotomise each of these 20,000,000 posterior probabilities into binary outcomes (1=Yes/event occurs, 0=No/event did not occur). For example to evaluate 0.1 and 0.65 futility thresholds the following SAS formats would be created:

$$Low - 0.1 = 0$$
 and  $Low - 0.65 = 0$   
 $0.1 - High = 1$   $0.65 - High = 1$ 

In turn, the dataset of posterior probabilities had each SAS formatted applied and was put through PROC FREQ to determine the proportion of inner loops where the posterior probability for futility exceeded the threshold implied by the SAS format (producing a record for each combination of SAS format \* outer loop \* potential IA2 timing \* dataset scenario).

Another set of SAS formats were created and applied in turn to the above dataset. These flagged when the proportion of the inner loops exceeded the proposed value implied by the associated SAS format, i.e. a Pause and Review outcome. Expressing this information as a proportion of Pause and Review outcomes gives a final dataset with one record per potential IA2 timing \* dataset scenario combination.

Table 16 details the combinations of dataset scenario, IA2 timing, futility proportions and proportion required to declare Pause and Review that were evaluated. A subset of the simulation results pertinent to the choices made for the protocol are summarised in Table 17. Other results are available on file. The highlighted column in Table 17 reflects the operating characteristics of the IA2 rules/criteria selected by the study team.

Table 16 Factors varied in evaluating IA2 operating characteristics

| Every com | Every combination of the following factors were evaluated | | |
|---|---|---|---|
| Hypothetical<br>Treatment<br>Profile | Interim Timings<br>(number of<br>observed<br>subjects per<br>arm) | Inner loop<br>futility threshold | Proportion of inner loops needed to declare "Pause and Review" |
| Null | | | |
| Active as BALTI<br>Pre-op<br>Half Active as | | 0.95, 0.9, 0.85,<br>0.8, 0.75, 0.7,<br>0.65, 0.6, 0.55, | 0.95, 0.9, 0.85,<br>0.8, 0.75, 0.7,<br>0.65, 0.6, 0.55, |
| BALTI Pre-op | 39, 25, 20, 15 | 0.5, 0.45, 0.4, | 0.5, 0.45, 0.4, |
| Quarter Active as<br>BALTI Pre-op | | 0.35, 0.3, 0.25,<br>0.2, 0.15, 0.1,<br>0.05 | 0.35, 0.3, 0.25,<br>0.2, 0.15, 0.1,<br>0.05 |
| Minimum desired profile | | | |

Table 17 Selected results from simulation exercise to evaluate IA2 operating characteristics

| Hypothetical<br>Treatment | % of simulated outer loops with Pause and Review outcome [Inner loop Futility threshold: 0.1 Proportion of inner loops to declare "Pause and Review": 0.3] | | | |
|---|---|---|---|---|
| Profile | IA2 @ 39 p.a. | IA2 @ 25 p.a. | IA2 @ 20 p.a. | IA2 @ 15 p.a. |
| Null | 71.69% | 76.15% | 76.26% | 75.98% |
| Active as BALTI Pre-op | 0.02% | 0.31% | 1.06% | 2.62% |
| Half Active as BALTI Pre-op | 6.17% | 15.69% | 20.59% | 25.82% |
| Quarter Active as BALTI Pre-<br>op | 31.65% | 44.41% | 48.13% | 51.46% |
| Minimum desired profile | 2.24% | 7.96% | 11.41% | 16.46% |

Note: Highlighted column (20 per arm) reflects the IA2 choices selected for the study protocol

**Note:** Whilst writing this RAP a minor error in the SAS code was discovered and corrected (results presented in this RAP reflect the corrected data). The SAS code was not adding dummy records to the first PROC FREQ output dataset to re-include the opposite outcome whenever all inner loops had identical results (i.e. either all 1,000 inner loops were futile, or all 1,000 inner loops were not futile). Therefore the denominators used in subsequent PROC FREQ's (number of input records) were not always as large as they should have been; but this situation was infrequent, so the impact is deemed minimal.

## 11.12.2. Simulations providing operating characteristics of the target sample size (40 per arm)

The simulated data relating to all 80 subjects within each of the 10,000 outer loops for each dataset scenario were used to obtain sets of sample summary statistics and then to obtain the parameters of the MVN distribution for the End of Study mean treatment differences (see Section 11.12.1 and Table 20). For clarification, since there are no inner loops non-informative priors were used (Table 14) along with the expected value of the inverse-Wishart distribution when deriving the parameters of the MVN distribution for the mean treatment difference.

Discussions within the study team led to the clinically relevant differences that make up Figure 2. The SAS PROBBNRM function was used to obtain the posterior probability of the mean treatment effects being in each region defined by Figure 2, for each outer loop, using the corresponding MVN distribution for the mean treatment difference. This probability only depends upon the location of the clinically relevant differences.

To get the process started an arbitrary probability threshold was assigned as a "trigger" for each region and if the posterior probability of being in the region exceeded the trigger it was deemed to have occurred. Since more than one region may be triggered the algorithm to combined triggered regions to obtain a single outcome was codified as

| Overall success | ≥1 of the "Success" outcomes | AND | 0 "Failures" |
|---|---|---|---|
| <b>Potentially Unsuccessful</b> | 0 "Success" outcomes | AND | 1 "Failure" |
| Inconclusive | 0 "Success" outcomes | AND | 0 "Failures" |
| Inconsistent | ≥1 of the "Success" outcomes | AND | 1 "Failure" |

Based on the arbitrary trigger thresholds each of the 10,000 outer loops was evaluated to determine which regions (if any) met their probability triggers, and subsequently, which outcome occurred for that outer loop (Note: The language used in Section 9.2.1 of the protocol refers to these probability triggers as "confidence levels"). The operating characteristic of each outcome is the number of observed occurrences expressed as a proportion of the 10,000 outer loops. These were presented to the study team and an iterative process was started to vary these thresholds and observe the impact on operating characteristics.

The "null" and "minimum desired profile" have different desired operating characteristics and the trigger thresholds were varied until the team were comfortable with the operating characteristics of both. This led to the criteria in Figure 2 (probability triggers of 0.75 for Step 1, 0.25 for Step 2 and 0.35 for Step 3; denoted {0.75, 0.25, 0.35}) and the resulting operating characteristics in Table 18 that were presented in Table 5 of the study protocol (re-produced here using all scenarios from Table 20).

Table 18 Results from Simulation exercise assuming 40 p.a. complete

| Hypothetical | % of simulated studies with outcome | | | |
|---|---|---|---|---|
| Treatment Profile | Overall Success | Potentially<br>Unsuccessful | Inconclusive | Inconsistent |
| Null | 4.65% | 92.81% | 2.54% | 0% |
| Active as BALTI Pre-op | 92.72% | 6.83% | 0.45% | 0% |
| Half Active as<br>BALTI Pre-op | 40.93% | 49.98% | 9.09% | 0% |
| Quarter Active as BALTI Pre-<br>op | 15.61% | 77.13% | 7.26% | 0% |
| Minimum desired profile | 80.64% | 13.63% | 5.73% | 0% |

A well performing end of study decision pathway should not be expected to conclude success for the "Null" profile whilst reliably concluding success for the "minimum desired profile". In the language of frequentist hypothesis testing the "Overall success"

probabilities for the Null and Minimum desired profile are akin to the Type I error rate and power for the study design respectively. These were estimated to be 4.65% and 80.64% respectively so the study design and end of study pathway was deemed acceptable (assuming 40 evaluable subjects per arm and residual variance covariance estimates in line with the BALTI trial (Perkins, 2014)).

An additional step evaluated the operating characteristics of the final end of study decision pathway (Figure 2) using 25, 30 and 35 subjects per arm. Unsurprisingly, the operating characteristics were not as good, given the reduced information content (see Table 19).

This exercise was also repeated using the following sets of probability triggers for the three steps of Figure 2: {0.75, 0.25, 0.50}, {0.70, 0.25, 0.50}, {0.95, 0.25, 0.50}, {0.95, 0.25, 0.25} and {0.75, 0.25, 0.25}; results presented in Table 21, Table 22, Table 23, Table 24 and Table 25 respectively.

Note: Candidate combinations of probability thresholds were selected based upon review of the distributions formed from the 10,000 outer loop probabilities associated with the 3x outcomes described in Figure 2 for each dataset in Table 20 and for 25, 30, 35 and 40 per arm total sample size. These are shown in Figure 5, Figure 6, Figure 7, Figure 8 and Figure 9. In these figures the boxid's titled "Fail", "Strong Success" and "Success" correspond to the Step 1, Step 2 and Step 3 probability thresholds respectively. A threshold would be a vertical slice placed on the x-axis and the proportion exceeding the slice would be the expected proportion triggering that rule (but the overall outcome requires the codifying rules described above).

Table 19 Results from Sensitivity analysis assuming 25, 30 and 35 p.a. complete

| Hypothetical | | | % of simulated stu | idies with outco | me |
|---|---|---|---|---|---|
| Treatment Profile | n (p.a.) | Overall Success | Potentially<br>Unsuccessful | Inconclusive | Inconsistent |
| | 25 | 9.38% | 86.03% | 4.59% | 0% |
| Null | 30 | 7.32% | 88.52% | 4.16% | 0% |
| | 35 | 5.65% | 90.91% | 3.44% | 0% |
| Active as BALTI Pre- | 25 | 88.49% | 9.98% | 1.53% | 0% |
| ор | 30 | 90.04% | 8.97% | 0.99% | 0% |
| | 35 | 91.51% | 7.86% | 0.63% | 0% |
| Half Active as BALTI | 25 | 44.57% | 46.42% | 9.01% | 0% |
| Pre-op | 30 | 42.84% | 47.68% | 9.48% | 0% |
| | 35 | 42.08% | 48.64% | 9.28% | 0% |
| Quarter<br>Active as | 25 | 21.96% | 68.95% | 9.09% | 0% |
| BALTI Pre- | 30 | 19.50% | 72.31% | 8.19% | 0% |
| ор | 35 | 17.49% | 74.95% | 7.56% | 0% |
| Minimum | 25 | 76.41% | 17.06% | 6.53% | 0% |
| desired | 30 | 77.71% | 15.91% | 6.38% | 0% |
| profile | 35 | 79.25% | 14.9% | 5.85% | 0% |

Table 20 Hypothetical scenarios for generating datasets

| DID | DID Desc' | Pbo Vector for Immediate | Active Vector for Post-op mean response | MAX n | nmc |
|---|---|---|---|---|---|
| | | Post-op mean response | | p.a. | |
| 1 | Null | $\begin{bmatrix} P/F \\ LN(PVPI) \end{bmatrix} : \mu_p = \begin{bmatrix} 42.27 \\ 0.765 \end{bmatrix}$ | $\mu_{a} = \begin{bmatrix} 42.27 \\ 0.765 \end{bmatrix} \mu_{dif \& rat} = \begin{bmatrix} 0 \\ 0 \end{bmatrix} \& \begin{bmatrix} 1 \\ 1 \end{bmatrix} = NOCHANGE$ | 40 | 10000 |
| 2 | Active as BALTI<br>Pre-op | $\begin{bmatrix} P/F \\ LN(PVPI) \end{bmatrix} : \mu_p = \begin{bmatrix} 42.27 \\ 0.765 \end{bmatrix}$ | $\mu_{a} = \begin{bmatrix} 53.14 \\ 0.577 \end{bmatrix} \mu_{dif \& rat} = \begin{bmatrix} 10.87 \\ -0.188 \end{bmatrix} \& \begin{bmatrix} 1.257 \\ 0.829 \end{bmatrix} = \frac{25.7\% \uparrow}{17.1\% \downarrow}$ | 40 | 10000 |
| 3 | Half Active as<br>BALTI Pre-op | $\begin{bmatrix} P/F \\ LN(PVPI) \end{bmatrix} : \mu_p = \begin{bmatrix} 42.27 \\ 0.765 \end{bmatrix}$ | $\mu_{a} = \begin{bmatrix} 47.705 \\ 0.671 \end{bmatrix} \mu_{dif \& rat} = \begin{bmatrix} 5.435 \\ -0.094 \end{bmatrix} \& \begin{bmatrix} 1.129 \\ 0.910 \end{bmatrix} = \frac{12.9\% \uparrow}{9.0\% \downarrow}$ | 40 | 10000 |
| 4 | Quarter Active as<br>BALTI Pre-op | $\begin{bmatrix} P/F \\ LN(PVPI) \end{bmatrix} : \mu_p = \begin{bmatrix} 42.27 \\ 0.765 \end{bmatrix}$ | $\mu_{a} = \begin{bmatrix} 44.985 \\ 0.718 \end{bmatrix} \mu_{dif \& rat} = \begin{bmatrix} 2.715 \\ -0.047 \end{bmatrix} \& \begin{bmatrix} 1.064 \\ 0.954 \end{bmatrix} = \frac{6.4\% \uparrow}{4.6\% \downarrow}$ | 40 | 10000 |
| 5 | Minimum desired profile | $\begin{bmatrix} P/F \\ LN(PVPI) \end{bmatrix} : \mu_p = \begin{bmatrix} 42.27 \\ 0.765 \end{bmatrix}$ | $\mu_{a} = \begin{bmatrix} 48.6105 \\ 0.602481 \end{bmatrix} \mu_{dif \& rat} = \begin{bmatrix} 6.3405 \\ -0.16252 \end{bmatrix} \& \begin{bmatrix} 1.15 \\ 0.85 \end{bmatrix} = \frac{15\% \uparrow}{15\% \downarrow}$ | 40 | 10000 |

DID = Dataset ID, p.a. = per arm, nmc = Number of MCMC iterations (Outer loops)

Table 21 Results from probability threshold set {0.75, 0.25, 0.50} and Sensitivity analysis assuming 25, 30, 35 and 40 p.a. complete

| Hypothetical | | % of simulated studies with outcome | | | |
|---|---|---|---|---|---|
| Treatment Profile | n (p.a.) | Overall Success | Potentially<br>Unsuccessful | Inconclusive | Inconsistent |
| | 25 | 6.06% | 86.03% | 7.91% | 0% |
| Madi | 30 | 4.46% | 88.52% | 7.02% | 0% |
| Null | 35 | 3.52% | 90.91% | 5.57% | 0% |
| | 40 | 2.65% | 92.81% | 4.54% | 0% |
| Active as BALTI Pre- | 25 | 88.15% | 9.98% | 1.87% | 0% |
| ор | 30 | 89.75% | 8.97% | 1.28% | 0% |
| | 35 | 91.31% | 7.86% | 0.83% | 0% |
| | 40 | 92.57% | 6.83% | 0.60% | 0% |
| Half Active as BALTI | 25 | 40.40% | 46.42% | 13.18% | 0% |
| Pre-op | 30 | 39.04% | 47.68% | 13.28% | 0% |
| | 35 | 37.90% | 48.64% | 13.46% | 0% |
| | 40 | 37.12% | 49.98% | 12.90% | 0% |
| Quarter<br>Active as | 25 | 17.42% | 68.95% | 13.63% | 0% |
| BALTI Pre- | 30 | 15.24% | 72.31% | 12.45% | 0% |
| ор | 35 | 13.32% | 74.95% | 11.73% | 0% |
| | 40 | 11.38% | 77.13% | 11.49% | 0% |
| | 25 | 73.06% | 17.06% | 9.88% | 0% |
| Minimum | 30 | 74.61% | 15.91% | 9.48% | 0% |
| desired profile | 35 | 76.04% | 14.90% | 9.06% | 0% |
| | 40 | 77.53% | 13.63% | 8.84% | 0% |

Table 22 Results from probability threshold set {0.70, 0.25, 0.50} and Sensitivity analysis assuming 25, 30, 35 and 40 p.a. complete

| Hypothetical | | | % of simulated stu | idies with outco | me |
|---|---|---|---|---|---|
| Treatment Profile | n (p.a.) | Overall Success | Potentially<br>Unsuccessful | Inconclusive | Inconsistent |
| | 25 | 6.06% | 87.89% | 6.05% | 0% |
| Nivill | 30 | 4.45% | 90.31% | 5.23% | 0.01% |
| Null | 35 | 3.50% | 92.73% | 3.75% | 0.02% |
| | 40 | 2.65% | 93.96% | 3.39% | 0% |
| Active as<br>BALTI Pre- | 25 | 86.71% | 10.60% | 1.25% | 1.44% |
| ор | 30 | 88.46% | 9.43% | 0.82% | 1.29% |
| | 35 | 89.92% | 8.12% | 0.57% | 1.39% |
| | 40 | 91.40% | 7.01% | 0.42% | 1.17% |
| Half Active as BALTI | 25 | 39.47% | 49.87% | 9.73% | 0.93% |
| Pre-op | 30 | 38.13% | 51.15% | 9.81% | 0.91% |
| | 35 | 37.13% | 51.98% | 10.12% | 0.77% |
| | 40 | 36.16% | 53.19% | 9.69% | 0.96% |
| Quarter<br>Active as | 25 | 17.16% | 72.28% | 10.30% | 0.26% |
| BALTI Pre- | 30 | 15.08% | 75.27% | 9.49% | 0.16% |
| ор | 35 | 13.12% | 78.02% | 8.66% | 0.20% |
| | 40 | 11.24% | 79.99% | 8.63% | 0.14% |
| | 25 | 72.40% | 19.14% | 7.80% | 0.66% |
| Minimum | 30 | 73.85% | 17.97% | 7.42% | 0.76% |
| desired profile | 35 | 75.39% | 16.76% | 7.20% | 0.65% |
| | 40 | 76.92% | 15.23% | 7.24% | 0.61% |

Table 23 Results from probability threshold set {0.95, 0.25, 0.50} and Sensitivity analysis assuming 25, 30, 35 and 40 p.a. complete

| Hypothetical | | % of simulated studies with outcome | | | |
|---|---|---|---|---|---|
| Treatment Profile | n (p.a.) | Overall<br>Success | Potentially<br>Unsuccessful | Inconclusive | Inconsistent |
| | 25 | 6.06% | 65.60% | 28.34% | 0% |
| Null | 30 | 4.46% | 71.10% | 24.44% | 0% |
| Null | 35 | 3.52% | 75.65% | 20.83% | 0% |
| | 40 | 2.65% | 79.01% | 18.34% | 0% |
| Active as BALTI Pre- | 25 | 88.15% | 2.44% | 9.41% | 0% |
| op | 30 | 89.75% | 2.30% | 7.95% | 0% |
| | 35 | 91.31% | 1.67% | 7.02% | 0% |
| | 40 | 92.57% | 1.55% | 5.88% | 0% |
| Half Active as BALTI | 25 | 40.40% | 22.09% | 37.51% | 0% |
| Pre-op | 30 | 39.04% | 23.24% | 37.72% | 0% |
| | 35 | 37.90% | 23.89% | 38.21% | 0% |
| | 40 | 37.12% | 24.84% | 38.04% | 0% |
| Quarter<br>Active as | 25 | 17.42% | 42.69% | 39.89% | 0% |
| BALTI Pre- | 30 | 15.24% | 46.59% | 38.17% | 0% |
| ор | 35 | 13.32% | 49.17% | 37.51% | 0% |
| | 40 | 11.38% | 52.51% | 36.11% | 0% |
| | 25 | 73.06% | 5.06% | 21.88% | 0% |
| Minimum | 30 | 74.61% | 4.64% | 20.75% | 0% |
| desired profile | 35 | 76.04% | 4.24% | 19.72% | 0% |
| | 40 | 77.53% | 3.94% | 18.53% | 0% |

Table 24 Results from probability threshold set {0.95, 0.25, 0.35} and Sensitivity analysis assuming 25, 30, 35 and 40 p.a. complete

| Hypothetical | | % of simulated studies with outcome | | | me |
|---|---|---|---|---|---|
| Treatment Profile | n (p.a.) | Overall Success | Potentially<br>Unsuccessful | Inconclusive | Inconsistent |
| | 25 | 9.38% | 65.60% | 25.02% | 0% |
| AlII | 30 | 7.32% | 71.10% | 21.58% | 0% |
| Null | 35 | 5.65% | 75.65% | 18.70% | 0% |
| | 40 | 4.65% | 79.01% | 16.34% | 0% |
| Active as BALTI Pre- | 25 | 88.49% | 2.44% | 9.07% | 0% |
| op | 30 | 90.04% | 2.30% | 7.66% | 0% |
| | 35 | 91.51% | 1.67% | 6.82% | 0% |
| | 40 | 92.72% | 1.55% | 5.73% | 0% |
| Half Active as BALTI | 25 | 44.57% | 22.09% | 33.34% | 0% |
| Pre-op | 30 | 42.84% | 23.24% | 33.92% | 0% |
| | 35 | 42.08% | 23.89% | 34.03% | 0% |
| | 40 | 40.93% | 24.84% | 34.23% | 0% |
| Quarter<br>Active as | 25 | 21.96% | 42.69% | 35.35% | 0% |
| BALTI Pre- | 30 | 19.50% | 46.59% | 33.91% | 0% |
| ор | 35 | 17.49% | 49.17% | 33.34% | 0% |
| | 40 | 15.61% | 52.51% | 31.88% | 0% |
| | 25 | 76.41% | 5.06% | 18.53% | 0% |
| Minimum | 30 | 77.71% | 4.64% | 17.65% | 0% |
| desired profile | 35 | 79.25% | 4.24% | 16.51% | 0% |
| | 40 | 80.64% | 3.94% | 15.42% | 0% |

Table 25 Results from probability threshold set {0.75, 0.25, 0.25} and Sensitivity analysis assuming 25, 30, 35 and 40 p.a. complete

| Hypothetical | | % of simulated studies with outcome | | | |
|---|---|---|---|---|---|
| Treatment Profile | n (p.a.) | Overall<br>Success | Potentially<br>Unsuccessful | Inconclusive | Inconsistent |
| | 25 | 12.70% | 86.03% | 1.27% | 0% |
| AlII | 30 | 10.36% | 88.52% | 1.12% | 0% |
| Null | 35 | 8.21% | 90.91% | 0.88% | 0% |
| | 40 | 6.62% | 92.81% | 0.57% | 0% |
| Active as BALTI Pre- | 25 | 88.89% | 9.98% | 1.13% | 0% |
| op | 30 | 90.26% | 8.97% | 0.77% | 0% |
| | 35 | 91.61% | 7.86% | 0.53% | 0% |
| | 40 | 92.80% | 6.83% | 0.37% | 0% |
| Half Active as BALTI | 25 | 48.33% | 46.42% | 5.25% | 0% |
| Pre-op | 30 | 46.59% | 47.68% | 5.73% | 0% |
| | 35 | 45.81% | 48.64% | 5.55% | 0% |
| | 40 | 44.63% | 49.98% | 5.39% | 0% |
| Quarter<br>Active as | 25 | 26.85% | 68.95% | 4.20% | 0% |
| BALTI Pre- | 30 | 23.87% | 72.31% | 3.82% | 0% |
| ор | 35 | 21.64% | 74.95% | 3.41% | 0% |
| | 40 | 19.92% | 77.13% | 2.95% | 0% |
| | 25 | 79.08% | 17.06% | 3.86% | 0% |
| Minimum | 30 | 80.15% | 15.91% | 3.94% | 0% |
| desired profile | 35 | 81.54% | 14.90% | 3.56% | 0% |
| | 40 | 83.04% | 13.63% | 3.33% | 0% |

Figure 5 Hypothetical Treatment Profile used to generate data (subjects)=Null



Figure 6 Hypothetical Treatment Profile used to generate data (subjects)=
Active as BALTI Pre-op



Figure 7 Hypothetical Treatment Profile used to generate data (subjects)= Half Active as BALTI Pre-op







Figure 9 Hypothetical Treatment Profile used to generate data (subjects)=
Minimum desired profile



## 11.13. Appendix 13: Abbreviations & Trade Marks

### 11.13.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> /CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| ELF | Epithelial Lining Fluid |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| GSK | GlaxoSmithKline |
| GUI | Guidance |
| LOC | Last Observation Carries Forward |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| SOFA | Sequential Organ Failure Assessment |
| SOFA | 1 0 |
| SUF | Standard Operation Procedure |

| Abbreviation | Description |
|---|---|
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| <b>Note:</b> See Table 13 for abbreviations used in Transpulmonary Thermodilution | |

### 11.13.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| Picco |
| SAS |
| Spotfire |
| WinNonlin |

### 11.14. Appendix 14: List of Data Displays

### 11.14.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Pharmacodynamic and / or Biomarker | 5.1 to 5.n | 5.1 to 5.n |
| Pharmacogenetics | 6.1 to 7.n | 6.1 to 7.n |
| Section | List | ings |
| ICH Listings | <br>1 t | 0 X |
| Other Listings | (x+1 | ) to z |

### 11.14.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 15: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacogenetics | PGX_Fn | PGX_Tn | PGX_Ln |

#### NOTES:

 Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

## 11.14.3. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|---|---|
| DS [X] | During Study |
| DE [X] | Dose Escalation |
| IAn [X] | Interim Analysis <n> Statistical Analysis Complete</n> |
| SAC [X] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.
### 11.14.4. Study Population Tables

| Study F | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Accountability | У | | | |
| 1.1. | n/a | POP_T1 | Summary of Subject Accountability (subjects constituting each Statistical Analysis Population) | Statistical analysis population by treatment. Create categories for the main treatment descriptors and for each of the alternative sets (grouping by study medication and BAL sampling location) | IA1 [1], IA2 [2],<br>SAC [1] |
| Subjec | t Disposition | | | | |
| 1.2. | Safety | ES1 | Summary of Subject Disposition | | SAC [1] |
| 1.3. | Screen<br>Failures | ES6 | Summary of Reasons for Screening Failure | Facilitates CONSORT diagram in publications. Therefore also sub-total the inclusion/exclusion category by the applicable individual criteria (e.g. exclusion due to presence of preexisting ADA antibodies). | SAC [1] |
| 1.4. | Safety | DV1b | Summary of Important Protocol Deviations | Create Separate "block" for each of the three per protocol populations in the style given in the shell. | SAC [1] |
| Demog | raphy | | | | |
| 1.5. | Safety | DM1 | Summary of Demographic Characteristics (by Treatment arm) | Use Main Treatment Group Descriptors | IA1 [1], IA2 [2],<br>SAC [1] |
| 1.6. | Safety | DM1 | Summary of Demographic Characteristics (by Study Medication) | Use Alternative Treatment Group<br>Descriptors #1 | IA1 [1], IA2 [2],<br>SAC [1] |
| 1.7. | Safety | DM1 | Summary of Demographic Characteristics (by BAL Location) | Use Alternative Treatment Group<br>Descriptors #2 | IA1 [1], IA2 [2],<br>SAC [1] |

| Study F | opulation Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.8. | Safety | DM5 | Summary of Race and Racial Combinations Details (by Treatment arm) | Use Main Treatment Group Descriptors | IA1 [1], IA2 [2],<br>SAC [1] |
| 1.9. | Safety | DM5 | Summary of Race and Racial Combinations Details (by Study Medication) | Use Alternative Treatment Group Descriptors #1 | IA1 [1], IA2 [2],<br>SAC [1] |
| 1.10. | Safety | DM5 | Summary of Race and Racial Combinations Details (by BAL Location) | Use Alternative Treatment Group<br>Descriptors #2 | IA1 [1], IA2 [2],<br>SAC [1] |
| 1.11. | Safety | SAFE_T1 | Number of Subjects per Country by Treatment Group | Macro: EMA_COUNTRY | SAC [1] |
| 1.12. | Safety | SAFE_T2 | Number of Subjects in each Age Group by Treatment Group | Macro: EMA_AGEGRP All age categories (in years) will be produced if they exist in the data, and according to the EMA requirements. If age unit is other than year, then programming modifications will be required. | SAC [1] |
| Medica | Condition & C | oncomitant Medic | cations | | |
| 1.13. | Safety | MH4 | Summary of Current Medical Conditions (by Treatment arm) | Use Main Treatment Group Descriptors | IA1 [1], IA2 [2],<br>SAC [1] |
| 1.14. | Safety | MH4 | Summary of Current Medical Conditions (by Study Medication) | Use Alternative Treatment Group<br>Descriptors #1 | IA1 [1], IA2 [2],<br>SAC [1] |
| 1.15. | Safety | MH4 | Summary of Current Medical Conditions (by BAL Location) | Use Alternative Treatment Group<br>Descriptors #2 | IA1 [1], IA2 [2],<br>SAC [1] |
| 1.16. | Safety | MH4 | Summary of Past Medical Conditions (by Treatment arm) | Use Main Treatment Group Descriptors | IA1 [1], IA2 [2],<br>SAC [1] |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.17. | Safety | MH4 | Summary of Past Medical Conditions (by Study Medication) | Use Alternative Treatment Group<br>Descriptors #1 | IA1 [1], IA2 [2],<br>SAC [1] |
| 1.18. | Safety | MH4 | Summary of Past Medical Conditions (by BAL Location) | Use Alternative Treatment Group<br>Descriptors #2 | IA1 [1], IA2 [2],<br>SAC [1] |
| 1.19. | Safety | CP_CM1 | Summary of Concomitant Medications by Generic Term (by Treatment arm) | Use Main Treatment Group Descriptors | IA1 [1], IA2 [2],<br>SAC [1] |
| 1.20. | Safety | CP_CM1 | Summary of Concomitant Medications by Generic Term (by Study Medication) | Use Alternative Treatment Group<br>Descriptors #1 | IA1 [1], IA2 [2],<br>SAC [1] |
| 1.21. | Safety | CP_CM1 | Summary of Concomitant Medications by Generic Term (by BAL Location) | Use Alternative Treatment Group<br>Descriptors #2 | IA1 [1], IA2 [2],<br>SAC [1] |

## 11.14.5. Efficacy Tables

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Primary | / Analysis | | | | |
| 2.1. | PP1 | EFF_T1 | Summary Statistics supporting Primary Analysis (Absolute and Change from Baseline): PVPI and PaO2/FiO2 (by Treatment arm) | Use Main Treatment Group Descriptors Only include timepoints associated with the primary analysis (i.e. the two assessments on Day 1: prior to surgery/post surgery). | IA2 [1], SAC [1] |
| 2.2. | PP2 | EFF_T1 | Summary Statistics supporting Primary Analysis (Absolute and Change from Baseline): PVPI and PaO2/FiO2 (by Study Medication) | Use Alternative Treatment Group Descriptors #1 Only include timepoints associated with the primary analysis (i.e. the two assessments on Day 1: prior to surgery/post surgery). | IA2 [1], SAC [1] |
| 2.3. | PP1 | EFF_T1 | Summary Statistics supporting Primary Analysis (Absolute and Change from Baseline): PVPI and PaO2/FiO2 (by BAL Location) | Use Alternative Treatment Group Descriptors #2 Only include timepoints associated with the primary analysis (i.e. the two assessments on Day 1: prior to surgery/post surgery). | IA2 [1], SAC [1] |
| 2.4. | PP2 | EFF_T2 | Summary of Primary Statistical Analysis: Joint Modelling of PVPI and PaO2/FiO2. | Example shell conditional on the Trt*BAL interaction term being nonsignificant. Use expert judgement to override the shell if an alternative layout is more informative / easier to review Assign a statistical analysis ID number to each analysis and page by this variable (mechanism to allow sensitivity analyses to be presented if applicable) | SAC [1] |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Second | lary Analyses | | | | |
| | Transpulmon | ary Thermodilutio | n | | |
| 2.5. | PP1 | EFF_T1 | Summary Statistics (Absolute and Change from Baseline):Transpulmonary Thermodilution (by Treatment arm) | Use Main Treatment Group Descriptors See Table 4 for endpoints (Arterial Line, Predicted body weight, predicted body surface area and body surface area only do need to be summarised at multiple timepoints). | SAC [1] |
| 2.6. | PP2 | EFF_T1 | Summary Statistics (Absolute and Change from Baseline):Transpulmonary Thermodilution (by Study Medication) | Use Alternative Treatment Group Descriptors #1 See above comments | SAC [1] |
| 2.7. | PP1 | EFF_T1 | Summary Statistics (Absolute and Change from Baseline):Transpulmonary Thermodilution (by BAL Location) | Use Alternative Treatment Group<br>Descriptors #2<br>See above comments | SAC [1] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.8. | PP2 | EFF_T2 | Summary of Statistical Analysis: Repeated Measures Joint Modelling of PVPI and PaO2/FiO2 | Example shell conditional on the Trt*BAL*Time interaction terms being non-significant. Use expert judgement to override the shell if an alternative layout is more informative / easier to review It is not possible to display all elements of the VCV from the actual MCMC modelling using this layout (e.g. the off diagonal elements across planned time). Add footnote to alert user that this has occurred. Assign a statistical analysis ID number to each analysis and page by this variable (mechanism to allow sensitivity analyses to be presented if applicable) | SAC [1] |
| 2.9. | PP2 | EFF_T5 | Summary of Statistical Analysis: Modelling of PVPI on Completion of Surgery | Example shell conditional on the Trt*BAL interaction term being non- significant. Use expert judgement to override the shell if an alternative layout is more informative / easier to review Assign a statistical analysis ID number to each analysis and page by this variable (mechanism to allow sensitivity analyses to be presented if applicable) | SAC [1] |
| 2.10. | PP2 | EFF_T5 | Summary of Statistical Analysis: Modelling of EVLWI on Completion of Surgery | See above comments | SAC [1] |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | Oxygenation | (especially P <sub>a</sub> O <sub>2</sub> /F | iO <sub>2</sub> ) | | |
| 2.11. | PP1 | EFF_T1 | Summary Statistics (Absolute and Change from Baseline):Oxygenation (by Treatment arm) | Use Main Treatment Group Descriptors See Table 4 for endpoints. Also include the imputed version of PaO2/FiO2 | SAC [1] |
| 2.12. | PP2 | EFF_T1 | Summary Statistics (Absolute and Change from Baseline): Oxygenation (by Study Medication) | Use Alternative Treatment Group<br>Descriptors #1<br>See above comments | SAC [1] |
| 2.13. | PP1 | EFF_T1 | Summary Statistics (Absolute and Change from Baseline):<br>Oxygenation (by BAL Location) | Use Alternative Treatment Group<br>Descriptors #2<br>See above comments | SAC [1] |
| 2.14. | PP2 | EFF_T5 | Summary of Statistical Analysis: Modelling of PaO2/FiO2 on Completion of Surgery | Example shell conditional on the Trt*BAL interaction term being nonsignificant. Use expert judgement to override the shell if an alternative layout is more informative / easier to review Assign a statistical analysis ID number to each analysis and page by this variable (mechanism to allow sensitivity analyses to be presented if applicable) | SAC [1] |
| | SOFA | | | | |
| 2.15. | PP2 | EFF_T1 | Summary Statistics (Absolute and Change from Baseline): Daily SOFA scores by Treatment and Time | Display Total SOFAs (observed then imputed). | SAC [1] |
| 2.16. | PP2 | EFF_T5 | Summary of Statistical Analysis of Repeated Measures Modelling of SOFA | Make appropriate modifications to account for the repeated measures | SAC [1] |

| Efficacy | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Explora | tory Analyses | | | | |
| | Clinical Outco | omes | | | |
| 2.17. | PP2 | | Summary of Diagnosed ARDS out to day 28 (by Study Medication) | Use Alternative Treatment Group Descriptors #1 | SAC [2] |
| 2.18. | PP2 | | Summary of 28 day survival status (by Study Medication) | Use Alternative Treatment Group<br>Descriptors #1 | SAC [2] |
| 2.19. | PP2 | | Summary of Organ Failure Free days out to day 28 (by Study Medication) | Use Alternative Treatment Group Descriptors #1 | SAC [2] |
| | Resource Util | isation | | · | |
| 2.20. | PP2 | | Summary of Ventilator Free Days (by Study Medication) | Use Alternative Treatment Group Descriptors #1 | SAC [2] |
| 2.21. | PP2 | | Summary of ICU Length of Stay (by Study Medication) | Use Alternative Treatment Group<br>Descriptors #1 | SAC [2] |
| 2.22. | PP2 | | Summary of Hospital Length of Stay (by Study Medication) | Use Alternative Treatment Group<br>Descriptors #1 | SAC [2] |
| Bespok | e outputs to si | upport the Interim | Analyses | | |
| 2.23. | PP2 | EFF_T3 | Summary of Futility Statistical Analysis at Interim Analysis 2 | | IA2 [1] |
| 2.24. | PP2 | EFF_T4 | Summary of Sample Size re-estimation process at Interim Analysis 2 | | IA2 [1] |

## 11.14.6. Efficacy Figures

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Primary | y Analysis | | | | |
| 2.1. | PP2 | EFF_F5 | Spaghetti plots of PVPI and PaO2/FiO2 Time Profiles (by Treatment arm) | Separate plot per endpoint. Identify subjects using the main treatment descriptors. Plot Ln(PVPI) by using Ln scale axis Only use Pre-Op and imm.Post Op timepoints | IA2 [1], SAC [1] |
| 2.2. | PP2 | EFF_F6 | Scatterplots of PVPI Vs PaO2/FiO2 by Study Medication and Timepoint | Identify subjects using the main treatment descriptors Only use Pre-Op and imm.Post Op timepoints | IA2 [1], SAC [1] |
| 2.3. | PP2 | EFF_F7 | Adjusted Medians and 95% Credible Intervals from the Marginal Posterior Distributions for each Study medication (PVPI and PaO2/FiO2) | | IA2 [1], SAC [1] |
| 2.4. | PP2 | EFF_F8 | Adjusted Medians and 95% Credible Intervals from the Marginal Posterior Distributions for Study medications comparisons (PVPI and PaO2/FiO2) | | IA2 [1], SAC[1] |
| 2.5. | PP2 | EFF_F4 | Joint Posterior Distribution and associated Marginals used to evaluate End of Study Decision Pathway | | IA2 [1], SAC[1] |
| Second | lary Analyses | | | | |
| | Transpulmon | ary Thermodilutio | n | | |
| 2.6. | PP2 | EFF_F1 | Individual Subject PVPI and EVLWI Time Profiles | Include all data for the subjects (inc<br>unscheduled). Use actual times. Try to<br>keep all endpoints on the same page<br>per subject and panel by endpoint | SAC[1] |

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.7. | PP2 | EFF_F5 | Spaghetti plots of PVPI and EVLWI Time Profiles (by Treatment arm) | Separate plot/page per endpoint. | SAC[1] |
| 2.8. | PP2 | EFF_F6 | Scatterplots of PVPI Vs PaO2/FiO2 by Study Medication and Timepoint | | SAC[1] |
| 2.9. | PP2 | EFF_F7 | Adjusted Medians and 95% Credible Intervals from the Marginal Posterior Distributions for each Study medication (PVPI and PaO2/FiO2) | Use Planned Timepoint as the x-axis of the plot but offset/group by treatment to avoid overlapping | SAC[1] |
| 2.10. | PP2 | EFF_F8 | Adjusted Medians and 95% Credible Intervals from the Marginal Posterior Distributions for Study medications comparisons (PVPI and PaO2/FiO2) | Use Planned Timepoint as the x-axis of the plot | SAC[1] |
| 2.11. | PP2 | EFF_F7 | Adjusted Medians and 95% Credible Intervals for each Study medication from the Modelling of PVPI on Completion of Surgery | | SAC[1] |
| 2.12. | PP2 | EFF_F8 | Adjusted Medians and 95% Credible Intervals for Study medication comparisons from the Modelling of PVPI on Completion of Surgery | | SAC[1] |
| 2.13. | PP2 | EFF_F7 | Adjusted Medians and 95% Credible Intervals for each Study medication from the Modelling of EVLWI on Completion of Surgery | | SAC[1] |
| 2.14. | PP2 | EFF_F8 | Adjusted Medians and 95% Credible Intervals for Study medication comparisons from the Modelling of EVLWI on Completion of Surgery | | SAC[1] |
| Oxyger | nation (especia | Ily P <sub>a</sub> O <sub>2</sub> /F <sub>i</sub> O <sub>2</sub> ) | | | |
| 2.15. | PP2 | EFF_F3 | Individual Subject Oxygenation Time Profiles | Include all data for the subjects (inc unscheduled). Use actual times. If possible put all endpoints on the same panel. Add the imputed PaO2/FiO2 profile as well. | SAC [1] |

| Efficacy | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.16. | PP2 | EFF_F5 | Spaghetti plots of PaO2/FiO2 and SpO2/FiO2 Time Profiles (by Treatment arm) | Separate plot/page per endpoint. Also add the impuited PaO2/FiO2 | SAC [1] |
| 2.17. | PP2 | EFF_F2 | Scatterplot of Observed PaO2/FiO2 and the PaO2/FiO2 value imputed from the associated SpO2/FiO2 | Only plot data where observed PaO2/FiO2 and SpO2/FiO2 data are present. Identify data points using the main treatment descriptor symbols and the b-splines using the associated line pattern. | SAC[1] |
| 2.18. | PP2 | EFF_F7 | Adjusted Medians and 95% Credible Intervals for each Study medication from the Modelling of PaO2/FiO2 on Completion of Surgery | | SAC[1] |
| 2.19. | PP2 | EFF_F8 | Adjusted Medians and 95% Credible Intervals for Study medication comparisons from the Modelling of PaO2/FiO2 on Completion of Surgery | | SAC[1] |
| SOFA | | | | | |
| 2.20. | PP2 | EFF_F1 | Individual Subject SOFA Time Profiles | Include all data for the subjects (inc unscheduled). Use actual times. | SAC [1] |
| 2.21. | PP2 | EFF_F7 /<br>EFF_F1 | Adjusted Medians and 95% Credible Intervals for each Study medication from the Repeated Measures Modelling of SOFA | Use Planned Timepoint as the x-axis of the plot but offset/group by treatment to avoid overlapping | SAC[1] |
| 2.22. | PP2 | EFF_F8 | Adjusted Medians and 95% Credible Intervals for Study medication comparisons from the Repeated Measures Modelling of SOFA | Use Planned Timepoint as the x-axis of the plot | SAC[1] |
| Explora | tory Analyses | • | | | |
| Clinical | Outcomes | | | | |
| 2.23. | PP2 | | Kaplan Meier survival curves for Day 28 Survival status (and approx 95% Cls) (by Study Medication) | Use Alternative Treatment Group<br>Descriptors #1 | SAC[2] |

## 11.14.7. Safety Tables

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 3.1. | Safety | CP_AE1p | Summary of All Serious Adverse Events (by Treatment arm) | Sort by System Organ Class Use Main Treatment Group Descriptors | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.2. | Safety | CP_AE1p | Summary of All Serious Adverse Events (by Study Medication) | Sort by System Organ Class Use Alternative Treatment Group Descriptors #1 | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.3. | Safety | CP_AE1p | Summary of All Serious Adverse Events (by BAL Location) | Sort by System Organ Class Use Alternative Treatment Group Descriptors #2 | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.4. | Safety | CP_AE1p | Summary of All Adverse Events (by Treatment arm) | Sort by System Organ Class Use Main Treatment Group Descriptors | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.5. | Safety | CP_AE1p | Summary of All Adverse Events (by Study Medication) | Sort by System Organ Class Use Alternative Treatment Group Descriptors #1 | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.6. | Safety | CP_AE1p | Summary of All Adverse Events (by BAL Location) | Sort by System Organ Class Use Alternative Treatment Group Descriptors #2 | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.7. | Safety | CP_AE1p | Summary of Drug-Related Adverse Events (by Treatment arm) | Sort by System Organ Class Use Main Treatment Group Descriptors | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.8. | Safety | CP_AE1p | Summary of Drug-Related Adverse Events (by Study Medication) | Sort by System Organ Class Use Alternative Treatment Group Descriptors #1 | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.9. | Safety | CP_AE1p | Summary of Drug-Related Adverse Events (by BAL Location) | Sort by System Organ Class Use Alternative Treatment Group Descriptors #2 | IA1 [1], IA2 [2],<br>SAC [1] |

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10. | Safety | AE2 | Relationship between System Organ Class and Verbatim Text | | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.11. | Safety | SAFE_T3 | All Non-Serious Adverse Event Counts that Occur in at least 5% of Any Treatment Group | Macro: EMA_AE | SAC [2] |
| 3.12. | Safety | SAFE_T4 | All Serious Adverse Event Counts | Macro: EMA_AE The 'Number of Related Fatalities' is only required at the Preferred Term level for reporting and is intentionally left out of the 'Any events' group | SAC [2] |
| Laborat | tory Values | | | | |
| 3.13. | Safety | LB1 | Summary of Chemistry Laboratory Values (by Treatment arm) | Exclude Pa02 from this summary Use Main Treatment Group Descriptors | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.14. | Safety | LB1 | Summary of Chemistry Laboratory Values (by Study Medication) | Exclude Pa02 from this summary Use Alternative Treatment Group Descriptors #1 | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.15. | Safety | LB1 | Summary of Chemistry Laboratory Values (by BAL Location) | Exclude Pa02 from this summary Use Alternative Treatment Group Descriptors #2 | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.16. | Safety | LB1 | Summary of Hematology Laboratory Values (by Treatment arm) | Use Main Treatment Group Descriptors | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.17. | Safety | LB1 | Summary of Hematology Laboratory Values (by Study Medication) | Use Alternative Treatment Group<br>Descriptors #1 | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.18. | Safety | LB1 | Summary of Hematology Laboratory Values (by BAL Location) | Use Alternative Treatment Group<br>Descriptors #2 | IA1 [1], IA2 [2],<br>SAC [1] |

| Safety : | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.19. | Safety | UR3b | Summary of Urinalysis Dipstick Results (by Treatment arm) | Use Main Treatment Group Descriptors Note: Consult with medical monitor to "map" results within each test to a common nomenclature prior to summarising | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.20. | Safety | UR3b | Summary of Urinalysis Dipstick Results (by Study Medication) | Use Alternative Treatment Group Descriptors #1 Note: Consult with medical monitor to "map" results within each test to a common nomenclature prior to summarising | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.21. | Safety | UR3b | Summary of Urinalysis Dipstick Results (by BAL Location) | Use Alternative Treatment Group Descriptors #2 Note: Consult with medical monitor to "map" results within each test to a common nomenclature prior to summarising | IA1 [1], IA2 [2],<br>SAC [1] |
| ECG | | | | | |
| 3.22. | Safety | EG1 | Summary of ECG Findings (by Treatment arm) | Use Main Treatment Group Descriptors | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.23. | Safety | EG1 | Summary of ECG Findings (by Study Medication) | Use Alternative Treatment Group Descriptors #1 | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.24. | Safety | EG1 | Summary of ECG Findings (by BAL Location) | Use Alternative Treatment Group Descriptors #2 | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.25. | Safety | EG2 | Summary of ECG Values (by Treatment arm) | Use Main Treatment Group Descriptors | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.26. | Safety | EG2 | Summary of ECG Values (by Study Medication) | Use Alternative Treatment Group<br>Descriptors #1 | IA1 [1], IA2 [2],<br>SAC [1] |

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.27. | Safety | EG2 | Summary of ECG Values (by BAL Location) | Use Alternative Treatment Group<br>Descriptors #2 | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.28. | Safety | EG2 | Summary of Change from Baseline in ECG Values (by Treatment arm) | Use Main Treatment Group Descriptors | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.29. | Safety | EG2 | Summary of Change from Baseline in ECG Values (by Study Medication) | Use Alternative Treatment Group Descriptors #1 | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.30. | Safety | EG2 | Summary of Change from Baseline in ECG Values (by BAL Location) | Use Alternative Treatment Group Descriptors #2 | IA1 [1], IA2 [2],<br>SAC [1] |
| Vital Sig | gns | | | | |
| 3.31. | Safety | VS1 | Summary of Vital Signs (by Treatment arm) | Use Main Treatment Group Descriptors | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.32. | Safety | VS1 | Summary of Vital Signs (by Study Medication) | Use Alternative Treatment Group<br>Descriptors #1 | IA1 [1], IA2 [2],<br>SAC [1] |
| 3.33. | Safety | VS1 | Summary of Vital Signs (by BAL Location) | Use Alternative Treatment Group Descriptors #2 | IA1 [1], IA2 [2],<br>SAC [1] |

| Safety : Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Immuno | ogenicity | | | | |
| 3.34. | Safety | IMM1 | Summary of Treatment emergent Positive Immunogenicity results (by Study Medication) | Use Alternative Treatment Group Descriptors #1 Note: The screening test results are not being databased (pre-requisite for Negative test was an inclusion criterion). Therefore this table should only contain treatment emergent positive samples | SAC [2] |

#### 11.14.8. Safety Figures

No Safety figures are currently planned. Spotfire is intended to be used in-stream to review safety data in an ongoing manner. If appropriate selected Spotfire visualisations may be reproduced within HARP.

#### 11.14.9. Pharmacokinetic Tables

| Pharmacokinetic : Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Plasma | 1 | | | | |
| 4.1. | PK | PKCT1 | Summary of Plasma GSK2862277 Pharmacokinetic Concentration – Time Data (by Treatment arm) | Use Main Treatment Group Descriptors<br>Planned time points: Day1: 0h, 1h, On<br>completion of surgery; Day 2: 24 h, Day<br>3: 48 h | SAC [1] |
| 4.2. | PK | PKCT1 | Summary of Plasma GSK2862277 Pharmacokinetic Concentration – Time Data (by Study Medication) | Use Alternative Treatment Group<br>Descriptors #2<br>Planned time points: Day1: 0h, 1h, On<br>completion of surgery; Day 2: 24 h, Day<br>3: 48 h | SAC [1] |
| 4.3. | PK | PKPT1 | Summary of Derived Plasma GSK2862277 Pharmacokinetic Parameters (by Treatment arm) | Use Main Treatment Group Descriptors | SAC [1] |
| 4.4. | PK | PKPT1 | Summary of Derived Plasma GSK2862277 Pharmacokinetic Parameters (by Study Medication) | Use Alternative Treatment Group<br>Descriptors #2 | SAC [1] |
| 4.5. | PK | PKPT3 | Summary of Derived Plasma GSK2862277 Pharmacokinetic Parameters (log transformed) (by Treatment arm) | Use Main Treatment Group Descriptors | SAC [1] |
| 4.6. | PK | PKPT3 | Summary of Derived Plasma GSK2862277 Pharmacokinetic Parameters (log transformed) (by Study Medication) | Use Alternative Treatment Group<br>Descriptors #2 | SAC [1] |
| BAL | | | | | |
| 4.7. | PK | Non-standard<br>PK_T1 | Summary of Derived Lung ELF Drug Concentrations and Volume Data (by Treatment arm) | Use Main Treatment Group Descriptors Exclude Placebo data. Only expecting pooled wash and pooled volume in this study. | SAC [1] |

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.8. | PK | Non-standard<br>PK_T1 | Summary of Derived Lung ELF Drug Concentrations and Volume Data (by Study Medication) | Use Alternative Treatment Group Descriptors #2 Exclude Placebo data. Only expecting pooled wash and pooled volume in this study. | SAC [1] |

#### 11.14.10. Pharmacokinetic Figures

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Plasma | | | | | |
| 4.1. | PK | PKCF3 | Median Plasma GSK2862277 Concentration-Time Plots (Linear and Semi-log) (by Treatment arm) | Use Main Treatment Group Descriptors Planned time points: Day1: 0h, 1h, On completion of surgery; Day 2: 24 h, Day 3: 48 h. Add a horizontal line at y-axis at LLQ and add footnote LLQ = | SAC [1] |
| 4.2. | PK | PKCF3 | Median Plasma GSK2862277 Concentration-Time Plots (Linear and Semi-log) (by Study Medication) | Use Alternative Treatment Group Descriptors #2 Planned time points: Day1: 0h, 1h, On completion of surgery; Day 2: 24 h, Day 3: 48 h. Add a horizontal line at y-axis at LLQ and add footnote LLQ = | SAC [1] |
| 4.3. | PK | PKCF1 | Individual Subject Plasma GSK2862277 Concentration – Time Plots (Linear and Semi-log) (by Treatment arm) | Use Main Treatment Group Descriptors Plot Planned time points: Day1: 0h, 1h, On completion of surgery; Day 2: 24 h, Day 3: 48 h and actual time points. Paginate by time point type. | SAC [1] |
| 4.4. | PK | PKCF1 | Individual Subject Plasma GSK2862277 Concentration – Time Plots (Linear and Semi-log) (by Study Medication) | Use Alternative Treatment Group Descriptors #2 Plot Planned time points: Day1: 0h, 1h, On completion of surgery; Day 2: 24 h, Day 3: 48 h and actual time points. Paginate by time point type. | SAC [1] |

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| BAL | | | | | |
| 4.5. | PK | Non-Standard PK_F1 (Study PII11115117 can provide examples) | Median Plasma and Individual Subject Derived Lung ELF<br>GSK2862277 Concentrations Plot (Semi-Log) (by Treatment<br>arm) | Use Main Treatment Group Descriptors Exclude Placebo data. Legend to identify subjid. Plasma based on planned rel. Time. Elf on actual rel. Time of Pooled wash. Elf data will be the pooled sample value. Include footnotes. Adjust x-axis to represent planned time points 0h, 1h, On completion of surgery; 24 h, 48 h. Use common y-axis range over this plot and the sister plot by study medication | SAC [1] |
| 4.6. | PK | Non-Standard<br>PK_F1 | Median Plasma and Individual Subject Derived Lung ELF GSK2862277 Concentrations Plot (Semi-Log) (by Study Medication) | Use Alternative Treatment Group Descriptors #2 Exclude Placebo data. Legend to identify subjid. Plasma based on planned rel. Time. Elf on actual rel. Time of Pooled wash. Elf data will be the pooled sample value. Include footnotes. Adjust x-axis to represent planned time points 0h, 1h, On completion of surgery; 24 h, 48 h. | SAC [1] |

### 11.14.11. Pharmacodynamic (Biomarker) Tables

| Pharma | Pharmacodynamic (Biomarker) : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| BAL Bi | omarkers | | | | |
| 5.1. | PP1 | EFF_T1 | Summary Statistics of BAL Biomarkers On Completion of Surgery (by Treatment arm) | No change form Baseline Add additional page by variable of the functional category of the biomarker Use Main Treatment Group Descriptors | SAC [1] |
| 5.2. | PP1 | EFF_T1 | Summary Statistics of BAL Biomarkers On Completion of Surgery (by Study Medication) | No change form Baseline Add additional page by variable of the functional category of the biomarker Use Alternative Treatment Group Descriptors #1 | SAC [1] |
| 5.3. | PP1 | EFF_T1 | Summary Statistics of BAL Biomarkers On Completion of Surgery (by BAL Location) | No change form Baseline Add additional page by variable of the functional category of the biomarker Use Alternative Treatment Group Descriptors #2 | SAC [1] |
| 5.4. | PP1 | | Summary of Statistical Analyses of BAL Biomarkers | Group by functional categories and Repeat table layouts for each BAL Biomarker Present only the final model per biomarker | SAC [1] |
| Serum | Biomarkers | | | · | |
| 5.5. | PP1 | EFF_T1 | Summary Statistics (Absolute and Change from Baseline):<br>Serum Biomarkers by Time (by Treatment arm) | Add additional page by variable of the functional category of the biomarker Use Main Treatment Group Descriptors | SAC [1] |

| Pharma | Pharmacodynamic (Biomarker) : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.6. | PP2 | EFF_T1 | Summary Statistics (Absolute and Change from Baseline):<br>Serum Biomarkers by Time (by Study Medication) | Add additional page by variable of the functional category of the biomarker Use Alternative Treatment Group Descriptors #1 | SAC [1] |
| 5.7. | PP1 | EFF_T1 | Summary Statistics (Absolute and Change from Baseline):<br>Serum Biomarkers by Time (by BAL Location) | Add additional page by variable of the functional category of the biomarker Use Alternative Treatment Group Descriptors #2 | SAC [1] |
| 5.8. | PP2 | | Summary of Statistical Analysis in Serum Biomarkers | Group by functional categories and Repeat table layouts for each BAL Biomarker Present only the final model per biomarker | SAC [1] |

### 11.14.12. Pharmacodynamic (Biomarker) Figures

| Pharma | Pharmacodynamic (and or Biomarker) : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| BAL Bi | omarkers | | | | |
| 5.1. | PP1 | | Box Plots of the BAL Biomarkers by Treatment Arm | Use imputed result. For each biomarker also plot individual data points alongside each box. Plot treatment arms side by side. Include LLQ and ULQ as reference lines where it makes sense to and footnote appropriately | SAC [1] |
| Serum | Biomarkers | | | | |
| 5.2. | PP2 | | Raw Time profiles of the Serum Biomarkers by Subject | Paginate by Treatment. For each subject plot biomarkers within a functional class on a single graph when units permit. Include LLQ and ULQ as reference lines where it makes sense to and footnote appropriately | SAC [1] |
| 5.3. | PP2 | | Spaghetti plots of the Serum Biomarkers by Treatment arm | For each biomarker plot time profiles of individuals within a treatment on a single graph. Use common axis ranges across pages/panels for each biomarker Include LLQ and ULQ as reference lines where it makes sense to and footnote appropriately | SAC [1] |

| Pharma | Pharmacodynamic (and or Biomarker) : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.4. | PP2 | | Spaghetti plots of the Serum Biomarkers by Study<br>Medication | For each biomarker plot time profiles of individuals within a study medication on a single graph. Plot study medications side by side but identify the BAL location within each study medication. Use common axis ranges across pages/panels for each biomarker Include LLQ and ULQ as reference | SAC [1] |
| | | | | lines where it makes sense to and footnote appropriately | |
| 5.5. | PP2 | | Scatterplot matrix of Serum Biomarkers by Treatment Arm | Plot all patients on same scatterplot. Indicate treatment groups by using different colours. Paginate by planned sampling times | SAC [1] |
| 5.6. | PP2 | | Scatterplot matrix of Serum Biomarkers by Time | Plot all patients and time points on same scatterplot. Indicate individual timepoints by using different colours. Paginate by Treatment Arm | SAC [1] |
| 5.7. | PP2 | EFF_F7 /<br>EFF_F1 | Adjusted Medians and 95% Credible Intervals for each Study medication from the Repeated Measures Modelling of Serum Biomarkers | Repeat for each biomarker Use Planned Timepoint as the x-axis of the plot but offset/group by treatment to avoid overlapping | |
| 5.8. | PP2 | EFF_F8 | Adjusted Medians and 95% Credible Intervals for Study medication comparisons from the Repeated Measures Modelling of Serum Biomarkers | Repeat for each biomarker Use Planned Timepoint as the x-axis of the plot | |

### 11.14.13. Pharmacogenetic Tables

| Pharmacogenetic : Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | cogenetics | | | | |
| 6.1. | 6.1 Safety GN1 Summary of Genetics Subject Accountability SAC [2] | | | | |
| 6.2. | 6.2 Safety GN2 Summary of Genetic Consent Not Obtained / Withdrawn SAC [2] | | | | |

#### 11.14.14. ICH Listings

| ICH : L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Accountabilit | y | | , | |
| 1. | n/a | POP_L1 | Listing of Subject Accountability (subjects constituting each Statistical Analysis Population) | Also list out the subject IDs who will participate in the Translational Sub-Study | IA1 [1], IA2 [2],<br>SAC [1] |
| Rando | misation | | | | |
| 2. | Safety | CP_TA1 | Listing of Randomised and Actual Treatments | Omit cohort column Include Site ID Include Randomisation number and Randomisation Date/Time (if only date available then modify column labels) Split Actual Treatment column into two separate columns ("Actual Study Medication" and "Actual BAL Sampled") Create corresponding Deviation columns for each actual treatment column | IA1 [1], IA2 [2],<br>SAC [1] |
| 3. | Safety | BL1 | Listing of Subjects for whom Treatment Blind was Broken (excluding when broken to support the interim analyses) | | SAC [2] |
| Subjec | t Disposition | | | | |
| 4. | Screen<br>Failures | ES7 | Listing of Reasons for Screening Failure | See notes for corresponding summary table | SAC [2] |
| 5. | Safety | DV2 | Listing of Important Protocol Deviations | Add additional columns to cover the 3x per protocol populations | IA1 [1], IA2 [2],<br>SAC [1] |
| 6. | Safety | IE3 | Listing of subjects with Inclusion/Exclusion Criteria Deviations | | SAC [1] |

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 7. | Safety | CP_ES10x | Listing of Subjects who Withdrew from Study | Modify the contents and re-label the cross over related column names as appropriate to a parallel group design. Keep the date of last contact. | SAC [2] |
| Demog | graphy | | | | |
| 8. | Safety | DM2 | Listing of Demographic Characteristics | | IA1 [1], IA2 [2],<br>SAC [1] |
| 9. | Safety | DM9 | Listing of Race | | IA1 [1], IA2 [2],<br>SAC [1] |
| Medica | al Condition & C | oncomitant Medi | cations | • | |
| 10. | Safety | MH2 | Listing of Current and Past Medical Conditions | Combine both current and past items into one listing | IA1 [1], IA2 [2],<br>SAC [1] |
| 11. | Safety | CP_CM3 | Listing of Concomitant Medications by Generic Term | | IA1 [1], IA2 [2],<br>SAC [1] |
| Expos | ure | | | | |
| 12. | Safety | EX3 | Listing of Exposure Data | | SAC [2] |
| Advers | se Events | | | • | |
| 13. | Safety | CP_AE8a | Listing of All Serious Adverse Events | | IA1 [1], IA2 [2],<br>SAC [1] |
| 14. | Safety | CP_AE8 | Listing of All Adverse Events | | IA1 [1], IA2 [2],<br>SAC [1] |
| 15. | Safety | CP_AE8 | Listing of Adverse Events Leading to Withdrawal from Study | | IA1 [1], IA2 [2],<br>SAC [1] |
| 16. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | IA1 [1], IA2 [2],<br>SAC [1] |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | Laboratory Values | | | | |
| 17. | Safety | CP_LB5 | Listing of Clinical Chemistry Abnormalities of Potential Clinical Importance | | IA1 [1], IA2 [2],<br>SAC [1] |
| 18. | Safety | CP_LB5 | Listing of All Clinical Chemistry Laboratory Data for Subjects with PCI Abnormalities | | IA1 [1], IA2 [2],<br>SAC [1] |
| 19. | Safety | CP_LB5 | Listing of Hematology Abnormalities of Potential Clinical Importance | | IA1 [1], IA2 [2],<br>SAC [1] |
| 20. | Safety | CP_LB5 | Listing of All Hematology Laboratory Data for Subjects with PCI Abnormalities | | IA1 [1], IA2 [2],<br>SAC [1] |
| 21. | n/a | LB13 | Listing of Laboratory Tests and Associated Reference Ranges | Add centre/site column if necessary to distinguish different sets of normal ranges (and add corresponding date range(s) if normal ranges have changed within a site during conduct of study) | IA1 [1], IA2 [2],<br>SAC [1] |
| 22. | Safety | Base on AE2 | Relationship between Urinalysis Summary Table Categories and Verbatim Text | Describes the mapping of test results to categories used in corresponding summary table. Base on AE2 shell (System Organ class becomes the Lab test name, Preferred term becomes the Category result was mapped onto) | IA1 [1], IA2 [2],<br>SAC [1] |
| ECG | | | | | |
| 23. | Safety | CP_EG3 | Listing of All ECG Values for Subjects with any Value of Potential Clinical Importance | | IA1 [1], IA2 [2],<br>SAC [1] |
| 24. | Safety | CP_EG3 | Listing of ECG Values of Potential Clinical Importance | | IA1 [1], IA2 [2],<br>SAC [1] |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 25. | Safety | CP_EG5 | Listing of Abnormal ECG Findings | | IA1 [1], IA2 [2],<br>SAC [1] |
| Vital Sig | gns | | | | |
| 26. | Safety | CP_VS4 | Listing of Vital Signs of Potential Clinical Importance | | IA1 [1], IA2 [2],<br>SAC [1] |
| 27. | Safety | CP_VS4 | Listing of All Vital Signs of for Subjects with any Value of Potential Clinical Importance | | IA1 [1], IA2 [2],<br>SAC [1] |
| Immund | Immunogenicity | | | | |
| 28. | Safety | IMM2 | Listing of Immunogenicity results | Omit drug concentration units column. Omit titre column if not applicable to observed data. | SAC [2] |

#### 11.14.15. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Efficacy Endpoints | | | | | |
| 29. | Safety | EFF_L2 | Listing of Transpulmonary Thermodilution Data | | IA2 [1] SAC [1] |
| 30. | Safety | EFF_L3 | Listing of Oxygenation Data | | IA2 [1] SAC [1] |
| 31. | Safety | EFF_L3 | Listing of Change from Baseline Oxygenation Data | Keep Baseline record (actual values)<br>but post baseline entries should contain<br>the change values (Vent mode changes<br>should be flagged) | IA2 [1] SAC [1] |
| 32. | Safety | EFF_L4 | Listing of SOFA Data | | SAC [1] |
| 33. | PP2 | Non-standard | SAS Output from Primary Statistical Analysis: Joint Modelling of PVPI and PaO2/FiO2. | | SAC [1] |
| 34. | PP2 | Non-standard | SAS Output from Statistical analysis: Modelling of PVPI on Completion of Surgery | | SAC [1] |
| 35. | PP2 | Non-standard | SAS Output from Statistical analysis: Modelling of PaO2/FiO2 on Completion of Surgery | | SAC [1] |
| 36. | PP2 | Non-standard | SAS Output from Statistical analysis: Modelling of EVLWI on Completion of Surgery | | SAC [1] |
| 37. | PP2 | Non-standard | SAS Output from Statistical analysis: Repeated Measures Modelling of SOFA | | SAC [1] |
| 38. | PP2 | Non-standard | SAS Output from PROC MCMC Futility analysis at Interim Analysis 2 | Interim analysis #2 only. | IA2 [1] |
| 39. | PP2 | Non-standard | SAS Output from Sample Size Re-estimation at Interim Analysis 2 | Interim analysis #2 only. | IA2 [1] |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Surgica | l Procedure | | | | |
| 40. | Safety | EFF_L1 | Listing of Information relating to the surgical procedure by Subject | New page per subject. Group and order subjects by Treatment, Centre and ID | IA1 [1], IA2 [2],<br>SAC [1] |
| PK (Pla | sma and BAL) | | | | |
| 41. | PK | PKCL1p | Listing of GSK2862277 Plasma Pharmacokinetic Concentration - Time Data | Use Main Treatment Descriptors | SAC [1] |
| 42. | PK | PKPL1p | Listing of Derived GSK2862277 Plasma Pharmacokinetic Parameters | Use Main Treatment Descriptors | SAC [1] |
| 43. | PK | PKLU1p | Listing of Derived GSK2862277 Lung ELF concentrations | Use Main Treatment Descriptors | SAC [1] |
| 44. | PK | Non-standard | Listing of Data required to obtain Lung ELF concentrations | Use Main Treatment Descriptors Create bespoke by-subject listing that includes the BAL Drug concentration, Plasma Urea and BAL Urea, dilution factor, Volume of ELF, Volume of BAL and Total drug in BAL fluid | SAC [1] |
| Pharma | codynamic (ar | nd or Biomarker) | | | |
| | BAL Biomark | ers | | | |
| 45. | Safety | | Listing of BAL Biomarker data | | SAC [1] |
| 46. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker Free sTNFR1 | | SAC [1] |
| 47. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker Total sTNFR1 | | SAC [1] |
| 48. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker Complex sTNFR1 | | SAC [1] |
| 49. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker TNFa | | SAC [1] |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 50. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker IL-6 | | SAC [1] |
| 51. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker IL-8 | | SAC [1] |
| 52. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker IL-1b | | SAC [1] |
| 53. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker MCP-1 | | SAC [1] |
| 54. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker CRP | | SAC [1] |
| 55. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker IL1-ra | | SAC [1] |
| 56. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker IL-10 | | SAC [1] |
| 57. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker Total Protein | | SAC [1] |
| 58. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker SP-D | | SAC [1] |
| 59. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker RAGE | | SAC [1] |
| 60. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker CC16 | | SAC [1] |
| 61. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker vWF | | SAC [1] |
| 62. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker sICAM-1 | | SAC [1] |
| 63. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker MPO | | SAC [1] |
| 64. | PP1 | Non-standard | SAS Output from Statistical Modelling of BAL biomarker Total Protein Ratio | | SAC [1] |
| Serum | Biomarkers | | | • | , |
| 65. | Safety | | Listing of Serum Biomarker data | | SAC [1] |
| 66. | PP2 | Non-standard | SAS Output from Statistical Modelling of Serum biomarker Free sTNFR1 | | SAC [1] |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 67. | PP2 | Non-standard | SAS Output from Statistical Modelling of Serum biomarker Total sTNFR1 | | SAC [1] |
| 68. | PP2 | Non-standard | SAS Output from Statistical Modelling of Serum biomarker Complex sTNFR1 | | SAC [1] |
| 69. | PP2 | Non-standard | SAS Output from Statistical Modelling of Serum biomarker IL-6 | | SAC [1] |
| 70. | PP2 | Non-standard | SAS Output from Statistical Modelling of Serum biomarker IL-8 | | SAC [1] |
| 71. | PP2 | Non-standard | SAS Output from Statistical Modelling of Plasma biomarker CRP | | SAC [1] |
| 72. | PP2 | Non-standard | SAS Output from Statistical Modelling of Plasma biomarker Total Protein | | SAC [1] |
| 73. | PP2 | Non-standard | SAS Output from Statistical Modelling of Serum biomarker SP-D | | SAC [1] |
| 74. | PP2 | Non-standard | SAS Output from Statistical Modelling of Serum biomarker RAGE | | SAC [1] |
| 75. | PP2 | Non-standard | SAS Output from Statistical Modelling of Serum biomarker CC16 | | SAC [1] |
| 76. | PP2 | Non-standard | SAS Output from Statistical Modelling of Serum biomarker vWF | | SAC [1] |
| 77. | PP2 | Non-standard | SAS Output from Statistical Modelling of Serum biomarker sICAM-1 | | SAC [1] |
| 78. | PP2 | Non-standard | SAS Output from Statistical Modelling of Serum biomarker MPO | | SAC [1] |
| Explor | atory | | | | • |
| 79. | Safety | EFF_L7 | Listing of Subjects Diagnosed with ARDS out to day 28 | | SAC [2] |
| 80. | Safety | EFF_L5 | Listing of day 28 survival status | | SAC [2] |
| 81. | Safety | EFF_L6 | Listing of Organ Failure Free days | Keep Subject and metadata and replace Vent free days with Organ failure free days | SAC [2] |
| 82. | Safety | EFF_L6 | Listing of day 28 Resource Usage | | SAC [2] |

#### 11.15. Appendix 15: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request


TFR116341

#### **Appendix 15: Example Mock Shells for Data Displays**

Example : PK\_T1 Page 1 of n

Protocol : TFR116341
Population : Pharmacokinetic

# Table X.X Summary of Derived Lung ELF Drug Concentrations and Volume Data

Treatment: 26.0 mcg

Planned 90% CI Relative Geometric Time Ν Mean (Lower, Upper) SD Logs CVb (%) ELF Drug Day 1(1) 10 110133.4 (52983.6,228927.1)1.09 151.6 Conc (pg/mL) Day 1(2) 10 63196.2 (40464.7,98697.4)0.66 74.7 Day 1(3) 48241.2 (35806.4,64994.2) 0.44 10 46.8 Pooled ELF Drug Day 1 10 55374.3 (39768.3,77104.4) 0.49 52.6 Conc (pg/mL) (Pooled Washes) Volume of ELF Day 1 (1) 10 0.0330 (0.0164, 0.0662)1.042 140.1 in BAL Fluid (mL) Day 1(2) 10 0.0996 (0.0526, 0.1886)0.953 121.6 Day 1(3) 0.1970 (0.1000, 0.3882)1.012 10 133.7
Example : PK\_F1 Page 1 of n

Protocol :TFR116341
Population : Pharmacokinetic

Table X.X

Median Plasma and Individual Subject Derived Lung ELF GSK2862277 Concentrations Plot (Semi-Log) Pooled Washes



PPD Subjid

TFR116341

: EFF\_T1 Example

Page 1 of 34 Protocol: TFR116343

Population: Biomaker Table 12.1

Summary of Raw Immune Function Biomarker data and change from Baseline

Endpoint (unit): PVPI (xxx)

| Planned n Visit Relative imp Mean | Min | |
|---|---|---|
| Treatment N Item [1] Time n [2] [3] 95% CI of Mean SD Median | [4] | Max |
| 0.002 6 Analyte P1D1 PRE-DOSE 6 0 8.40 (6.65, 10.15) 1.664 8.60 mg/kg IV numeric (BL) sD result | 5.6 | 10.5 |
| 2 HOUR 6 0 7.95 (6.17, 9.73) 1.697 7.55 | 5.8 | 10.8 |
| 6 HOUR 6 0 8.30 (5.88, 10.72) 2.308 7.40 | 6.2 | 11.9 |
| 24 HOUR 6 0 9.03 (6.46, 11.60) 2.449 8.80 | 6.3 | 12.1 |
| 48 HOUR 6 0 8.42 (5.99, 10.84) 2.309 7.90 | 5.7 | 11.8 |
| Change P1D1 2 HOUR 6 0 -4.86 (-15.68, 5.97) 10.318 -1.37 from Baseline | -23.4 | 3.6 |
| 6 HOUR 6 0 -0.79 (-20.78, 19.20) 19.046 0.20 | -21.3 | 19.5 |
| 24 HOUR 6 0 7.47 (-11.68, 26.62) 18.245 7.09 | -18.2 | 33.3 |
| 48 HOUR 6 0 -0.19 (-15.45, 15.07) 14.543 -2.64 | -16.0 | 20.7 |

<sup>[1]</sup> P=Study Part, D=Study day relative to 1st dose

Programming Notes: Paginate by endpoint. Indicate the baseline timepoint (e.g. suffix with "(BL)"). If no imputations for the endpoints then drop the nimp column and any associated footnotes. Modify as appropriate to the endpoint(s) being summarised.

<sup>[2]</sup> Number of imputed observations (imputed using 1/2 of the LLQ)

<sup>[3]</sup> NA = Not Applicable (due to  $\geq$  75% of values being LLQ )

<sup>[4]</sup> NC = Non-Calculable (due to presence of LLQ values)

Example : EFF\_T1 (contd)

Protocol: TFR116343 Page 2 of 34

Population: Biomaker

Table 12.1

Summary of Raw Immune Function Biomarker data and percentage change from Baseline

Endpoint (unit): PVPI (xxx)

| Treatment | · | Item | Visit<br>[1] | Planned<br>Relative<br>Time | n<br> | n<br>imp<br>[2] | Geo.<br>Mean | 95% CI of Geo.<br>Mean | SD<br>Logs | CV (%) |
|---|---|---|---|---|---|---|---|---|---|---|
| 0.002<br>mg/kg IV<br>SD | 6 | Analyte numeric result | P1D1 | PRE-DOSE<br>(BL) | 6 | 0 | 8.25 | (6.57, 10.35) | 0.216 | 21.9 |
| | | | | 2 HOUR | 6 | 0 | 7.81 | (6.27, 9.72) | 0.209 | 21.1 |
| | | | | 6 HOUR | 6 | 0 | 8.05 | (6.11, 10.62) | 0.263 | 26.8 |
| | | | | 24 HOUR | 6 | 0 | 8.76 | (6.56, 11.69) | 0.275 | 28.0 |
| | | | | 48 HOUR | 6 | 0 | 8.16 | (6.14, 10.85) | 0.272 | 27.7 |
| | | Change<br>from<br>Baseline | P1D1 | 2 HOUR | 6 | 0 | NA | NA | NA | NA |
| | | | | 6 HOUR | 6 | 0 | NA | NA | NA | NA |
| | | | | 24 HOUR | 6 | 0 | NA | NA | NA | NA |
| | | | | 48 HOUR | 6 | 0 | NA | NA | NA | NA |

<sup>[1]</sup> P=Study Part, D=Study day relative to 1st dose

<sup>[2]</sup> Number of imputed observations (imputed using 1/2 of the LLQ)

<sup>[3]</sup> NA = Not Applicable (due to  $\geq$  75% of values being LLQ )

<sup>[4]</sup> NC = Non-Calculable (due to presence of LLQ values)

TFR116341

Example : EFF\_T2
Protocol: TFR116341

Protocol: TFR116341


Population: Safety

Table 12.207

Summary of Primary Statistical Analysis: Joint Modelling of PVPI and PaO2/FiO2.

------ Statistical Analysis ID=1 ------

| Treatment | N | Planned.<br>Relative<br>Time | Endpoint | n | Sample<br>Mean<br>Vector | Sample<br>Variance<br>Matrix | Covariance | Sample<br>Correlation |
|---|---|---|---|---|---|---|---|---|
| Placebo (BAL Collapsed lung) | 20 | Pre-Op (BL) | Ln{PVPI}<br>PaO2/FiO2 | XX<br>XX | XX.X<br>XX.X | XX.XXX<br>XX.XXX | XX.XXX<br>XX.XXX | x.xx |
| | | Imm. Post Op. | <pre>Ln{PVPI} Pa02/Fi02</pre> | | XX.X<br>XX.X | XX.XXX<br>XX.XXX | XX.XXX<br>XX.XXX | X.XX |
| Placebo (BAL Ventilated lung) | 20 | Pre-Op (BL) | Ln{PVPI}<br>PaO2/FiO2 | XX<br>XX | XX.X<br>XX.X | XX.XXX<br>XX.XXX | XX.XXX<br>XX.XXX | X.XX |
| | | Imm. Post Op. | Ln{PVPI}<br>PaO2/FiO2 | | XX.X<br>XX.X | XX.XXX<br>XX.XXX | XX.XXX<br>XX.XXX | X.XX |
| GSK2862277 26mg IH (BAL Collapsed lung) | 20 | Pre-Op (BL) | Ln{PVPI}<br>PaO2/FiO2 | XX<br>XX | XX.X<br>XX.X | XX.XXX<br>XX.XXX | XX.XXX<br>XX.XXX | X.XX |
| | | Imm. Post Op. | Ln{PVPI}<br>PaO2/FiO2 | | XX.X<br>XX.X | XX.XXX<br>XX.XXX | XX.XXX<br>XX.XXX | X.XX |

Example : EFF\_T2 (Contd)

Protocol: TFR116341 

Population: Safety

Table 12.207

Summary of Primary Statistical Analysis: Joint Modelling of PVPI and PaO2/FiO2.

------ Statistical Analysis ID=1 ------

| Item | Planned.<br>Relative<br>Time | Endpoint | Median<br>Mean<br>Vector | Median<br>Variance<br>Matrix | Covariance | Median<br>Correlation |
|---|---|---|---|---|---|---|
| Adjusted Placebo (averaging over BAL) | Imm. Post Op. | Ln{PVPI}<br>PaO2/FiO2 | XX.X<br>XX.X | XX.XXX<br>XX.XXX | XX.XXX<br>XX.XXX | X.XX |
| Adjusted Active (averaging over BAL) | Imm. Post Op. | Ln{PVPI}<br>PaO2/FiO2 | XX.X<br>XX.X | XX.XXX<br>XX.XXX | XX.XXX<br>XX.XXX | X.XX |
| Adjusted Active Vs Placebo<br>Joint Distribution<br>(averaging over BAL) | Imm. Post Op. | PVPI Ratio<br>PaO2/FiO2 Diff | XX.X<br>XX.X | XX.XXX<br>XX.XXX | XX.XXX<br>XX.XXX | X.XX |

TFR116341

Example : EFF\_T2 (Contd)

Protocol: TFR116341 

Population: Safety

Table 12.207

Summary of Primary Statistical Analysis: Joint Modelling of PVPI and PaO2/FiO2.

------ Statistical Analysis ID=1 ------

| Item<br>(units) | Planned.<br>Relative<br>Time | Median | 95% Credible<br>Interval | MCSE/SD |
|---|---|---|---|---|
| Adjusted Pbo PVPI averaging over BAL (xxx) | Imm. Post Op. | XX.XX | (X.XXX, XX.XXX) | X.XXX |
| Adjusted Pbo PaO2/FiO2 averaging over BAL (kPa) | Imm. Post Op. | XX.XX | (X.XXX, XX.XXX) | X.XXX |
| Adjusted Act PVPI averaging over BAL (xxx) | Imm. Post Op. | XX.XX | (X.XXX, XX.XXX) | X.XXX |
| Adjusted Act PaO2/FiO2 averaging over BAL (kPa) | Imm. Post Op. | XX.XX | (X.XXX, XX.XXX) | X.XXX |

Note: Values used for continuous covariates in model adjustment: Baseline PVPI = xxx (unit), Baseline PaO2/FiO2 = xxx (unit), Age = 36 Years, Height = xx cm, etc

TFR116341

Example : EFF\_T2 (contd)

Protocol: TFR116341 

Population: Safety

Table 12.207

Summary of Primary Statistical Analysis: Joint Modelling of PVPI and PaO2/FiO2.

------ Statistical Analysis ID=1 ------

| <pre>Item (units)</pre> | Planned.<br>Relative<br>Time | Median | 95% Credible<br>Interval | MCSE/SD |
|---|---|---|---|---|
| Ratio of Act/Pbo PVPI averaging over BAL | Imm. Post Op. | XX.XX | (X.XXX, XX.XXX) | x.xxx |
| Difference Act-Pbo P/F averaging over BAL (kPa) | Imm. Post Op. | XX.XX | (X.XXX, XX.XXX) | X.XXX |

Note: Values used for continuous covariates in model adjustment: Baseline PVPI = xxx (unit), Baseline PaO2/FiO2 = xxx (unit), Age = 36 Years, Height = xx cm, etc

TFR116341

Example : EFF\_T2 (contd)

Protocol: TFR116341 

Population: Safety

Table 12.207

Summary of Primary Statistical Analysis: Joint Modelling of PVPI and PaO2/FiO2.

------ Statistical Analysis ID=1 ------

| End of Study Decision Pathway | Criteria | Threshold<br>Probability | Observed<br>Probability | Met |
|---|---|---|---|---|
| Outcome 1: Robust Success | Pr(PVPI ratio (A/P) < 0.884 AND PaO2/FiO2 Diff (A-P) >= 5.3 kPa) | 0.25 | 0.0328 | N |
| Outcome 2: Success | Pr(PVPI ratio (A/P) < 0.884) | 0.35 | 0.0856 | N |
| Outcome 3: Potentially Unsuccessful | Pr(PVPI ratio (A/P) >= 0.884) | 0.75 | 0.9144 | Y |
| OVERALL END OF STUDY OUTCOME | Potentially Unsuccessful | | | |

#### PPD

**Programming note:** Use more appropriate descriptors for the labels (e.g. update when timeslicing keys are set). Add any other posterior probability statements in a similar manner to those in GSK2586881 ACE114622 (e.g. PD Table 12.207), for example....

| (units) | Comparison | Posterior Probability Statement | Value |
|---|---|---|---|
| XXXXX | (Act / Pbo) Imm. Post Op. | < 0.10 i.e. More than 90% reduction | 0.0740 |

TFR116341


Example : EFF\_T3
Protocol : TFR116341
Population : Safety

Table X.XX

#### The SAS System

#### TFR116341 Interim Analysis 2 (IA2) Statistical Analysis Outcome

"PAUSE and REVIEW"

Number of Observed Placebo Subjects at IA2 = 22

Number of Observed Active Subjects at IA2 = 18

Number of Placebo Subjects required (per simulated dataset) to reach end of study target of 40 = 18

Number of Active Subjects required (per simulated dataset) to reach end of study target of 40 = 22

Number of simulated datasets = 1000

Futility criteria for each simulated dataset: If the joint probability of  $\{Any\ Decrease\ in\ P/F\ AND\ Any\ Increase\ in\ PVPI\}\ is > 0.1$  then simulated study is futile

If the proportion of future simulated datasets meeting futility criteria is > 0.3 then statistical analysis recommendation is to "Pause and Review", otherwise recommendation is to "Continue"

Note: As per protocol, this statistical analysis recommendation is not binding and may be over-ruled by expert judgement of GSK Study Team if deemed appropriate

Proportion of future datasets meeting futility criteria = 0.932, therefore...

Statistical analysis recommendation is to "PAUSE and REVIEW"

TFR116341

Example : EFF\_T4 Page 1 of n

Protocol : TFR116341 Population : Safety

Table X.XX

Precise specification up to the expert judgement of the statistician/programmer. Should contain...

Selected SAS output from sample size re-estimation procedure: Assumed VCV matrix used in protocol, the estimated VCV matrix from the IA2 data, and the recommended number of subjects and the operating characteristics under the re-estimated number assuming a Null and Minimum desired profile for the remaining (unobserved) subjects

>>>

TFR116341

Example : EFF\_T5

Protocol: TFR116341 

Population: Safety

Table 12.207

Summary of Statistical Analysis: Modelling of PVPI on Completion of Surgery.

------ Statistical Analysis ID=1 ------

| Item (units) | Planned.<br>Relative<br>Time | Median | 95% Credible<br>Interval | MCSE/SD |
|---|---|---|---|---|
| Adjusted Pbo PVPI averaging over BAL (xxx) | Imm. Post Op. | XX.XX | (X.XXX, XX.XXX) | X.XXX |
| Adjusted Act PVPI averaging over BAL (xxx) | Imm. Post Op. | XX.XX | (X.XXX, XX.XXX) | X.XXX |

Note: Values used for continuous covariates in model adjustment: Baseline PVPI = xxx (unit), Baseline PaO2/FiO2 = xxx (unit), Age = 36 Years, Height = xx cm, etc

TFR116341

Example : EFF\_T5 (contd)

Protocol: TFR116341 

Population: Safety

Table 12.207

Summary of Statistical Analysis: Modelling of PVPI on Completion of Surgery.

------ Statistical Analysis ID=1 ------

Planned.

Item Relative 95% Credible (units) Time Median Interval MCSE/SD Ratio of Act/Pbo PVPI averaging over BAL Imm. Post Op. XX.XX (X.XXX, XX.XXX) X.XXX

Note: Values used for continuous covariates in model adjustment: Baseline PVPI = xxx (unit), Baseline PaO2/FiO2 = xxx (unit), Age = 36 Years, Height = xx cm, etc

TFR116341

Example : EFF\_T5 (contd)

Protocol: TFR116341 

Population: Safety

Table 12.207

Summary of Statistical Analysis: Modelling of PVPI on Completion of Surgery.

------ Statistical Analysis ID=1 ------

Item

| (units) | Comparison | Posterior Probability Statement | Value |
|---|---|---|---|
| Ratio of Act/Pbo | (Act / Pbo) Imm. Post Op. | < 1.00 i.e. Any reduction | 0.6740 |
| PVPI averaging over BAL | | < 0.10 i.e. More than 90% reduction | 0.0740 |

## PPD

**Programming note:** Use more appropriate descriptors for the labels (e.g. update when timeslicing keys are set). Add any other posterior probability statements in a similar manner to those above


Protocol : TFR116341 Population : Safety

Figure X.XX




Protocol : TFR116341 Population : Safety

Figure X.XX



Page 3 of 59

Protocol : TFR116341

Protocol : TFR11 Population : Safety

Figure X.XX
Protocol: AL1111592
Population: All Subjects

Figure 10.998
By Subject Time Profiles of SaO2, PaO2, FiO2 and P/F ratio



Note: RA = Room Air, NP = Nasal Prongs, FM = Face Mask and VT = Ventilator. Dashed lines left axis, Solid lines right axis Note: NA = Not Applicable (not on Ventilator), IMV = IMV/sIMV, PCV = Pressure controlled ventilation, PS = Pressure support N ote: NI PPV = Non-invasive positive pressure ventilation and Other = Other method (see listings for details) PPD

: EFF\_F4 Page 1 of n Example

Protocol : TFR116341 Population : Safety






Example : EFF\_F5
Protocol : TFR116341
Population : Safety




Example : EFF\_F6
Protocol : TFR116341
Population : Safety




Example : EFF\_F7
Protocol : TFR116341
Population : Safety



Protocol : TFR116341

Protocol : TFR110 Population : Safety



TFR116341


Protocol : TFR116341 Population : Safety

Listing X.XX

Actual Treatment: Placebo BAL Collapsed Lung, Subject ID xxx, (Inv ID: xxx)

#### Subject Demographics

Derived Age

Sex

Race

#### Subject Background

```
Prior Oesophageal Chemotherapy : [No] or [Yes and end date of treatment]

Smoking History: [Never Smoked] or [Current Smoker] or [Former Smoker and date last smoked]

Medical History: {Exclude the GSK cardiovascular risk factor items, Group by Past and Current}
```

#### Study treatment

Actual Study Drug received: [Name and date/time of Start of nebulisation]

#### Oesophagectomy procedure

```
Type of Surgery: [Trans Thoracic Oesophagectomy] or [Free text box from eCRF]

Start (rel to Dosing): [Start date and time of procedure] ([Start of procedure relative to dosing (hh:mm)])

Stop (rel to Dosing): [Stop date and time of procedure] ([End of procedure relative to dosing (hh:mm)])

Duration of Oesophagectomy procedure: [Duration of procedure (hh:mm)]

Did subject receive blood transfusion (amount and units): [Yes: amount and units] or [No]
```

#### Ventilation: Two Lung Ventilation

TFR116341

Example : EFF\_L1 (Contd) Page 1 of n

Protocol : TFR116341 Population : Safety

# Listing X.XX

# Actual Treatment: Placebo BAL Collapsed Lung, Subject ID xxx, (Inv ID: xxx)

All information from "Two-lung ventilation (At start of ventilation)" item of eCRF: [Mode of Ventilation, Tidal Volume, PEEP, Peal Pressure and Plateau Pressure]

Did ventilation continue post surgery: [No] or [Yes and Mode of ventilation]

### Ventilation: One Lung Ventilation (OLV)

Start of OLV (rel to Dosing and Surgery): [Start date and time of OLV] ([Start of OLV relative to dosing (hh:mm)], [Start rel' to surgery (hh:mm)])

End of OLV: [End date/time of OLV] ([End of OLV relative to dosing (hh:mm)], [End rel' to surgery (hh:mm)])

Duration of One Lung Ventilation: [Duration of One Lung ventilation (hh:mm)]

All information from "One-lung ventilation (baseline)" item of eCRF: [Mode of Ventilation, Tidal Volume, PEEP, Peal Pressure and Plateau Pressure]

#### Anaesthetic

Start of anaesthia (rel to Dosing and Surgery): [Start date and time of anaesthia] ([Start of anaesthia relative to dosing (hh:mm)],[Start rel' to surgery (hh:mm)])

End of anaesthia (rel to Dosing and Surgery): [End of anaesthia], [End of anaesthia relative to dosing (hh:mm)], [End rel' to surgery (hh:mm)]

Duration of anaesthia: [Duration of anaesthia (hh:mm)]

Anaesthetic and operative agents: [Epidural Anasthesia] or [free text box from eCRF]

Method of maintenance: [Volatile anaesthetic] or [TIVA]

Was Inotrope used intra-op?: [No] or [Drug Used and For how long (hh:mm)]

Was Inotrope used post-op?: [No] or [Drug Used and For how long (hh:mm)]

TFR116341

Example : EFF\_ L1 (Contd) Page 1 of n

Protocol: TFR116341

Population : Safety Listing X.XX

Actual Treatment: Placebo BAL Collapsed Lung, Subject ID xxx, (Inv ID: xxx)

#### BAL Procedure

```
Start of BAL (rel to Dosing and Surgery): [Start date and time of BAL] ([Start of BAL relative to dosing (hh:mm)], [Start rel' to surgery (hh:mm)])

Lung BAL performed on: [Left] or [Right]

Actual Lung BAL performed on: [Deflated (Collapsed)] or [Inflated (Ventilated)]
```

#### Fluid balance in 24hr period from start of surgery

```
Fluid intake start date/time: [Fluid intake start date/time]

Fluid intake stop date/time: [Fluid intake stop date/time]

Total Input (ml): [Total input]

Total Output (ml): [Total output]

Net total: [Derived as Total Input - Total Output]

Urine Output (ml): [Urine output]

Other Output (ml): [Other output]
```

#### Post operative complications

```
Did the subject receive antibiotics for a suspected respiratory tract infection?: [Yes] or [No]

Did the subject develop a significant pleural effusion?: [Yes] or [No]

Did the subject develop an Empyema?: [Yes] or [No]

Did the patient suffer from aspiration pneumonitis?: [Yes] or [No]
```

Example : EFF\_L2
Protocol : TFR116341
Population : Safety


Listing X.XX
Listing of Transpulmonary Thermodilution Data

| Treatment/<br>Inv ID/<br>Subject | Weight (kg)/ Pred. Weight (kg)/ Pred. BSA (m**2) | Visit /<br>Planned<br>Relative<br>Time | Actual Date/Time | Time since<br>start of<br>Surgery | Item (units) | Result | Change from<br>Baseline (BL) |
|---|---|---|---|---|---|---|---|
| Placebo (BAL<br>Collapsed<br>lung)/<br>PPD | 89/<br>100/<br>233 | Day 1 /<br>Imm. Prior<br>to Surgery<br>(BL) | DDMMMYYY /<br>HH:MM | +/- XXh<br>XXm | Arterial Line used | Femoral | n/a |
| | | | | | Cardiac output rep1 (xxx) Cardiac output rep2 (xxx) Cardiac output rep3 (xxx) Cardiac output Mean (xxx) Mean Arterial Pressure (xxx) etc | XX<br>XX<br>XX<br>XX<br>XX | n/a<br>n/a<br>n/a<br>n/a<br>n/a |
| | | Day 1 /<br>Imm. Post<br>Surgery | DDMMMYYY /<br>HH:MM | +/- XXh<br>XXm | Arterial Line used | Femoral | |
| | | | | | Cardiac output rep1 (xxx) Cardiac output rep2 (xxx) Cardiac output rep3 (xxx) Cardiac output Mean (xxx) Mean Arterial Pressure (xxx) | XX<br>XX<br>XX<br>XX<br>XX | n/a<br>n/a<br>n/a<br>XX<br>XX |

TFR116341

Protocol : TFR116341

Protocol : TFR11
Population : Safety

Listing X.XX Listing of Oxygenation Data

Treatment: Placebo (BAL Collapsed lung) Inv.ID: PPD Subject: PPD

Visit/
Planned
Relative

Time/Time Peak Plateau

Since Vent. Vent. Mean Pa02/ Tidal Dose Oxy. Peep Pr. Pr. Airway Fi02 Pa02/ Ind. Sa02 Sa02/ Fi02 Vent Planned Pa02 (cm (cm Pressure Volume (cm Fi02 (%) (%) FiO2 H20) H20) H20) Actual Vent (mmHg) (%) (Imp) Mode (cm H2O) (mL) SCREENING/ Y 4 XX XX XX.X XX XX.X XX XX XX Pressure XX XX XX XXX.XX SCREENING/ controlled -0.38 XX.X XXX.XX

PART B/ Y 4 XX XX XX XX XX XX XX Pressure XX XX XX O.5 H/

0.5 H/ 0.02

TFR116341


Protocol : TFR116341 Population : Safety

Listing 227

Listing of SOFA and Change from Baseline SOFA Scores (Sequential Organ Failure Assessment)

Treatment: Placebo BID

| Inv.ID<br>/Subj | Visit | Study<br>Day | Respi-<br>ration | <br>Coagu- | _ | Central Nervous System | Renal | Observed<br>SOFA<br>Score<br>(Total) | Observed<br>Chg.<br>Baseline<br>SOFA [2] |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXXX | Baseline | 1 | 4 | 0 | 1 | 4 | 0 | 12 | 0 |
| | Day 4 | 4 | | | | | | | |
| | Follow-up<br>Day 7 | 7 | | | | | | | |
| XXXXXX/<br>XXXXX | Baseline | 1 | 1 | 0 | 2 | 4 | 0 | 11 | 0 |
| | Day 4 | 4 | 2 | 2 | 2 | 1 | 2 | 11 | 0 |
| | Follow-up<br>Day 7 | 7 | | 3 | 2 | 2 | 2 | | |

<sup>[1]:</sup> Individual organ function scored on a 0-4 point scale (0: Normal, 4: Most Abnormal)

<sup>[2]:</sup> String Assumptions made to obtain a baseline SOFA value

TFR116341


Protocol : TFR116341
Population : Safety

Listing of Day 28 Survival Status

Treatment: Placebo BID

| Inv./<br>Subj. | Age/<br>Sex | Randomization Date/<br>Event or Censoring<br>Date | Endpoint Description for 28 Day Survival | 28 Day<br>Survival<br>(days) |
|---|---|---|---|---|
| PPD<br>XXXXX | XX/<br>Male | XXOCT201X/<br>XXOCT201X | Event: Died | 6 |
| PPD<br>XXXXX | XX/<br>Male | XXAPR201X/<br>XXMAY201X | Censor: Last adequate asmt | 28 |

TFR116341


Protocol : TFR116341 Population : Safety

Listing 225

Listing of Day 28 Resource usage

Treatment: Placebo BID

| Subject | Inv. ID/Sex/Age/<br>Race/Death Date<br>(blank if alive) | Hospital-<br>isation Start/<br>End Date/<br>Discharged | ICU Start/<br>End Date/<br>Discharged | Vent.<br>free<br>days | Days<br>Alive in<br>Hospital | Days<br>Alive in<br>ICU |
|---|---|---|---|---|---|---|
| XXXXX | XXXXXX/M/XX/White -<br>White/Caucasian/European<br>Heritage/XXOCT201X | XXOCT201X/<br>XXOCT201X/<br>Y | XXOCT201X/<br>XXOCT201X/<br>Y | 0 | 6 | 6 |
| XXXXX | XXXXXX/M/XX/White -<br>White/Caucasian/European<br>Heritage/ | XXAPR201X/<br>/<br>N | XXAPR201X/<br>XXAPR201X/<br>Y | 8 | 28 | 4 |

Note: Evaluation Interval: Day of first dose to Day of first dose +27 days

Note: Partial days rounded up during computations

TFR116341

Page 1 of n : EFF\_L7 Example

Protocol : TFR116341 Population : Safety

Listing 229
Listing of Date and Time of Individual Subjects Surgical Procedures

| Treatment | Invid./<br>Subj. | Did the subject develop ARDS while in hospital? |
|---|---|---|
| Placebo BID | XXXXXX/<br>XXXXXX | Y |

TFR116341


Example : POP\_T1 Protocol : TFR116341

Population : n/a

Summary X.XX Summary of Subject Accountability (subjects constituting each Statistical Analysis Population)

| Treatment | Treatment | Number of individuals in population | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Descriptors | | Screen<br>Failures | Safety | PK | PP1 | PP2 | PP3 | IA1 | IA2 |
| Screening failures | n/a | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Main Treatment<br>Group<br>Descriptions | Placebo (BAL<br>Collapsed lung) | 0 | 15 | Х | х | x | x | x | х |
| • | Placebo (BAL | 0 | 25 | X | Χ | Х | X | X | Х |
| | Ventilated lung)<br>GSK2862277 26mg<br>IH (BAL Collapsed<br>lung) | 0 | 18 | Х | x | X | Х | Х | Х |
| | GSK2862277 26mg<br>IH (BAL Ventilated<br>lung) | 0 | 22 | X | Х | X | X | Х | Х |
| Alternative<br>Treatment Group | Placebo | 0 | 40 | Х | Х | Х | Х | Х | х |
| Descriptions #1 | GSK2862277 26mg<br>IH | 0 | 40 | Х | Х | Х | X | Х | х |
| Alternative<br>Treatment Group<br>Descriptions #2 | BAL Collapsed lung | 0 | 33 | Х | х | Х | Х | Х | X |
| | BAL Ventilated lung | 0 | 47 | Х | Х | Х | Х | Х | Х |

TFR116341

Example : POP\_L1 Protocol : TFR116341

Population : n/a

# Listing X.XX Listing of Subject Accountability (subjects constituting each Statistical Analysis Population)

| Inv ID | Screening<br>ID or<br>Subject ID | Actual<br>treatment | Screen<br>Failures | Safety | PK | PP1 | PP2 | PP3 | IA1 | IA2 | Translational<br>Sub-Study |
|---|---|---|---|---|---|---|---|---|---|---|---|
| PPD | | n/a | Y | • | • | • | • | | | • | |
| | | n/a | Y | | • | | | • | • | | • |
| | | n/a | Y | | | | | | - | • | |
| | | Placebo<br>BAL<br>Collapsed | · | Y | Y | Y | Y | Y | Y | Y | |
| | | Placebo<br>BAL<br>Collapsed | | Y | Υ | | | Y | ٠ | | Y |

Note: n/a = not applicable, PP = Per Protocol, Y = Included in population, "." = Excluded from population

Programming note: Label Center ID as Inv Id. If a subject was not a screen failure use their Subject ID. Break on Centres. Add additional columns if required